Apixaban versus Warfarin in Patients with Atrial Fibrillation (ARISTOTLE trial) **DUPLICATE-ARISTOTLE** May 26, 2021

#### 1. RCT Details

#### 1.1 Title

Apixaban versus Warfarin in Patients with Atrial Fibrillation (ARISTOTLE trial)

## 1.2 Intended aim(s)

To compare the risk of stroke or systemic embolism in atrial fibrillation (AF) patients with at least 1 risk factor for stroke with apixaban versus warfarin use.

## 1.3 Primary endpoint for replication

The primary outcome of the study was stroke (ischemic or hemorrhage) or systemic embolism.

## 1.3.1 Required power for primary endpoint and noninferiority margin (if applicable)

The test was designed for noninferiority. For non-inferiority, the 95% CI should not include  $\geq$  1.38 to declare noninferiority and 99% CI should not include  $\geq$  1.44 to declare noninferiority. Assuming average follow-up period of 1.8 years and a stroke or systemic embolism rate of 1.67 per 100 subject-years, the power of the study will be 90% with 18,000 randomized patients and 448 patients with primary outcome.

## 1.4 Secondary endpoint for replication (assay sensitivity) and RCT finding

Major bleeding; HR = 0.69 (95% CI 0.60-0.80)

## 1.5 Trial estimate

HR = 0.79 (95% CI 0.66-0.95) comparing apixaban vs warfarin (Granger et al., 2011)

## 2. Person responsible for implementation of replication in Aetion

Ajinkya Pawar, Ph.D., Hemin Lee, MD, MPH, and Dureshahwar Jawaid, MPH implemented the study design in the Aetion Evidence Platform. They are not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

## 3. Data Source(s)

United/Optum, MarketScan, Medicare

## 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

## **Design Diagram - ARISTOTLE TRIAL REPLICATION**



#### 5. Cohort Identification

#### 5.1 Cohort Summary

This study will involve a new user, parallel group, propensity score-matched, retrospective cohort study design comparing apixaban (any dose) to warfarin users. The patients will be required to have continuous enrollment during baseline period of 180 days before initiation of apixaban or warfarin (index date). We restrict the analyses to patients with a diagnosis of atrial fibrillation or atrial flutter in the 12 months prior to drug initiation along with risk factors for stroke or systemic embolism.

## 5.2 Important steps for cohort formation

New users (defined as no use in 180 days prior to index date) of an exposure and a comparator drug will be identified.

## 5.2.1 Eligible cohort entry dates

Market availability of apixaban in the U.S. started on December 28, 2012.

- For Medicare: January 01, 2013- December 31, 2017 (end of available data)
- For Marketscan: January 01, 2013- December 31, 2018 (end of available data)
- For Optum: January 01, 2013- December 31, 2019 (end of available data)

## 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date

Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in **Appendix A** and are summarized in the flowcharts below.

## 5.3 Flowchart of the study cohort assembly

## For apixaban vs. warfarin

| | Optum | | Truven | | Medicare | |
|---|---|---|---|---|---|---|
| | Less Excluded Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients | | 75,894,642 | | 200,203,908 | | 6,886,908 |

| Patients with claim for apixaban or warfarin | -74,955,393 | 939,249 | -199,377,918 | 825,990 | -2,374,503 | 4,512,405 |
|---|---|---|---|---|---|---|
| Excluded due to insufficient enrollment | -87,255 | 851,994 | -66,419 | 759,571 | -1,340,098 | 3,172,307 |
| Excluded due to prior use of warfarin | -390,759 | 461,235 | -426,157 | 333,414 | -1,802,129 | 1,370,178 |
| Excluded due to prior use of apixaban 5mg | -250,816 | 210,419 | -139,097 | 194,317 | -545,919 | 824,259 |
| Excluded because patient qualified in >1 exposure category | -21 | 210,398 | -5 | 194,312 | -51 | 824,208 |
| Excluded based on missing Age | -563 | 209,835 | 0 | 194,312 | -136 | 824,072 |
| Excluded based on missing Gender | 0 | 209,835 | 0 | 194,312 | 0 | 824,072 |
| Inclusion 3 - Age >= 18 | -82 | 209,753 | -187 | 194,125 | -68 | 824,004 |
| Inclusion #2- Afib (Inpatient, principal) 7 days prior OR Afib or flutter (any setting, any position) 2 diagnoses separated by 14 to 351 days, measured 365 days prior to drug initiation | -86406 | 123,347 | -96150 | 97,975 | -275611 | 548,393 |
| Inclusion #3- One or more of the 5 risk factor(s) for stroke | -2636 | 120,711 | -2941 | 95,034 | -5239 | 543,154 |
| Excluded based on Exclusion #2- Mitral Stenosis (any position, any setting) | -320 | 120,391 | -127 | 94,907 | -626 | 542,528 |
| Excluded based on Exclusion #3 - intracranial hemorrhage | -503 | 119,888 | -309 | 94,598 | -1823 | 540,705 |
| Excluded based on Exclusion #4 - Prosthetic heart valve | -1916 | 117,972 | -1004 | 93,594 | -8562 | 532,143 |
| Excluded based on Exclusion #5 - Uncontrolled hypertension | -701 | 117,271 | -218 | 93,376 | -1753 | 530,390 |
| Excluded based on Exclusion #6 - Active infective endocarditis | -83 | 117,188 | -43 | 93,333 | -456 | 529,934 |
| Excluded based on Exclusion #11 - Aspirin and Thienopyridine days supply overlap >7 days, measured 14 days prior to drug initiation | -10 | 117,178 | -24 | 93,309 | ** | ** |
| Excluded based on Exclusion #12- CCI (180 days)>=10 | -5059 | 112,119 | -1788 | 91,521 | -6685 | 523,239 |
| Excluded based on Exclusion #13- Active alcohol or drug abuse | -1381 | 110,738 | -563 | 90,958 | -5143 | 518,096 |
| Excluded based on Exclusion #14 - Ischemic stroke (w and w/o mention of cerebral infarction)- 7 days prior | -1178 | 109,560 | -558 | 90,400 | -5741 | 512,355 |
| Excluded based on Exclusion #15 - Severe renal impairment | -9885 | 99,675 | -5151 | 85,249 | -50219 | 462,136 |
| Excluded based on Exclusion #17 - Thrombocytopenia | -411 | 99,264 | -290 | 84,959 | -2040 | 460,096 |
| Excluded based on Exclusion #18 - Anemia | -933 | 98,331 | -1034 | 83,925 | -7386 | 452,710 |
| Excluded based on Exclusion #23b - Pregnancy | -3 | 98,328 | -9 | 83,916 | -11 | 452,699 |
| Final cohort | | 98,328 | | 83,916 | | 452,699 |

<sup>\*</sup> Medicare database includes all patients using a novel oral anticoagulant and a subset of patients using warfarin during 2011-2017.

\*\* = Data redacted to maintain compliance with CMS cell suppression policy

#### 6. Variables

## 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is initiation of apixaban. Initiation will be defined by no use of apixaban or a comparator in the prior 6 months before treatment initiation (washout period).

#### Comparator agents-

- Initiators of apixaban will be compared to initiators of-
  - Warfarin

#### 6.2 Covariates:

- Age
- Sex
- Combined Comorbidity Index (CCI), measured over the baseline covariate assessment period, defined as 180 days prior to and including index date

Covariates listed above represent only a small subset of covariates that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

## 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Primary Effectiveness outcomes of interest (definitions provided in **Appendix A**):

- Primary outcome: Stroke (hemorrhagic, ischemic) and systemic embolism
- Secondary outcomes: Individual components:
  - o Hospital admission for stroke (principal diagnosis position)

Hospital admission for systemic embolism (principal diagnosis position)

Control outcomes of interest (control outcomes only serve to assess aspects of study validity but are not further interpreted):

1. Major bleeding

#### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on the day of cohort entry. Because adherence in the real-world databases is expected to be much worse than in the trial, the AT analysis is the **primary** analysis, as it targets the relative hazard of outcomes on treatment.

For the AT analyses, the follow-up will start the day after initiation of apixaban and comparator and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Nursing home admission
  - Nursing home admissions are considered a censoring event because the data sources utilized typically provide little to no data on a patient, particularly on drug utilization, after admission. We will utilize this as an exclusion reason for cohorts for the same reason.
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (apixaban and comparator) plus a defined grace period (i.e., 10 days after the end of the last prescription's days' supply in main analyses).
- The date of augmentation or switching from exposure to comparator or vice versa or augmentation/switching to any other NOAC (e.g. switching from apixaban or warfarin to rivaroxaban would be a censoring event);
  - o A dosage change on the index treatment does not fulfill this criterion
  - o An added treatment that is not part of the exposure or comparator group does not fulfill this criterion

For the intention-to-treat (ITT) analyses, the censoring based on the augmentation/switching and treatment discontinuation will be replaced with a maximum allowed follow-up time of 365 days.

#### 7. Initial Feasibility Analysis

#### Aetion report name:

Optum- <a href="https://bwh-dope.aetion.com/projects/details/707/results/58231/result/0">https://bwh-dope.aetion.com/projects/details/707/results/58231/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/709/results/58232/result/0">https://bwh-dope.aetion.com/projects/details/708/results/58232/result/0</a>
Medicare- <a href="https://bwh-dope.aetion.com/projects/details/709/results/58233/result/0">https://bwh-dope.aetion.com/projects/details/709/results/58233/result/0</a>

Date conducted: 9/4/2020

Complete Aetion feasibility analysis using age, sex, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed nor will incidence rates stratified by treatment group.

- Report patient characteristics by treatment group
- Report summary parameters of study population
- Report median follow-up time by treatment group
- Report reasons for censoring in the overall study population

#### 8. Initial Power Assessment

## Aetion report name:

For apixaban vs. warfarin

Optum- https://bwh-dope.aetion.com/projects/details/711/results/53838/result/0
Marketscan- https://bwh-dope.aetion.com/projects/details/712/results/53839/result/0
Medicare- https://bwh-dope.aetion.com/projects/details/713/results/53840/result/0

Date conducted: 05/12/2020

In order to complete the initial power analysis, the dummy outcome of a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. Complete a 1:1 PS-matched comparative analysis using this outcome. PS should include only 3 covariates: age, sex, and combined

comorbidity index. Power calculations are based on the formulas from Chow et al. (2008).

• Stop analyses until feasibility and power are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 6/3/20 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 6/30/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

#### Aetion report name:

For apixaban vs. warfarin

Optum- https://bwh-dope.aetion.com/projects/details/711/results/57927/result/0

Marketscan- https://bwh-dope.aetion.com/projects/details/712/results/57928/result/0

Medicare- https://bwh-dope.aetion.com/projects/details/713/results/57982/result/0

Date conducted: 8/27/2020 (Medicare 8/30/2020)

After review of initial feasibility and power analyses, complete creation of the remaining covariates (see Table 1 below for list of covariates). Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates (excluding laboratory values, which are missing in some patients).

• Provide plot of PS distributions stratified by treatment group.

Note- Please refer to **Appendix B**.

Report covariate balance after matching.

Note- For Table 1, please refer to Appendix B.

• Report reasons for censoring by treatment group.

| | Overall | Referent | Exposure |
|---|---|---|---|
| Dummy Outcome | 0 (0.00%) | 0 (0.00%) | 0 (0.00%) |
| Death | 3,281 (1.49%) | 1,664 (1.51%) | 1,617 (1.47%) |
| Start of an additional exposure | 4,890 (2.22%) | 3,122 (2.83%) | 1,768 (1.60%) |
| End of index exposure | 157,724 (71.52%) | 78,153 (70.88%) | 79,571<br>(72.17%) |
| Specified date reached (Dec 17/Dec 18/Dec 19) | 23,353 (10.59%) | 10,720 (9.72%) | 12,633<br>(11.46%) |
| End of patient enrollment | 9,203 (4.17%) | 4,146 (3.76%) | 5,057 (4.59%) |
| Switch to other NOACs (for censoring) + nursing home admission | 22,067 (10.01%) | 12,454 (11.30%) | 9,613 (8.72%) |

• Report follow-up time by treatment group.

| Median Follow-Up Time (Days) [IQR] | | | |
|---|---|---|---|
| Patient Group Optum Truven Medicare | | | |
| Overall Patient Population | 98 [38-192] | 98 [38-213] | 98 [38-213] |
| Referent | 98 [38-182] | 98 [38-180] | 98 [39-191] |
| Exposure | 98 [38-211] | 98 [38-264] | 98 [38-242] |

• Report overall risk of the primary outcome.

| | Optum | MarketScan | Medicare | Pooled |
|-------------------------|-------|------------|----------|--------|
| Risk per 1,000 patients | 3.61 | 3.6 | 5.64 | 5.06 |

## 10. Final Power Assessment

## Date conducted:

• Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9.

All other parameters in the table should be the same as in Section 8.

• For apixaban vs. warfarin

## o Pooled

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 110,259 | Reference | 110,259 |
| Exposed | 110,259 | Exposed | 110,259 |
| Risk per 1,000 patients | 5.06 | Risk per 1,000 patients | 5.06 |
| Desired HR from RCT | 0.79 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.38 |
| Number of events expected | 1115.82108 | Number of events expected | 1115.82108 |
| Power | 0.975982555 | Power | 0.999686272 |

o Optum

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 15,273 | Reference | 15,273 |
| Exposed | 15,273 | Exposed | 15,273 |
| Risk per 1,000 patients | 3.61 | Risk per 1,000 patients | 3.61 |
| Desired HR from RCT | 0.79 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.38 |
| Number of events expected | 110.27106 | Number of events expected | 110.27106 |
| Power | 0.235746761 | Power | 0.394017124 |

## o MarketScan

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 14,849 | Reference | 14,849 |
| Exposed | 14,849 | Exposed | 14,849 |
| Risk per 1,000 patients | 3.6 | Risk per 1,000 patients | 3.60 |
| Desired HR from RCT | 0.79 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.38 |
| Number of events expected | 106.9128 | Number of events expected | 106.9128 |
| Power | 0.229997009 | Power | 0.384067948 |

Effectiveness research with Real World Data to support FDA's regulatory decision making

Medicare

| Superiority Analysis | | Non-inferiority Analysis | |
|---|---|---|---|
| Number of patients matched | | Number of patients matched | |
| Reference | 80,137 | Reference | 80,137 |
| Exposed | 80,137 | Exposed | 80,137 |
| Risk per 1,000 patients | 5.64 | Risk per 1,000 patients | 5.64 |
| Desired HR from RCT | 0.79 | Assumed HR from RCT | 1 |
| Alpha (2-sided) | 0.05 | Alpha (2-sided) | 0.05 |
| | | Non-inferiority margin | 1.38 |
| Number of events expected | 903.94536 | Number of events expected | 903.94536 |
| Power | 0.943359069 | Power | 0.998023363 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Jessica Franklin | Date reviewed: | 9/8/20 |
|-------------------------|------------------|----------------|---------|
| Reviewed by FDA: | Ken Quinto | Date reviewed: | 9/29/20 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

## 11. Study Confidence and Concerns

<u>Deadline for voting on study confidence and listing concerns:</u>

Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the

success of the RWD study in the <u>Google Form</u>. This form also provides space for reviewers to list any concerns that they feel may contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the individual respondent.

• After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

## 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

• Register the study on clinicalTrials.gov and upload this document.

## 13. Comparative Analyses

Aetion report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 For sensitivity analyses:

## 14. Requested Results

## 14.1 <u>Table 1: Baseline characteristics before and after adjustment</u>

| Variable | Before adjustment | | After adjustment | | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

## 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

## 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

## 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |
| Analysis 1 | | | | | |
| Analysis 2 | | | | | |

HR, Hazard Ratio; Cl, Confidence Interval.

Effectiveness research with Real World Data to support FDA's regulatory decision making

## 14.5 Table 5: Results from secondary analyses;

## 15. References

Chow S, Shao J, Wang H. 2008. *Sample Size Calculations in Clinical Research*. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. **page** 177

Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC. Apixaban versus warfarin in patients with atrial fibrillation. New England Journal of Medicine. 2011; 365(11):981-92.

| # | ARISTOTLE trial definitions | Implementation in routine care | References/Rationale | Color coding |
|---|---|---|---|---|
| | Trial details- Primary approval, Unintended | S with label change | Please see the following Google Drive for further details or any missing information: <a href="https://drive.google.com/open7id=1WD618wrvwV/EaXrfl.TcuK-VCcnb6b-gV">https://drive.google.com/open7id=1WD618wrvwV/EaXrfl.TcuK-VCcnb6b-gV</a> | Criteria |
| | EXPOSURE vs. COMPARI: | SON | ICD-10 codes are not listed in this document because of excel cell size<br>limitations and excessive number of ICD-10 codes. Full ICD-10 code lists will<br>be available in the above Google Drive Folder (link above). ICD-9 to ICD-10<br>code conversions were completed using a SAS macro that implements<br>forward/backward mapping based on the CMS ICD-9 to ICD-10 mapping:<br>https://www.hbber.org/data/icd9-icd-10-cm-and-ocs-crosswalk-general-<br>squivalence-mapping.html | Adequate mapping in claims |
| | apixaban (at a dose of 5 mg twice daily) versus warfarin (target international normalized ratio, 2.0 to 3.0) | Apixaban 5 mg vs warfarin | | Intermediate mapping in claims |
| | PRIMARY OUTCOME | | | Poor mapping or cannot be measured in claims |
| | The primary outcome was ischemic or hemorrhagic stroke or systemic embolism. | Measured 1 days after drug initiation in diagnosis position specified below and inpatient care setting: For stroke: For stroke: Primary diagnosis position in inpatient care setting 430.xx Subarachnoid hemorrhage (SAH) 431.xx Intracerebral hemorrhage (ICH) 433.xx Intracerebral hemorrhage (ICH) 433.xx (excluding 434.xx) Occlusion and stenosis of precerebral arteries with cerebral infarction 434.xx (excluding 434.xx) Occlusion and stenosis of cerebral arteries with cerebral infarction 436.x Acute, but ill-defined cerebrovascular events Systemic embolism: (inpatient, any position) ICD-9:444.xx (arterial embolism) ICD-10:174.x arterial embolism and thrombosis | For stroke: PPV of 85% or higher for ischemic stroke PPV ranging from 80% to 98% for hemorrhagic stroke PPV ranging from 80% to 98% for hemorrhagic stroke PPV ranging from 80% to 98% for hemorrhagic stroke PAndrade SE, Harrod LR, Tijla, et al. A systematic review of validated methods for identifying cerebrovascular accident or transient ischemic attack using administrative data. Pharmacoepidemiology and Drug Safety 2012;21 Suppl 1:100-28.] → Tirschwell DL, Longstreth WT, Jr. Validating administrative data in stroke research. Stroke, a journal of cerebral circulation 2002;33:2465-70.] → Tillowinie CL, Mitchel E, Gideon PS, Varas-Lorenzo C, Castellsague J, Griffin MR. Validation of ICO 9 codes with a high positive predictive value for incident strokes resulting in hospitalization using Medicaid health data. Pharmacoepidemiology and drug safety 2008;17:20-6.] | Can't be measured in claims but not important for the analysis |
| | INCLUSION CRITERIA | Measured on the day of drug initiation | | |
| 1 | Age≥18 years | Age>=18 years | | |
| | In atrial fibrillation or atrial flutter not due to a reversible cause and documented by ECG at the time of enrollment. | Measured 7 days prior to and including day of drug initiation in primary diagnosis position and inpatient care setting <u>Atrial fibrillation</u> (CD-9 diagnosis: 427.31, 427.32 Reversible causes listed in exclusion criteria. | | |
| 2b | • If not in atrial fibrillation/flutter at the time of enrollment, must have atrial fibrillation/flutter documented on two separate occasions, not due to a reversible cause at least 2 weeks apart in the 12 months prior to enrollment. Atrial fibrillation/flutter may be documented by ECG, or as an episode lasting at least one minute on a rhythm strip, Holter recording, or intracardiac electrogram (from an implanted pacemaker or defibrillator). | Measured 365 days prior to and including day of drug initiation 2 diagnoses of Atrial fibrillation/flutter separated by 14 to 351 days in any diagnosis position and inpatient or outpatient care setting Atrial fibrillation or flutter ICD-9 diagnosis: 427.31, 427.32 Reversible causes listed in exclusion criteria. | | |
| 3 | One or more of the following risk factor(s) for stroke: | | | |
| 3a | • Age 75 years or older | Measured on the day of drug initiation Age >= 75 | | |
| 3b | • Prior stroke, TIA or systemic embolus | Measured any time prior to and including day of drug initiation in diagnosis position and care setting specified below Stroke (Inpatient care setting, primary diagnosis position) ICD-9 diagnosis: 430.x, 431.xx, 433.xx, 434.xx, 436.xx ICD-10 diagnosis: ICB.5x, ICB.3x, ICB.3x, ICB.3x, ICB.3x, ICB.5x, I | | |
| 30 | ■ Either <u>symptomatic</u> congestive heart failure within 3 months or left ventricular dysfunction with an <u>LV ejection fraction</u> ( <u>LVEF) ≤ 40%</u> by echocardiography, radionuclide study or contrast angiography | Measured 90 days prior to and including day of drug initiation in any diagnosis position and inpatient care setting Heart failure ICD-9 diagnosis: 428.x, 398.91, 402.01, 402.11, 402.91, 404.01, 404.11, 404.91, 404.03, 404.13, 404.93 ICD-10 diagnosis: 109.81, I11.0, I13.0, I13.2, I50.1x, I50.2x, I50.3x, I50.4x, I50.9 | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study," BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRISS) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA 118.039177 | |

| 3d | Diabetes mellitus | Measured any time prior to and including day of drug initiation in any diagnosis position and any care setting Type 1. Type 2 diabetes mellitus ICD-9 diagnosis: 250.x1, 250.x3, 250.x0, 250.x2 ICD-10 diagnosis: E10.x, E11.x | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with<br>canagliflozin versus other non-gliflozin antidiabetic drug:s population based<br>chohort study." MBM 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin<br>Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr<br>8. doi:10.1167/CIRCULATIONAHA.118.039177 |
|---|---|---|---|
| Зе | Hypertension requiring pharmacological treatment | Measured 180 days to 3650 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Hypertension ICD-9 diagnosis: 401.x - 405.x ICD-10 diagnosis: 101.x - 113.x, 115.x Plus following medication use on the same day: (Hypertension Medications sheet) ACE/ARB/beta-blocker/Calcium channel blockers/thiazides/loop diuretics/other diuretics/other medications | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Fallure Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin Comparative Effectiveness and Safety (EMPRIS) Study." Circulation. 2019 Apr 8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| 4 | Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the treatment period of the study or for 2 weeks after the last dose of study medication, whichever is longer, in such a manner that the risk of pregnancy is minimized. | N/A - Incorporated in the exclusion criteria. | |
| 5 | WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within | N/A - Incorporated in the exclusion criteria. | |
| - | 48 hours prior to the start of investigational product. All subjects must provide signed written informed consent. | N/A | |
| ٣ | EXCLUSION CRITERIA | | |
| 1 | Atrial fibrillation or flutter due to <b>reversible causes</b> (e.g. thyrotoxicosis, pericarditis) | N/A | |
| 2 | Clinically significant (moderate or severe) mitral stenosis | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care settling Mitral stenosis (ICD-9 diagnosis: 96.0x, 396.1x, 394, 746.5 ICD-10 diagnosis: 134.2x, 105.1x, 105.2x | |
| 3 | Increased bleeding risk that is believed to be a contraindication to oral anticoagulation (e.g. previous intracranial hemorrhage) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient care setting Intracranial hemorrhage ICD-9 diagnosis: 430.x, 431.x, 432.x | |
| 4 | Conditions other than atrial fibrillation that require chronic anticoagulation (e.g. prosthetic mechanical heart valve) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting ICD-9 diagnosis: V43.3x ICD-10 diagnosis: 295.2x CPT procedure codes: (TAVR with prosthetic valve) 33361, 33362, 33363, 33364, 33365, 33366, 33367, 33368, 33369, 33477, 0483T, 0484T, 0569T, 0570T | |
| 5 | Persistent, uncontrolled hypertension (systolic BP > 180 mm Hg, or diastolic BP > 100 mm Hg) | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or ED care setting Malignant hypertension ICD-9 diagnosis: 401.0x Hypertensive urgency/ Hypertensive crisis ICD-10 diagnosis: 116.xx | |
| | Active infective endocarditis | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Endocarditis ICD-9 diagnosis: 421.xx ICD-10 diagnosis: 133.xx | |
| 7 | Planned major surgery Planned atrial fibrillation or flutter ablation procedure | N/A | |
| 8 | Planned atrial fibrillation or flutter ablation procedure Use of an <b>unapproved</b> , investigational drug or device within the past 30 days | N/A<br>N/A | |
| 10 | Required treatment with aspirin > 165 mg/day | N/A | |
| | Simultaneous treatment with both aspirin and a thienopyridine (e.g., clopidogrel, ticlopidine) | Measured 14 days prior to and including day of drug initiation Days supply overlap of >7 days of: 1) Prescription for any dose of Aspirin (Note: Unable to capture over the counter use.) AND 2) Prescription for any dose of Clopidogrel/Ticlopidine/prasugrel | |
| 12 | Severe comorbid condition with life expectancy of ≤ 1 year | Measured 180 days prior to and including day of drug initiation<br>CCI ≥ 10 | |

| 13 | Active alcohol or drug abuse, or psychosocial reasons that make study participation impractical | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting <u>Alcohol abuse or dependence</u> ICD-9 diagnosis: 291.xx, 303.xx, 305.0x, 571.0x, 571.1x, 571.2x, 571.3x, 357.5x, 425.5x, | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with<br>canagilflozin versus other non-gliflozin antidiabetic drugs: population based<br>chohort study." BMJ 2018;366:119 http://dx.doi.org/10.1136/bmj.kl.19 Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure |
|---|---|---|---|
| | | E860.0x, V1.1.3x<br><u>Drux abuse or dependence</u><br>ICD-9 diagnosis: 292.xx, 304.xx, 305.2x-305.9x, 648.3x, 965.0x, 967.x, 969.x, 970.81 | Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin<br>Comparative Effectiveness and Safety (EMPRISE) Study." Circulation. 2019 Apr<br>8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | | Measured 7 days prior to and including day of drug initiation in primary diagnosis position and inpatient care setting | Patorno, Elisabetta et al. "Cardiovascular outcomes associated with canagliflozin versus other non-gliflozin antidiabetic drugs: population based cohort study." BMJ 2018;360:k119 http://dx.doi.org/10.1136/bmj.k119 |
| 14 | Recent ischemic stroke (within 7 days) | Ischemic stroke<br>ICD-9 diagnosis: 433.xx, 434.xx, 436.xx | Patorno, Elisabetta et al. "Empagliflozin and the Risk of Heart Failure<br>Hospitalization in Routine Clinical Care: A First Analysis from the Empagliflozin<br>Comparative Effectivenes and Safety (EMPRIS) Study." Circulation. 2019 Apr<br>8. doi: 10.1161/CIRCULATIONAHA.118.039177 |
| | | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting | |
| 15 | Severe renal insufficiency (serum creatinine > 2.5 mg/dL or a calculated creatinine clearance < 25 mL/min, See Section 6.3.2.2) | CKD stage 4/5/ESRD<br>ICD-9 diagnosis: 585.4x, 585.5x, 585.6x<br>ICD-10 diagnosis: N18.4x, N18.5x, N18.6x | |
| | | OR | |
| _ | ALT or AST > 2X ULN or a Total Bilirubin ≥ 1.5X ULN (unless an alternative causative factor [e.g., Gilbert's syndrome] is | <u>Dialysis/ Renal transplant</u> code list in sheet "Dialysis and Renal Transplant" | |
| 16 | identified) | N/A | |
| 17 | Platelet count ≤ 100,000/ mm3 | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting <u>Thrombocytopenia</u> | |
| | | ICD-9 diagnosis: 287.3x, 287.4x, 287.5x<br>ICD-10 diagnosis: D69.3x, D69.4x, D69.5x, D69.6x | |
| 18 | Hemoglobin < 9 g/dL | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting | |
| | | Anemia (non-deficiency/neoplastic/chemotherapy/hemorrhagic assoicated) ICD-9 diagnosis: 282.x, 283.x, 284.x, 285.0, 285.2 (acute posthemorrhagic anemia), 285.22 (anemia of neoplastic disease), 285.3 (antineoplastic chemotherapy induced anemia) ICD-10 diagnosis: D55 - D62, D63.0 | |
| | Inability to comply with INR monitoring | N/A | |
| | Prior randomization into an apixaban clinical study | N/A | |
| | Prisoners or subjects who are involuntarily incarcerated Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness | N/A<br>N/A | |
| | Women of child bearing potential (WOCBP) unwilling or unable to use an acceptable method to avoid pregnancy: | N/A | |
| | WOCBP using a prohibited contraceptive method | N/A | |
| | •WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal [defined as amenor/thea≥12 consecutive months; or women on hormone replacement therapy (HRT) with documented serum folliclestimulating hormone (FSH) level > 35 milly IMpL. | Measured 180 days prior to and including day of drug initiation in any diagnosis position and inpatient or outpatient care setting Codes are in the sheet "Pregnancy" | |
| 23b | Even women who are using <b>oral contraceptives</b> , other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of child bearing potential | | |
| | Women who are pregnant or breastfeeding | | |
| 23d | Women with a positive pregnancy test on enrollment or prior to administration of investigational product. | | |

| Comparator | Active | |
|---|---|---|
| No. of Patients | | 18,201 |
| Blinding | Double-blinded | |
| Trial finding | HR 0.79; 95% CI, 0.66 to 0.95; P<0.001 for noninferiority; P = 0.01 for superiority | |
| Measurable endpoint | Primary outcomes:<br>Effectiveness: ischemic or hemorrhagic stroke or systemic embolism<br>Safety: Major bleeding | |
| pNDA Indication | For the prevention of stroke and systemic embolism resulting from nonvalvular atrial fibrillation | |
| <u>Year</u> | | 2012 |
| <u>Sponsor</u> | Bristol-Myers Squibb | |
| Generic Name | apixaban | |
| Brand Name | <u>Eliquis</u> | _ |
| Therapeutic Area | Cardiology/Vascular Diseases | |
| <u>NCT</u> | NCT00412984 | |
| Trial Name (with web links) | <u>ARISTOTLE</u> | |
| <u>Trial ID</u> | pNDA15 | |

| Hypertension medication | |
|---|---|
| ACE inhibitor | Benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril |
| ARB | Azilsartan, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan |
| Beta blocker | Acebutolol, atenolol, betaxolol, bisoprolol, carteolol, carvedilol, esmolol, labetalol, metoprolol tartrate, metoprolol succinate, propranolol, penbutolol, pindolol, nadolol, nebivolol, sotalol, timolol |
| Calcium channel blocker | Diltiazem, mibefradil, verapamil, amlodipine, clevidipine,<br>bepridil, felodipine, isradipine, nicardipine, nifedipine,<br>nimodipine, nisoldipine |
| Other hypertension drugs | Doxazosin, eplerenone, prazosin, terazosin, clonidine, guanabenz, guanadrel, guanethidine, guanfacine, hydralazine, methyldopa, metyrosine, reserpine, minoxidil, aliskiren |
| Thiazides | Benzthiazide, chlorothiazide, chlorthalidone, cyclothiazide, hydrochlorothiazide, hydroflumethiazide, indapamide, methyclothiazide, metolazone, polythiazide, quinethazone, trichlormethiazide, bendroflumethiazide |
| Loop diuretics | Furosemide, bumetanide, torsemide, ethacrynic acid |
| Other diuretics | Amiloride, eplerenone, spironolactone, triamterene |

#### Dialysis codes

ESRD, defined as 2 codes (either inpatient or outpatient), separated by at least 30 days

Codes include:

- ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

- ICD9 dx codes:

585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis)

585.6x, End stage renal disease (for ESRD with dialysis)

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

- CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per month

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription

90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older

90989, Dialysis training, patient, including helper where applicable, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512, Home visit for hemodialysis

- HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility

G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/2 or 3 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.

G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem

S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per diem

OR

Kidney transplant, defined as either 1 inpatient or 1 outpatient code

Codes include:

-ICD9 dx codes:

V42.0x, Kidney transplant status

996.81 Complications of transplanted kidney

-ICD9 prox codes:

55.6x, Transplant of kidney (Exclude 55.61)

- CPT/L codes

## Pregnancy Dx codes 650 NORMAL DELIVERY 660 OBSTRUCTED LABOR 661 ABNORMALITY OF FORCES OF LABOR 662 LONG LABOR 663 UMBILICAL CORD COMPLICATIONS DURING LABOR AND DELIVERY 664 TRAUMA TO PERINEUM AND VULVA DURING DELIVERY 665 OTHER OBSTETRICAL TRAUMA 667 RETAINED PLACENTA OR MEMBRANES WITHOUT HEMORRHAGE 668 COMPLICATIONS OF THE ADMINISTRATION OF ANESTHETIC OR OTHER SEDATION IN LABOR AND DELIVERY 669.94 UNSPECIFIED COMPLICATION OF LABOR AND DELIVERY POSTPARTUM CONDITION OR COMPLICATION V24 POSTPARTUM CARE AND EXAMINATION V24.0 POSTPARTUM CARE AND EXAMINATION IMMEDIATELY AFTER DELIVERY V24.1 POSTPARTUM CARE AND EXAMINATION OF LACTATING MOTHER V24.2 ROUTINE POSTPARTUM FOLLOW V27 OUTCOME OF DELIVERY V27.0 MOTHER WITH SINGLE LIVEBORN V27.1 MOTHER WITH SINGLE STILLBORN V27.2 MOTHER WITH TWINS BOTH LIVEBORN V27.3 MOTHER WITH TWINS ONE LIVEBORN AND ONE STILLBORN V27.4 MOTHER WITH TWINS BOTH STILLBORN V27.5 MOTHER WITH OTHER MULTIPLE BIRTH ALL LIVEBORN V27.6 MOTHER WITH OTHER MULTIPLE BIRTH SOME LIVEBORN V27.7 MOTHER WITH OTHER MULTIPLE BIRTH ALL STILLBORN V27.9 MOTHER WITH UNSPECIFIED OUTCOME OF DELIVERY **Procedure codes** 72.0 LOW FORCEPS OPERATION 72.1 LOW FORCEPS OPERATION WITH EPISIOTOMY 72.2 MID FORCEPS OPERATION 72.21 MID FORCEPS OPERATION WITH EPISIOTOMY 72.29 OTHER MID FORCEPS OPERATION 72.3 HIGH FORCEPS OPERATION 72.31 HIGH FORCEPS OPERATION WITH EPISIOTOMY 72.39 OTHER HIGH FORCEPS OPERATION

- 72.4 FORCEPS ROTATION OF FETAL HEAD
- 72.5 BREECH EXTRACTION
- 72.51 PARTIAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.52 OTHER PARTIAL BREECH EXTRACTION
- 72.53 TOTAL BREECH EXTRACTION WITH FORCEPS TO AFTERCOMING HEAD
- 72.54 OTHER TOTAL BREECH EXTRACTION
- 72.6 FORCEPS APPLICATION TO AFTERCOMING HEAD
- 72.7 VACUUM EXTRACTION
- 72.71 VACUUM EXTRACTION WITH EPISIOTOMY
- 72.79 OTHER VACUUM EXTRACTION
- 72.8 OTHER SPECIFIED INSTRUMENTAL DELIVERY
- 72.9 UNSPECIFIED INSTRUMENTAL DELIVERY
- 73.0 ARTIFICIAL RUPTURE OF MEMBRANES
- 73.01 INDUCTION OF LABOR BY ARTIFICIAL RUPTURE OF MEMBRANES
- 73.09 OTHER ARTIFICIAL RUPTURE OF MEMBRANES
- 73.1 OTHER SURGICAL INDUCTION OF LABOR
- 73.2 INTERNAL AND COMBINED VERSION AND EXTRACTION
- 73.21 INTERNAL AND COMBINED VERSION WITHOUT EXTRACTION
- 73.22 INTERNAL AND COMBINED VERSION WITH EXTRACTION
- 73.3 FAILED FORCEPS
- 73.4 MEDICAL INDUCTION OF LABOR
- 73.5 MANUALLY ASSISTED DELIVERY
- 73.51 MANUAL ROTATION OF FETAL HEAD
- 73.59 OTHER MANUALLY ASSISTED DELIVERY
- 73.6 EPISIOTOMY
- 73.8 OPERATIONS ON FETUS TO FACILITATE DELIVERY
- 73.9 OTHER OPERATIONS ASSISTING DELIVERY
- 73.91 EXTERNAL VERSION ASSISTING DELIVERY
- 73.92 REPLACEMENT OF PROLAPSED UMBILICAL CORD
- 73.93 INCISION OF CERVIX TO ASSIST DELIVERY
- 73.94 PUBIOTOMY TO ASSIST DELIVERY
- 73.99 OTHER OPERATIONS ASSISTING DELIVERY
- 74.0 CLASSICAL CESAREAN SECTION
- 74.1 LOW CERVICAL CESAREAN SECTION
- 74.2 EXTRAPERITONEAL CESAREAN SECTION

- 74.3 REMOVAL OF EXTRATUBAL ECTOPIC PREGNANCY
- 74.4 CESAREAN SECTION OF OTHER SPECIFIED TYPE
- 74.9 CESAREAN SECTION OF UNSPECIFIED TYPE
- 74.91 HYSTEROTOMY TO TERMINATE PREGNANCY
- 74.99 OTHER CESAREAN SECTION OF UNSPECIFIED TYPE
- 75.4 MANUAL REMOVAL OF RETAINED PLACENTA
- 75.5 REPAIR OF CURRENT OBSTETRIC LACERATION OF UTERUS
- 75.6 REPAIR OF OTHER CURRENT OBSTETRIC LACERATION
- 75.7 MANUAL EXPLORATION OF UTERINE CAVITY, POSTPARTUM
- 75.9 OTHER OBSTETRIC OPERATIONS

Appendix B: Apixaban vs Warfarin



# Table 1: Unmatched

| | | | | Unmatched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Optur<br>Reference - Warfarin | n<br>Apixaban (any dose) | Truv<br>Reference - Warfarin | Apixaban (any dose) | Medic<br>Reference - Warfarin | Apixaban (any dose) | Reference - Warfarin | POOLED<br>Apixaban (any dose) | St. Diff. |
| Number of patients<br>Age | 46,518 | 51,684 | 47,096 | 36,714 | 277,248 | 174,898 | 370,862 | 263,296 | |
| mean (sd)<br>median (IQR) | 75.30 (8.70)<br>77.00 (70.00, 82.00) | 74.09 (9.49)<br>75.00 (68.00, 81.00) | 74.33 (11.29)<br>76.00 [66.00, 83.00] | 69.50 (12.30)<br>69.00 (60.00, 79.00) | 77.79 (8.41)<br>78.00 (72.00.84.00) | 77.33 (8.13)<br>77.00 (72.00, 83.00) | 77.04 (8.86) | 75.60 (9.09) | 0.16 |
| Age categories without zero category | | | | | , | | | | |
| 18 - 54; n (%)<br>55 - 64; n (%) | 1,093 (2.3%)<br>4,064 (8.7%) | 1,861 (3.6%)<br>5,668 (11.0%) | 2,201 (4.7%)<br>8,470 (18.0%) | 3,698 (10.1%)<br>11,308 (30.8%) | 2,803 (1.0%)<br>8,161 (2.9%) | 1,281 (0.7%)<br>4,224 (2.4%) | 6,097 (1.6%)<br>20,695 (5.6%) | 6,840 (2.6%)<br>21,200 (8.1%) | -0.01<br>-0.01 |
| 65 - 74; n (%)<br>>= 75; n (%) | 13,880 (29.8%)<br>27,481 (59.1%) | 16,773 (32.5%)<br>27,382 (53.0%) | 10,436 (22.2%)<br>25,989 (55.2%) | 7,808 (21.3%)<br>13,900 (37.9%) | 83,745 (30.2%)<br>182.539 (65.8%) | 59,633 (34.1%)<br>109,760 (62.8%) | 108,061 (29.1%)<br>236,009 (63.6%) | 84,214 (32.0%)<br>151,042 (57.4%) | -0.01<br>0.01 |
| Gender without zero category- United<br>Males: n (%) | 25.508 (54.8%) | 25,542 (49.4%) | 26,865 (57.0%) | 20,513 (55.9%) | 135.230 (48.8%) | 76,603 (43.8%) | 187,603 (50.6%) | 122,658 (46.6%) | 0.01 |
| Females; n (%) | 21,010 (45.2%) | 26,142 (50.6%) | 20,231 (43.0%) | 16,201 (44.1%) | 142,018 (51.2%) | 98,295 (56.2%) | 183,259 (49.4%) | 140,638 (53.4%) | -0.01 |
| Race without zero categoryWhite; n (%) | N/A | N/A | N/A | N/A | 259,440 (93.6%) | 162,140 (92.7%) | 259,440 (93.6%) | 162,140 (92.7%) | #REF! |
| Black; n (%)<br>Asian; n (%) | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | 8,892 (3.2%)<br>2,208 (0.8%) | 5,772 (3.3%)<br>1.884 (1.1%) | 8,892 (3.2%)<br>2.208 (0.8%) | 5,772 (3.3%)<br>1.884 (1.1%) | 0.00 |
| Hispanic; n (%)<br>North American Native: n (%) | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | 2,251 (0.8%)<br>773 (0.3%) | 1,567 (0.9%)<br>394 (0.2%) | 2,251 (0.8%)<br>773 (0.3%) | 1,567 (0.9%)<br>394 (0.2%) | 0.00 |
| Other/Unknown; n (%) | N/A | N/A | N/A | N/A | 3,684 (1.3%) | 3,141 (1.8%) | 3,684 (1.3%) | 3,141 (1.8%) | 0.00 |
| Region without zero category-United v3 (lumping<br>missing&other category with West) | | | | | | | | | |
| Northeast; n (%)<br>South; n (%) | 6,849 (14.7%)<br>15.118 (32.5%) | 6,040 (11.7%)<br>23,275 (45.0%) | 11,511 (24.4%)<br>15,235 (32.3%) | 7,944 (21.6%)<br>9,410 (25.6%) | 62,468 (22.5%)<br>95,216 (34.3%) | 32,667 (18.7%)<br>77.615 (44.4%) | 80,828 (21.8%)<br>125,569 (33.9%) | 46,651 (17.7%)<br>110,300 (41.9%) | 0.01<br>-0.01 |
| Midwest; n (%) | 10,705 (23.0%) | 10,011 (19.4%) | 12,823 (27.2%)<br>7.324 (15.6%) | 14,967 (40.8%)<br>4,225 (11.5%) | 73,735 (26.6%) | 36,209 (20.7%) | 97,263 (26.2%) | 61,187 (23.2%) | 0.01 |
| West; n (%)<br>Unknown+missing; n (%) | 13,846 (29.8%)<br>N/A | 12,358 (23.9%)<br>N/A | 7,324 (15.6%)<br>203 (0.4%) | 4,225 (11.5%)<br>168 (0.5%) | 45,829 (16.5%)<br>N/A | 28,407 (16.2%)<br>N/A | 66,999 (18.1%)<br>203 (0.4%) | 44,990 (17.1%)<br>168 (0.5%) | 0.00<br>0.00 |
| Calendar Time by day (March 29, 2013 to CED)mean (sd) | 1.024.53 (739.16) | 1.652.15 (579.60) | 535.68 (509.15) | 1,132.76 (552.83) | 3,905 (1.4%) | 2,792 (1.6%) | 3115.82 (318.51) | 2336.89 (329.48) | 2.40 |
| median (IOR) | 943.00 (351.00,<br>1.649.00) | 1,757.00 [1,289.00, | 389.00 [121.00, 838.00] 1 | | 8,444 (3.0%) | 4,048 (2.3%) | | | |
| CV Covariates | , | | | | | | | | |
| Ischemic heart disease; n (%)<br>Acute MI; n (%) | 15,366 (33.0%)<br>1,062 (2.3%) | 18,835 (36.4%)<br>1,789 (3.5%) | 15,378 (32.7%)<br>1,106 (2.3%) | 12,189 (33.2%)<br>1,178 (3.2%) | 85,977 (31.0%)<br>5,202 (1.9%) | 61,345 (35.1%)<br>4,915 (2.8%) | 116,721 (31.5%)<br>7,370 (2.0%) | 92,369 (35.1%)<br>7,882 (3.0%) | -0.01<br>-0.01 |
| ACS/unstable angina; n (%) Old MI; n (%) | 996 (2.1%)<br>2,154 (4.6%) | 1,826 (3.5%)<br>3,103 (6.0%) | 1,029 (2.2%)<br>1,390 (3.0%) | 1,272 (3.5%)<br>1,228 (3.3%) | 5,178 (1.9%)<br>12,481 (4.5%) | 5,389 (3.1%)<br>9,804 (5.6%) | 7,203 (1.9%)<br>16,025 (4.3%) | 8,487 (3.2%)<br>14,135 (5.4%) | -0.01<br>0.00 |
| Stable angina; n (%) | 1,906 (4.1%) | 3,373 (6.5%) | 1,430 (3.0%) | 1,709 (4.7%) | 7,700 (2.8%) | 7,862 (4.5%) | 11,036 (3.0%) | 12,944 (4.9%) | -0.01 |
| Coronary atherosclerosis and other forms of chronic<br>ischemic heart disease; n (%) | 14,190 (30.5%) | 16,844 (32.6%) | 14,344 (30.5%) | 10,912 (29.7%) | 80,277 (29.0%) | 55,930 (32.0%) | 108,811 (29.3%) | 83,686 (31.8%) | 0.00 |
| Other atherosclerosis with ICD10 v2 Copy; n (%) Previous cardiac procedure (CABG or PTCA or Stent) | 640 (1.4%) | 482 (0.9%) | 767 (1.6%) | 353 (1.0%) | 3,716 (1.3%) | 1,837 (1.1%) | 5,123 (1.4%) | 2,672 (1.0%) | 0.00 |
| v4; n (%) History of CABG or PTCA; n (%) | 466 (1.0%)<br>3,408 (7.3%) | 590 (1.1%)<br>5,202 (10.1%) | 582 (1.2%)<br>1,986 (4.2%) | 378 (1.0%)<br>1,679 (4.6%) | 2,737 (1.0%)<br>21,847 (7.9%) | 1,850 (1.1%)<br>17,991 (10.3%) | 3,785 (1.0%)<br>27,241 (7.3%) | 2,818 (1.1%)<br>24,872 (9.4%) | 0.00 |
| Any stroke; n (%) | 3,408 (7.3%)<br>3,889 (8.4%) | 5,202 (10.1%)<br>5,294 (10.2%) | 1,986 (4.2%)<br>4,154 (8.8%) | 1,679 (4.6%)<br>3,107 (8.5%) | 21,847 (7.9%)<br>22,265 (8.0%) | 17,991 (10.3%)<br>16,801 (9.6%) | 27,241 (7.3%)<br>30,308 (8.2%) | 24,872 (9.4%)<br>25,202 (9.6%) | -0.01<br>0.00 |
| Ischemic stroke (w and w/o mention of cerebral infarction); n (%) | 3,868 (8.3%) | 5,274 (10.2%) | 4,139 (8.8%) | 3,089 (8.4%) | 22,171 (8.0%) | 16,733 (9.6%) | 30,178 (8.1%) | 25,096 (9.5%) | 0.00 |
| Hemorrhagic stroke; n (%)<br>TIA: n (%) | 39 (0.1%)<br>1 324 (2.8%) | 43 (0.1%) | 33 (0.1%)<br>1 325 (2.8%) | 29 (0.1%)<br>1.405 (3.8%) | 140 (0.1%)<br>6.957 (2.5%) | 110 (0.1%) | 212 (0.1%)<br>9,606 (2.6%) | 182 (0.1%)<br>10.139 (3.9%) | 0.00 |
| Other cerebrovascular disease; n (%) | 1,133 (2.4%) | 1,895 (3.7%) | 1,082 (2.3%) | 1,018 (2.8%) | 6,167 (2.2%) | 5,465 (3.1%) | 8,382 (2.3%) | 8,378 (3.2%) | -0.01 |
| Late effects of cerebrovascular disease; n (%)<br>Cerebrovascular procedure; n (%) | 1,203 (2.6%)<br>36 (0.1%) | 1,446 (2.8%)<br>74 (0.1%) | 1,059 (2.2%)<br>40 (0.1%) | 660 (1.8%)<br>37 (0.1%) | 6,565 (2.4%)<br>272 (0.1%) | 4,464 (2.6%)<br>239 (0.1%) | 8,827 (2.4%)<br>348 (0.1%) | 6,570 (2.5%)<br>350 (0.1%) | 0.00<br>0.00 |
| Heart failure (CHF); n (%)<br>Peripheral Vascular Disease (PVD) or PVD Surgery v2; | 11,451 (24.6%) | 13,056 (25.3%) | 10,527 (22.4%) | 7,845 (21.4%) | 57,750 (20.8%) | 37,998 (21.7%) | 79,728 (21.5%) | 58,899 (22.4%) | 0.00 |
| n (%) Atrial fibrillation; n (%) | 4,031 (8.7%)<br>44,976 (96.7%) | 4,290 (8.3%)<br>50,504 (97.7%) | 3,753 (8.0%)<br>45,020 (95.6%) | 2,213 (6.0%)<br>36,026 (98.1%) | 22,154 (8.0%)<br>258,810 (93.3%) | 13,347 (7.6%)<br>162,538 (92.9%) | 29,938 (8.1%)<br>348.806 (94.1%) | 19,850 (7.5%)<br>249,068 (94.6%) | 0.00 |
| Other cardiac dysrhythmia; n (%) | 28,564 (61.4%) | 46,297 (89.6%) | 18,736 (39.8%) | 27,343 (74.5%) | 128,350 (46.3%) | 124,814 (71.4%) | 175,650 (47.4%) | 198,454 (75.4%) | -0.04 |
| Cardiac conduction disorders; n (%)<br>Other CVD; n (%) | 3,879 (8.3%)<br>15,662 (33.7%) | 6,455 (12.5%)<br>21,521 (41.6%) | 3,318 (7.0%)<br>15.575 (33.1%) | 3,652 (9.9%)<br>14.236 (38.8%) | 18,316 (6.6%)<br>74,638 (26.9%) | 16,705 (9.6%)<br>58,184 (33.3%) | 25,513 (6.9%)<br>105,875 (28.5%) | 26,812 (10.2%)<br>93,941 (35.7%) | -0.01<br>-0.01 |
| Diabetes-related complications | | | .,,. | , , | | | | | |
| Diabetic retinopathy; n (%) Diabetes with other ophthalmic manifestations; n | 618 (1.3%) | 532 (1.0%) | 530 (1.1%) | 251 (0.7%) | 2,648 (1.0%) | 1,270 (0.7%) | 3,796 (1.0%) | 2,053 (0.8%) | 0.00 |
| (%) Retinal detachment, vitreous hemorrhage, | 70 (0.2%) | 105 (0.2%) | 394 (0.8%) | 152 (0.4%) | 1,768 (0.6%) | 753 (0.4%) | 2,232 (0.6%) | 1,010 (0.4%) | 0.00 |
| vitrectomy; n (%) | 46 (0.1%)<br>36 (0.1%) | 38 (0.1%)<br>42 (0.1%) | 54 (0.1%)<br>55 (0.1%) | 32 (0.1%)<br>21 (0.1%) | 278 (0.1%)<br>331 (0.1%) | 132 (0.1%)<br>169 (0.1%) | 378 (0.1%)<br>#VALUE! | 202 (0.1%)<br>232 (0.1%) | 0.00<br>#VALUE! |
| Retinal laser coagulation therapy; n (%) Occurrence of Diabetic Neuropathy v2 Copy; n (%) | 2,516 (5.4%) | 2,284 (4.4%) | 2,055 (4.4%) | 1,237 (3.4%) | 10,444 (3.8%) | 5,519 (3.2%) | 15,015 (4.0%) | 9,040 (3.4%) | 0.00 |
| Occurrence of diabetic nephropathy V3 with ICD10<br>Copy; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| Hypoglycemia v2; n (%)<br>Hyperglycemia; n (%) | 362 (0.8%)<br>2,214 (4.8%) | 146 (0.3%)<br>3,478 (6.7%) | 523 (1.1%)<br>1,225 (2.6%) | 168 (0.5%)<br>1,520 (4.1%) | 3,539 (1.3%)<br>14,276 (5.1%) | 2,349 (1.3%)<br>12,139 (6.9%) | 4,424 (1.2%)<br>17,715 (4.8%) | 2,663 (1.0%)<br>17,137 (6.5%) | 0.00<br>-0.01 |
| Disorders of fluid electrolyte and acid-base balance; n | 3,947 (8.5%) | 6,950 (13.4%) | 3,246 (6.9%) | 3,753 (10.2%) | 20,433 (7.4%) | | | 20,306 (7.7%) | 0.00 |
| Diabetic ketoacidosis; n (%) | 38 (0.1%) | 27 (0.1%) | 48 (0.1%) | 28 (0.1%) | 266 (0.1%) | 9,603 (5.5%)<br>142 (0.1%) | 27,626 (7.4%)<br>352 (0.1%) | 197 (0.1%) | 0.00 |
| Hyperosmolar hyperglycemic nonketotic syndrome<br>(HONK); n (%) | 42 (0.1%) | 58 (0.1%) | 35 (0.1%) | 31 (0.1%) | 227 (0.1%) | 171 (0.1%) | 304 (0.1%) | 260 (0.1%) | 0.00 |
| Diabetes with peripheral circulatory disorders with ICD-10 v2 Copy; n (%) | 1,168 (2.5%) | 1,166 (2.3%) | 912 (1.9%) | 460 (1.3%) | 7,176 (2.6%) | 3,365 (1.9%) | 9,256 (2.5%) | 4,991 (1.9%) | 0.00 |
| Diabetic Foot; n (%) | 1,114 (2.4%) | 882 (1.7%) | 1,235 (2.6%) | 568 (1.5%) | 8,445 (3.0%) | 3,903 (2.2%) | 10,794 (2.9%) | 5,353 (2.0%) | 0.01 |
| Gangrene v2; n (%)<br>Lower extremity amputation; n (%) | 55 (0.1%)<br>193 (0.4%) | 56 (0.1%)<br>158 (0.3%) | 74 (0.2%)<br>116 (0.2%) | 46 (0.1%)<br>64 (0.2%) | 434 (0.2%)<br>995 (0.4%) | 236 (0.1%)<br>494 (0.3%) | 563 (0.2%)<br>1,304 (0.4%) | 338 (0.1%)<br>716 (0.3%) | 0.00 |
| Osteomyelitis; n (%)<br>Skin infections v2: n (%) | 179 (0.4%)<br>2 805 (6.0%) | 166 (0.3%)<br>2 863 (5.5%) | 211 (0.4%)<br>3.119 (6.6%) | 116 (0.3%)<br>1 972 (5 4%) | 1,256 (0.5%)<br>17.378 (6.3%) | 633 (0.4%)<br>9.518 (5.4%) | 1,646 (0.4%) | 915 (0.3%)<br>14.353 (5.5%) | 0.00 |
| Erectile dysfunction; n (%) Diabetes with unspecified complication; n (%) | 831 (1.8%)<br>558 (1.2%) | 1,104 (2.1%)<br>813 (1.6%) | 743 (1.6%)<br>441 (0.9%) | 766 (2.1%)<br>487 (1.3%) | 1,957 (0.7%)<br>2,180 (0.8%) | 1,418 (0.8%) | 3,531 (1.0%)<br>3,179 (0.9%) | 3,288 (1.2%)<br>2,871 (1.1%) | 0.00 |
| Diabetes mellitus without mention of complications; | | | | | | 1,571 (0.9%) | | | |
| n (%)<br>Hypertension: 1 inpatient or 2 outpatient claims | 12,418 (26.7%) | 11,942 (23.1%) | 12,169 (25.8%) | 8,307 (22.6%) | 72,769 (26.2%) | 39,895 (22.8%) | 97,356 (26.3%) | 60,144 (22.8%) | 0.01 |
| within 365 days; n (%)<br>Hyperlipidemia v2; n (%) | 38,202 (82.1%)<br>26,248 (56.4%) | 44,939 (86.9%)<br>31,513 (61.0%) | 34,957 (74.2%)<br>22,282 (47.3%) | 30,224 (82.3%)<br>20,521 (55.9%) | 240,781 (86.8%)<br>132,828 (47.9%) | 156,352 (89.4%)<br>95,142 (54.4%) | 313,940 (84.7%)<br>181,358 (48.9%) | 231,515 (87.9%)<br>147,176 (55.9%) | 0.00<br>-0.01 |
| Edema; n (%) | 5,070 (10.9%) | 6,386 (12.4%) | 4,232 (9.0%) | 3,436 (9.4%) | 22,434 (8.1%) | 15,113 (8.6%) | 31,736 (8.6%) | 24,935 (9.5%) | 0.00 |
| Renal Dysfunction (non-diabetic) v2; n (%)<br>Occurrence of acute renal disease v2; n (%) | 33 (0.1%)<br>27 (0.1%) | 33 (0.1%)<br>23 (0.0%) | 36 (0.1%)<br>31 (0.1%) | 16 (0.0%)<br>13 (0.0%) | 140 (0.1%)<br>102 (0.0%) | 91 (0.1%)<br>74 (0.0%) | #VALUE! | 140 (0.1%)<br>110 (0.0%) | #VALUE! |
| Occurrence of chronic renal insufficiency; n (%)<br>Chronic kidney disease v2: n (%) | 0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | #VALUE!<br>000 (0.0%) | #VALUE! |
| CKD Stage 3-4; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| Occurrence of hypertensive nephropathy; n (%) Occurrence of miscellaneous renal insufficiency v2; n | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | 000 (0.0%) | #VALUE! |
| (%)<br>Glaucoma or cataracts v2: n (%) | 3 (0.0%)<br>9.485 (20.4%) | 10 (0.0%)<br>10.339 (20.0%) | 9 917 (21 1%) | 6 637 (18 1%) | 28 (0.0%)<br>3,434 (1.2%) | 2.714 (1.6%) | #VALUE!<br>22,836 (6.2%) | #VALUE!<br>19,690 (7.5%) | #VALUE!<br>0.00 |
| Cellulitis or abscess of toe; n (%) | 741 (1.6%)<br>1,122 (2.4%) | 968 (1.9%)<br>873 (1.7%) | 490 (1.0%)<br>1,259 (2.7%) | 504 (1.4%) | #REF! | #REF! | #REF! | #REF! | #REF! |
| Foot ulcer; n (%)<br>Bladder stones; n (%) | 68 (0.1%) | 73 (0.1%) | 50 (0.1%) | 569 (1.5%)<br>55 (0.1%) | 3,748 (1.4%) | 2,644 (1.5%) | 3,866 (1.0%) | 2,772 (1.1%) | 0.00 |
| Kidney stones; n (%)<br>Urinary tract infections (UTIs); n (%) | 610 (1.3%)<br>4,369 (9.4%) | 909 (1.8%)<br>5,714 (11.1%) | 750 (1.6%)<br>3,794 (8.1%) | 703 (1.9%)<br>2,807 (7.6%) | 32,381 (11.7%)<br>92,251 (33.3%) | 22,757 (13.0%)<br>65,655 (37.5%) | 33,741 (9.1%)<br>100,414 (27.1%) | 24,369 (9.3%)<br>74,176 (28.2%) | 0.00<br>0.00 |
| Dipstick urinalysis; n (%)<br>Non-dipstick urinalysis; n (%) | 13,186 (28.3%)<br>5,387 (11.6%) | 17,082 (33.1%)<br>5,784 (11.2%) | 10,409 (22.1%)<br>2,901 (6.2%) | 9,436 (25.7%)<br>2,362 (6.4%) | 30,263 (10.9%)<br>11,517 (4.2%) | 17,838 (10.2%)<br>7,449 (4.3%) | 53,858 (14.5%)<br>19,805 (5.3%) | 44,356 (16.8%)<br>15,595 (5.9%) | -0.01<br>0.00 |
| Urine function test; n (%) | 1,455 (3.1%) | 1,651 (3.2%) | 1,846 (3.9%) | 1,279 (3.5%) | 6,355 (2.3%) | 4,126 (2.4%) | 9,656 (2.6%) | 7,056 (2.7%) | 0.00 |
| Cytology; n (%)<br>Cystoscopy; n (%) | 783 (1.7%)<br>887 (1.9%) | 904 (1.7%)<br>926 (1.8%) | 1,128 (2.4%)<br>1,187 (2.5%) | 750 (2.0%)<br>772 (2.1%) | 6,641 (2.4%)<br>#REF! | 4,090 (2.3%)<br>#REF! | 8,552 (2.3%)<br>#REF! | 5,744 (2.2%)<br>#REF! | 0.00<br>#REF! |
| Other Covariates<br>Liver disease; n (%) | 1,283 (2.8%) | 1,887 (3.7%) | 1,178 (2.5%) | 1.168 (3.2%) | 6,381 (2.3%) | 4,922 (2.8%) | 8,842 (2.4%) | 7,977 (3.0%) | 0.00 |
| Osteoarthritis; n (%) | 1,283 (2.8%)<br>9,198 (19.8%) | 1,887 (3.7%) | 1,178 (2.5%)<br>8,391 (17.8%) | 1,168 (3.2%)<br>6,628 (18.1%) | 54,070 (19.5%) | 4,922 (2.8%)<br>39,271 (22.5%) | 71,659 (19.3%) | 58,183 (22.1%) | -0.01 |
| Other arthritis, arthropathies and musculoskeletal<br>pain; n (%) | 17,803 (38.3%) | 21,436 (41.5%) | 18,046 (38.3%) | 13,933 (38.0%) | 99,452 (35.9%) | 65,655 (37.5%) | 135,301 (36.5%) | 101,024 (38.4%) | 0.00 |
| Dorsopathies; n (%)<br>Fractures; n (%) | 9,910 (21.3%)<br>2,192 (4.7%) | 12,917 (25.0%)<br>2,353 (4.6%) | 9,393 (19.9%)<br>2,232 (4.7%) | 8,215 (22.4%)<br>1,440 (3.9%) | 54,493 (19.7%)<br>13,695 (4.9%) | 38,821 (22.2%)<br>8,779 (5.0%) | 73,796 (19.9%)<br>18,119 (4.9%) | 59,953 (22.8%)<br>12,572 (4.8%) | -0.01<br>0.00 |
| Falls v2; n (%) | 2,600 (5.6%)<br>3.562 (7.7%) | 3,404 (6.6%)<br>4.642 (9.0%) | 1,210 (2.6%)<br>2,679 (5.7%) | 1,061 (2.9%)<br>1,895 (5.2%) | 5,600 (2.0%)<br>23,503 (8.5%) | 4,195 (2.4%)<br>17.259 (9.9%) | 9,410 (2.5%) | 8,660 (3.3%)<br>23,796 (9.0%) | 0.00 |
| Osteoporosis; n (%)<br>Hyperthyroidism; n (%) | 503 (1.1%) | 708 (1.4%) | 390 (0.8%) | 492 (1.3%) | 2,653 (1.0%) | 2,180 (1.2%) | 3,546 (1.0%) | 3,380 (1.3%) | 0.00<br>0.00 |
| Hypothyroidism v2; n (%)<br>Other disorders of thyroid gland V2; n (%) | 7,899 (17.0%)<br>1,449 (3.1%) | 10,367 (20.1%)<br>2,396 (4.6%) | 6,211 (13.2%)<br>1,396 (3.0%) | 5,753 (15.7%)<br>1,570 (4.3%) | 34,405 (12.4%)<br>8,147 (2.9%) | 17,156 (9.8%)<br>6,371 (3.6%) | 48,515 (13.1%)<br>10,992 (3.0%) | 33,276 (12.6%)<br>10,337 (3.9%) | 0.00<br>0.00 |
| Depression; n (%) | 3,549 (7.6%) | 4,771 (9.2%)<br>6,666 (12.9%) | 3,003 (6.4%)<br>2,601 (5.5%) | 2,603 (7.1%) | 20,125 (7.3%) | 14,758 (8.4%) | 26,677 (7.2%) | 22,132 (8.4%)<br>27,007 (10.3%) | 0.00<br>-0.01 |
| Anxiety; n (%)<br>Sleep_Disorder; n (%) | 3,653 (7.9%)<br>4,189 (9.0%) | 2,487 (4.8%) | 5,819 (12.4%) | 3,574 (9.7%)<br>3,549 (9.7%) | 17,650 (6.4%)<br>20,780 (7.5%) | 16,767 (9.6%)<br>9,518 (5.4%) | 30,788 (8.3%) | 15,554 (5.9%) | 0.01 |
| Dementia; n (%)<br>Delirium; n (%) | 2,848 (6.1%)<br>691 (1.5%) | 3,687 (7.1%)<br>1,059 (2.0%) | 2,376 (5.0%)<br>733 (1.6%) | 1,622 (4.4%)<br>532 (1.4%) | 16,857 (6.1%)<br>4,542 (1.6%) | 12,337 (7.1%)<br>3,724 (2.1%) | 22,081 (6.0%)<br>5,966 (1.6%) | 17,646 (6.7%)<br>5,315 (2.0%) | 0.00<br>0.00 |
| Psychosis; n (%)<br>Obesity; n (%) | 481 (1.0%)<br>6,410 (13.8%) | 482 (0.9%)<br>10,641 (20.6%) | 500 (1.1%)<br>4,779 (10.1%) | 235 (0.6%)<br>6,689 (18.2%) | 3,738 (1.3%)<br>30,638 (11.1%) | 2,232 (1.3%)<br>22,749 (13.0%) | 4,719 (1.3%)<br>41,827 (11.3%) | 2,949 (1.1%)<br>40,079 (15.2%) | 0.00 |
| Overweight; n (%) | 1,900 (4.1%) | 4,100 (7.9%) | 813 (1.7%) | 1,462 (4.0%) | 7,636 (2.8%) | 7,748 (4.4%) | 10,349 (2.8%) | 13,310 (5.1%) | -0.01 |
| Smoking; n (%)<br>Alcohol abuse or dependence; n (%) | 6,155 (13.2%)<br>0 (0.0%) | 11,928 (23.1%)<br>0 (0.0%) | 2,707 (5.7%)<br>0 (0.0%) | 3,811 (10.4%)<br>0 (0.0%) | 46,166 (16.7%)<br>0 (0.0%) | 42,054 (24.0%)<br>0 (0.0%) | 55,028 (14.8%)<br>#VALUE! | 57,793 (21.9%)<br>00 (0.0%) | -0.02<br>#VALUE! |
| Drug abuse or dependence; n (%)<br>COPD; n (%) | 0 (0.0%)<br>7,249 (15.6%) | 0 (0.0%)<br>8,641 (16.7%) | 0 (0.0%)<br>5,994 (12.7%) | 0 (0.0%)<br>4,383 (11.9%) | 0 (0.0%)<br>37,766 (13.6%) | 0 (0.0%)<br>26,713 (15.3%) | #VALUE!<br>51,009 (13.8%) | 00 (0.0%)<br>39,737 (15.1%) | #VALUE!<br>0.00 |
| Asthma; n (%) | 2,805 (6.0%) | 4,018 (7.8%) | 2,515 (5.3%) | 2,517 (6.9%) | 15,333 (5.5%) | 12,262 (7.0%) | 20,653 (5.6%) | 18,797 (7.1%) | -0.01 |
| Obstructive sleep apnea; n (%)<br>Pneumonia; n (%) | 5,531 (11.9%)<br>2,506 (5.4%) | 8,010 (15.5%)<br>3,423 (6.6%) | 5,762 (12.2%)<br>2,722 (5.8%) | 6,537 (17.8%)<br>2,155 (5.9%) | 20,547 (7.4%)<br>14,911 (5.4%) | 16,157 (9.2%)<br>11,869 (6.8%) | 31,840 (8.6%)<br>20,139 (5.4%) | 30,704 (11.7%)<br>17,447 (6.6%) | -0.01<br>0.00 |
| Imaging; n (%) Diabetes Medications | 90 (0.2%) | 126 (0.2%) | 91 (0.2%) | 40 (0.1%) | 7,508 (2.7%) | 3,335 (1.9%) | 7,689 (2.1%) | 3501 (1.3%) | 0.01 |
| DM Medications - AGIs; n (%) | 27 (0.1%) | 25 (0.0%) | 37 (0.1%) | 26 (0.1%) | 189 (0.1%) | 96 (0.1%) | 253 (0.1%) | 147 (0.1%) | 0.00 |
| DM Medications - Glitazones; n (%)<br>DM Medications - GLP-1 RA; n (%) | 386 (0.8%)<br>269 (0.6%) | 463 (0.9%)<br>428 (0.8%) | 498 (1.1%)<br>405 (0.9%) | 373 (1.0%)<br>452 (1.2%) | 2,191 (0.8%)<br>1,300 (0.5%) | 1,445 (0.8%)<br>944 (0.5%) | 3,075 (0.8%)<br>1,974 (0.5%) | 2,281 (0.9%)<br>1,824 (0.7%) | 0.00<br>0.00 |
| DM Medications - Insulin; n (%) DM Medications - Meglitinides; n (%) | 1,928 (4.1%)<br>67 (0.1%) | 1,470 (2.8%)<br>58 (0.1%) | 2,484 (5.3%)<br>187 (0.4%) | 1,267 (3.5%)<br>84 (0.2%) | 700 (0.3%)<br>36,304 (13.1%) | 377 (0.2%)<br>21,098 (12.1%) | 5,112 (1.4%)<br>36,558 (9.9%) | 3,114 (1.2%)<br>21,240 (8.1%) | 0.00<br>0.01 |
| DM Medications - Metformin; n (%) Alogliptin; n (%) | 6,525 (14.0%) | 6,660 (12.9%) | 6,133 (13.0%) | 4,912 (13.4%) | 17 (0.0%)<br>0.03 (0.17) | ** | 12,675 (3.4%)<br>#VALUE! | #VALUE! | #VALUE! |
| | - | | | - | 0.03 (0.17) | 0.04 (0.21) | #VALUE! | #VALUE! | #VALUE! |

# Table 1: Unmatched

| Linagliptin; n (%) Savagliptin; n (%) Concomitant initiation or current use of 2nd | 76 (0.2%)<br>130 (0.3%)<br>519 (1.1%) | 128 (0.2%)<br>115 (0.2%)<br>513 (1.0%) | 125 (0.3%)<br>164 (0.3%)<br>1,048 (2.2%) | 106 (0.3%)<br>76 (0.2%)<br>603 (1.6%) | 0.00 (0.00, 0.00)<br>0<br>0.08 (0.40) | 0.00 [0.00, 0.00]<br>0<br>0.10 (0.44) | #VALUE!<br>#VALUE!<br>1,567 (0.4%) | #VALUE!<br>#VALUE!<br>1116 (0.4%) | #VALUE!<br>0.00 |
|---|---|---|---|---|---|---|---|---|---|
| Generation SUs; n (%) Concomitant initiation or current use of AGIs: n (%) | 2,811 (6.0%)<br>22 (0.0%) | 2,013 (3.9%)<br>20 (0.0%) | 2,878 (6.1%)<br>20 (0.0%) | 1,524 (4.2%)<br>20 (0.1%) | 222 (0.1%)<br>85 (0.0%) | 87 (0.0%)<br>59 (0.0%) | 5,911 (1.6%)<br>127 (0.0%) | 3,624 (1.4%)<br>99 (0.0%) | 0.00<br>#DIV/0! |
| Concomitant initiation or current use of Glitazones;<br>n (%) | 296 (0.6%) | 383 (0.7%) | 394 (0.8%) | 295 (0.8%) | 10,008 (3.6%) | 4,508 (2.6%) | 10,698 (2.9%) | 5.186 (2.0%) | 0.01 |
| Concomitant initiation or current use of GLP-1 RA; n | , | | | | | | | .,, | |
| (%) Concomitant initiation or current use of Insulin; n | 175 (0.4%) | 313 (0.6%) | 295 (0.6%) | 325 (0.9%) | 75 (0.0%) | 24 (0.0%) | #VALUE! | #VALUE! | #VALUE! |
| (%) Concomitant initiation or current use of | 1,335 (2.9%) | 1,061 (2.1%) | 1,855 (3.9%) | 943 (2.6%) | 5,097 (1.8%) | 1,483 (0.8%) | 8,287 (2.2%) | 3,487 (1.3%) | 0.01 |
| Meglitinides; n (%)<br>Concomitant initiation or current use of Metformin; | 41 (0.1%) | 46 (0.1%) | 147 (0.3%) | 61 (0.2%) | 0 | 0 | #VALUE! | #VALUE! | #VALUE! |
| n (%) Past use of 2nd Generation SUs Copy; n (%) | 5,447 (11.7%)<br>536 (1.2%) | 5,502 (10.6%)<br>437 (0.8%) | 5,060 (10.7%)<br>638 (1.4%) | 3,953 (10.8%)<br>322 (0.9%) | 0.09 (0.06) | 0.08 (0.06) | 10,507 (2.8%)<br>#VALUE! | 9,455 (3.6%)<br>#VALUE! | 0.00<br>#VALUE! |
| Past use of AGIs Copy; n (%) | ** | ** | 17 (0.0%) | ** | 40 (0 00) | 40 (0.00) | #VALUE! | #VALUE! | #VALUE! |
| Past use of Glitazones Copy; n (%)<br>Past use of GLP-1 RA Copy; n (%) | 90 (0.2%)<br>96 (0.2%) | 80 (0.2%)<br>119 (0.2%) | 104 (0.2%)<br>113 (0.2%) | 78 (0.2%)<br>128 (0.3%) | 40 (0.0%) | 19 (0.0%) | #VALUE! | 177 (0.1%)<br>#VALUE! | #VALUE! |
| Past use of Insulin Copy; n (%) Past use of Meglitinides Copy; n (%) | 593 (1.3%)<br>26 (0.1%) | 410 (0.8%)<br>12 (0.0%) | 630 (1.3%)<br>40 (0.1%) | 324 (0.9%)<br>23 (0.1%) | 42 (0.0%)<br>0 | 21 (0.0%) | 1,265 (0.3%)<br>#VALUE! | 755 (0.3%)<br>#VALUE! | 0.00<br>#VALUE! |
| Past use of metformin (final) Copy; n (%) Other Medications | 1,078 (2.3%) | 1,158 (2.2%) | 1,073 (2.3%) | 959 (2.6%) | 365.00 (0.00) | 365.00 (0.00) | 2,516 (0.7%) | 2,482 (0.9%) | 0.00 |
| Use of ACE inhibitors; n (%) | 16,031 (34.5%) | 16,348 (31.6%) | 15,709 (33.4%) | 11,934 (32.5%)<br>9.485 (25.8%) | 94,664 (34.1%) | 55,262 (31.6%) | 126,404 (34.1%) | 83,544 (31.7%)<br>67 114 (25.5%) | 0.00 |
| Use of Loop Diuretics - United; n (%) | 9,327 (20.1%)<br>13,519 (29.1%) | 12,884 (24.9%)<br>12,517 (24.2%) | 10,532 (22.4%)<br>14,343 (30.5%) | 8,029 (21.9%) | 58,704 (21.2%)<br>88,917 (32.1%) | 44,745 (25.6%)<br>46,134 (26.4%) | 78,563 (21.2%)<br>116,779 (31.5%) | 66,680 (25.3%) | -0.01<br>0.01 |
| Use of other diuretics- United; n (%) Use of nitrates-United; n (%) | 2,991 (6.4%)<br>3,113 (6.7%) | 2,857 (5.5%)<br>3,398 (6.6%) | 3,338 (7.1%)<br>3,604 (7.7%) | 2,090 (5.7%)<br>2,376 (6.5%) | 18,938 (6.8%)<br>23,060 (8.3%) | 9,440 (5.4%)<br>14,532 (8.3%) | 25,267 (6.8%)<br>29,777 (8.0%) | 14,387 (5.5%)<br>20,306 (7.7%) | 0.01<br>0.00 |
| Use of other hypertension drugs; n (%) Use of digoxin- United; n (%) | 3,138 (6.7%)<br>7,261 (15.6%) | 3,262 (6.3%)<br>3,916 (7.6%) | 3,277 (7.0%)<br>8,724 (18.5%) | 2,136 (5.8%)<br>3,451 (9.4%) | 19,290 (7.0%)<br>48,844 (17.6%) | 11,843 (6.8%)<br>17,770 (10.2%) | 25,705 (6.9%)<br>64,829 (17.5%) | 17,241 (6.5%)<br>25,137 (9.5%) | 0.00<br>0.02 |
| Use of Anti-arrhythmics; n (%) | 7,019 (15.1%) | 11,603 (22.4%) | 8,401 (17.8%) | 9,912 (27.0%) | 43,026 (15.5%) | 41,098 (23.5%) | 58,446 (15.8%) | 62,613 (23.8%) | -0.02 |
| Use of COPD/asthma meds- United; n (%) Use of statins; n (%) | 7,511 (16.1%)<br>25,912 (55.7%) | 10,113 (19.6%)<br>28,245 (54.6%) | 8,597 (18.3%)<br>26,335 (55.9%) | 7,219 (19.7%)<br>19,285 (52.5%) | 50,139 (18.1%)<br>156,203 (56.3%) | 36,786 (21.0%)<br>97,740 (55.9%) | 66,247 (17.9%)<br>208,450 (56.2%) | 54,118 (20.6%)<br>145,270 (55.2%) | -0.01<br>0.00 |
| Use of other lipid-lowering drugs; n (%) Use of antiplatelet agents; n (%) | 2,792 (6.0%)<br>3,472 (7.5%) | 2,670 (5.2%)<br>5,766 (11.2%) | 4,079 (8.7%)<br>4,580 (9.7%) | 2,525 (6.9%)<br>4,623 (12.6%) | 19,312 (7.0%)<br>23,628 (8.5%) | 11,011 (6.3%)<br>22,256 (12.7%) | 26,183 (7.1%)<br>31,680 (8.5%) | 16,206 (6.2%)<br>32,645 (12.4%) | 0.00<br>-0.01 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban,<br>Apixaban, Warfarin); n (%) | 46,518 (100.0%) | 51,684 (100.0%) | 47,096 (100.0%) | 36,714 (100.0%) | 277,248 (100.0%) | 174,898 (100.0%) | 370,862 (100.0%) | 263,296 (100.0%) | 0.00 |
| Use of heparin and other low-molecular weight heparins; n (%) | 1.826 (3.9%) | 262 (0.5%) | 17 (0.0%) | 9 (0.0%) | 11.736 (4.2%) | 1.025 (0.6%) | 13.579 (3.7%) | 1.296 (0.5%) | 0.02 |
| Use of NSAIDs; n (%) | 3,545 (7.6%) | 6,273 (12.1%) | 3,897 (8.3%) | 4,968 (13.5%) | 23,704 (8.5%) | 22,086 (12.6%) | 31,146 (8.4%) | 33,327 (12.7%) | -0.01 |
| Use of oral corticosteroids; n (%) Use of bisphosphonate (United); n (%) | 8,410 (18.1%)<br>1,626 (3.5%) | 11,399 (22.1%)<br>1,754 (3.4%) | 8,644 (18.4%)<br>1,385 (2.9%) | 7,663 (20.9%)<br>849 (2.3%) | 55,726 (20.1%)<br>9,601 (3.5%) | 40,611 (23.2%)<br>5,899 (3.4%) | 72,780 (19.6%)<br>12,612 (3.4%) | 59,673 (22.7%)<br>8,502 (3.2%) | -0.01<br>0.00 |
| Use of opioids- United; n (%) Use of antidepressants; n (%) | 11,125 (23.9%)<br>9.146 (19.7%) | 11,856 (22.9%)<br>11,418 (22.1%) | 12,311 (26.1%)<br>8.850 (18.8%) | 8,801 (24.0%)<br>7,378 (20.1%) | 73,353 (26.5%)<br>60.026 (21.7%) | 44,667 (25.5%)<br>40.727 (23.3%) | 96,789 (26.1%)<br>78,022 (21.0%) | 65,324 (24.8%)<br>59,523 (22.6%) | 0.00 |
| Use of antipsychotics; n (%) Use of antipsychotics: n (%) | 720 (1.5%)<br>5,473 (11.8%) | 918 (1.8%)<br>6,369 (12.3%) | 680 (1.4%)<br>4,883 (10.4%) | 531 (1.4%)<br>3,637 (9.9%) | 5,996 (2.2%)<br>34,654 (12.5%) | 4,070 (2.3%)<br>22,276 (12.7%) | 7,396 (2.0%) | 5,519 (2.1%) | 0.00<br>0.00 |
| Use of lithium- United; n (%) | 38 (0.1%) | 38 (0.1%) | 29 (0.1%) | 29 (0.1%) | 200 (0.1%) | 173 (0.1%) | 45,010 (12.1%)<br>267 (0.1%) | 32,282 (12.3%)<br>240 (0.1%) | 0.00 |
| Use of Benzos- United; n (%) Use of anxiolytics/hypnotics- United; n (%) | 5,108 (11.0%)<br>2,139 (4.6%) | 6,832 (13.2%)<br>2,540 (4.9%) | 5,792 (12.3%)<br>2,857 (6.1%) | 4,959 (13.5%)<br>2,470 (6.7%) | 36,471 (13.2%)<br>16,581 (6.0%) | 27,284 (15.6%)<br>11,562 (6.6%) | 47,371 (12.8%)<br>21,577 (5.8%) | 39,075 (14.8%)<br>16,572 (6.3%) | -0.01<br>0.00 |
| Use of dementia meds- United; n (%) Use of antiparkinsonian meds- United; n (%) | 1,633 (3.5%)<br>1,231 (2.6%) | 1,682 (3.3%)<br>1,449 (2.8%) | 1,713 (3.6%)<br>1,232 (2.6%) | 885 (2.4%)<br>836 (2.3%) | 12,226 (4.4%)<br>8,890 (3.2%) | 7,476 (4.3%)<br>5,878 (3.4%) | 15,572 (4.2%)<br>11,353 (3.1%) | 10,043 (3.8%)<br>8,163 (3.1%) | 0.00 |
| Any use of pramlintide; n (%) | ** | ** | 1,232 (2.0%) | 830 (2.376) | ** | ** | #VALUE! | #VALUE! | #VALUE! |
| Any use of 1st generation sulfonylureas; n (%)<br>Entresto (sacubitril/valsartan); n (%) | 0 (0.0%)<br>142 (0.3%) | 0 (0.0%)<br>387 (0.7%) | 51 (0.1%) | 139 (0.4%) | 18 (0.0%)<br>9,353 (3.4%) | 12 (0.0%)<br>6,025 (3.4%) | 9,546 (2.6%) | #VALUE!<br>6,551 (2.5%) | 0.00<br>0.00 |
| Initiation as monotherapy v4 Copy; n (%) Dual therapy with metformin v4 (latest based on | | ** | | ** | 585 (0.2%) | 519 (0.3%) | #VALUE! | #VALUE! | #VALUE! |
| Aetion's suggestion)- not adding to PS; n (%)<br>Labs | 22 (0.0%) | 69 (0.1%) | 29 (0.1%) | 67 (0.2%) | #REF! | #REF! | #REF! 93,614 | #REF!<br>88,398 | #REF! |
| Lab values- HbA1c (%) v3; n (%)<br>Lab values- HbA1c (%) (within 3 months) v3: n (%) | 5,987 (12.9%) | 8,246 (16.0%) | 614 (1.3%) | 450 (1.2%)<br>311 (0.8%) | N/A | N/A | 6,601 (7.1%)<br>4,154 (4.4%) | 8,696 (9.8%)<br>5,415 (6.1%) | -0.01<br>-0.01 |
| Lab values- HbA1c (%) (within 6 months) v3; n (%) | 3,745 (8.1%)<br>5,987 (12.9%) | 5,104 (9.9%)<br>8,246 (16.0%) | 409 (0.9%)<br>614 (1.3%) | 450 (1.2%) | N/A<br>N/A | N/A<br>N/A | 6,601 (7.1%) | 8,696 (9.8%) | -0.01 |
| Lab values- BNP; n (%)<br>Lab values- BNP (within 3 months); n (%) | 745 (1.6%)<br>450 (1.0%) | 999 (1.9%)<br>709 (1.4%) | 67 (0.1%)<br>47 (0.1%) | 52 (0.1%)<br>40 (0.1%) | N/A<br>N/A | N/A<br>N/A | 812 (0.9%)<br>497 (0.5%) | 1,051 (1.2%)<br>749 (0.8%) | 0.00 |
| Lab values- BNP (within 6 months); n (%)<br>Lab values- BUN (mg/dl); n (%) | 745 (1.6%)<br>12,115 (26.0%) | 999 (1.9%)<br>16,732 (32.4%) | 67 (0.1%)<br>734 (1.6%) | 52 (0.1%)<br>690 (1.9%) | N/A<br>N/A | N/A<br>N/A | 812 (0.9%)<br>12,849 (13.7%) | 1,051 (1.2%)<br>17,422 (19.7%) | 0.00<br>-0.01 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) | 7,935 (17.1%) | 11,391 (22.0%) | 495 (1.1%) | 494 (1.3%) | N/A | N/A | 8,430 (9.0%) | 11,885 (13.4%) | -0.01 |
| Lab values- BUN (mg/dl) (within 6 months); n (%)<br>Lab values- Creatinine (mg/dl) v2; n (%) | 12,115 (26.0%)<br>12,356 (26.6%) | 16,732 (32.4%)<br>17,327 (33.5%) | 734 (1.6%)<br>755 (1.6%) | 690 (1.9%)<br>724 (2.0%) | N/A<br>N/A | N/A<br>N/A | 12,849 (13.7%)<br>13,111 (14.0%) | 17,422 (19.7%)<br>18,051 (20.4%) | -0.01<br>-0.02 |
| Lab values- Creatinine (mg/dl) (within 3 months) v2;<br>n (%) | 8,090 (17.4%) | 11,865 (23.0%) | 510 (1.1%) | 511 (1.4%) | N/A | N/A | 8,600 (9.2%) | 12,376 (14.0%) | -0.01 |
| Lab values- Creatinine (mg/dl) (within 6 months) v2;<br>n (%) | 12,356 (26.6%) | 17,327 (33.5%) | 755 (1.6%) | 724 (2.0%) | N/A | N/A | 13,111 (14.0%) | 18,051 (20.4%) | -0.02 |
| Lab values- HDL level (mg/dl); n (%) | 8,381 (18.0%) | 11,485 (22.2%) | 545 (1.2%) | 482 (1.3%) | N/A | N/A | 8,926 (9.5%) | 11,967 (13.5%) | -0.01 |
| Lab values- HDL level (mg/dl) (within 3 months); n (%) | 4,958 (10.7%) | 6,825 (13.2%) | 352 (0.7%) | 313 (0.9%) | N/A | N/A | 5,310 (5.7%) | 7,138 (8.1%) | -0.01 |
| Lab values- HDL level (mg/dl) (within 6 months); n (%)<br>Lab values- LDL level (mg/dl) v2; n (%) | 8,381 (18.0%)<br>8,846 (19.0%) | 11,485 (22.2%)<br>12,078 (23.4%) | 545 (1.2%)<br>636 (1.4%) | 482 (1.3%)<br>481 (1.3%) | N/A | N/A | 8,926 (9.5%)<br>9,482 (10.1%) | 11,967 (13.5%)<br>12,559 (14.2%) | -0.01<br>-0.01 |
| Lab values- LDL level (mg/dl) (within 3 months) v2; n | | | | | N/A | N/A | | | |
| (%)<br>Lab values- LDL level (mg/dl) (within 6 months) v2; n | 5,236 (11.3%) | 7,197 (13.9%) | 412 (0.9%) | 312 (0.8%) | N/A | N/A | 5,648 (6.0%) | 7,509 (8.5%) | -0.01 |
| (%)<br>Lab values- NT-proBNP; n (%) | 8,846 (19.0%)<br>107 (0.2%) | 12,078 (23.4%)<br>230 (0.4%) | 636 (1.4%) | 481 (1.3%) | N/A<br>N/A | N/A<br>N/A | 9,482 (10.1%)<br>#VALUE! | 12,559 (14.2%)<br>#VALUE! | -0.01 |
| Lab values- NT-proBNP (within 3 months); n (%)<br>Lab values- NT-proBNP (within 6 months); n (%) | 77 (0.2%)<br>107 (0.2%) | 174 (0.3%)<br>230 (0.4%) | :: | :: | N/A<br>N/A | N/A<br>N/A | #VALUE! | #VALUE! | - |
| Lab values-Total cholesterol (mg/dl) v2; n (%) | 8,532 (18.3%) | 11,722 (22.7%) | 532 (1.1%) | 483 (1.3%) | N/A | N/A | 9,064 (9.7%) | 12,205 (13.8%) | -0.01 |
| Lab values-Total cholesterol (mg/dl) (within 3 months) v2; n (%) | 5,050 (10.9%) | 6,978 (13.5%) | 340 (0.7%) | 312 (0.8%) | N/A | N/A | 5,390 (5.8%) | 7,290 (8.2%) | -0.01 |
| Lab values- Total cholesterol (mg/dl) (within 6 months) v2; n (%) | 8,532 (18.3%) | 11,722 (22.7%) | 532 (1.1%) | 483 (1.3%) | N/A | N/A | 9,064 (9.7%) | 12,205 (13.8%) | -0.01 |
| Lab values- Triglyceride level (mg/dl); n (%)<br>Lab values- Triglyceride level (mg/dl) (within 3 | 8,377 (18.0%) | 11,624 (22.5%) | 531 (1.1%) | 482 (1.3%) | N/A | N/A | 8,908 (9.5%) | 12,106 (13.7%) | -0.01 |
| months); n (%)<br>Lab values- Triglyceride level (mg/dl) (within 6 | 4,953 (10.6%) | 6,914 (13.4%) | 343 (0.7%) | 311 (0.8%) | N/A | N/A | 5,296 (5.7%) | 7,225 (8.2%) | -0.01 |
| months); n (%)<br>Lab result number-HbA1c (%) mean (only 2 to 20 | 8,377 (18.0%) | 11,624 (22.5%) | 531 (1.1%) | 482 (1.3%) | N/A | N/A | 8,908 (9.5%) | 12,106 (13.7%) | -0.01 |
| included) v4<br>mean (sd) | 6.50 (1.17) | 6.23 (1.06) | 7.03 (1.38) | 6.79 (1.44) | N/A<br>N/A | N/A<br>N/A | 93,614<br>6.77 (1.28) | 88,398<br>6.46 (1.23) | 0.25 |
| median [IQR] | 6.20 [5.80, 6.90] | 6.00 [5.60, 6.60] | 6.68 [6.10, 7.60] | 6.40 [5.90, 7.20] | N/A | N/A | | | 0.23 |
| Missing; n (%)<br>Lab result number-BNP mean v2 | 40,583 (87.2%) | 43,466 (84.1%) | 46,544 (98.8%) | 36,271 (98.8%) | N/A<br>N/A | N/A<br>N/A | 87,127 (93.1%) | 79,737 (90.2%) | |
| mean (sd)<br>median [IQR] | 302.74 (403.46)<br>195.00 [103.08, 347.00] | 318.02 (487.53)<br>193.80 [98.90, 363.00] | 425.66 (678.07)<br>207.00 (80.00, 445.00) | 473.61 (790.82)<br>180.50 (110.50, 418.00) | N/A<br>N/A | N/A<br>N/A | 364.58 (455.54) | 382.64 (631.44) | -0.03 |
| Missing; n (%)<br>Lab result number-BUN (mg/dl) mean v2 | 45,773 (98.4%) | 50,685 (98.1%) | 47,029 (99.9%) | 36,662 (99.9%) | N/A<br>N/A | N/A<br>N/A | | | |
| mean (sd) | 18.61 (6.76) | 17.56 (5.86) | 495.31 (9,425.53) | 829.31 (12,410.83) | N/A | N/A | 258.43 (6685.44) | 354.70 (7998.29) | -0.01 |
| median [IQR]<br>Missing; n (%) | 18.00 [14.00, 21.80]<br>34,403 (74.0%) | 17.00 [14.00, 20.50]<br>34,952 (67.6%) | 18.00 [14.00, 22.00]<br>46,362 (98.4%) | 17.33 [14.00, 21.00]<br>36,024 (98.1%) | N/A<br>N/A | N/A<br>N/A | | | |
| Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included) v3 | | | | | N/A | N/A | | | |
| mean (sd)<br>median (IQR) | 0.99 (0.26)<br>0.96 [0.82, 1.12] | 0.95 (0.23)<br>0.92 [0.79, 1.07] | 1.01 (0.28)<br>0.97 [0.82, 1.14] | 0.97 (0.23)<br>0.95 [0.82, 1.09] | N/A<br>N/A | N/A<br>N/A | 1.00 (0.27) | 0.96 (0.23) | 0.16 |
| Missing; n (%) | 34,278 (73.7%) | 34,562 (66.9%) | 46,368 (98.5%) | 35,998 (98.0%) | N/A | N/A | | | |
| Lab result number-HDL level (mg/dl) mean (only<br>=<\$000 included) v2 | | | | | N/A | N/A | | | |
| mean (sd)<br>median [IQR] | 50.77 (16.18)<br>48.00 (40.00, 59.00) | 53.45 (17.10)<br>51.00 (42.00, 63.00) | 43.18 (16.42)<br>42.00 (34.50, 51.00) | 47.27 (15.00)<br>45.00 (37.00, 54.62) | N/A<br>N/A | N/A<br>N/A | 46.95 (16.30) | 50.88 (16.26) | -0.24 |
| Missing; n (%) Lab result number-LDL level (mg/dl) mean (only | 38,137 (82.0%) | 40,199 (77.8%) | 46,552 (98.8%) | 36,234 (98.7%) | N/A | N/A | | | |
| = <s000 included)="" v2<br="">mean (sd)</s000> | 87.02 (32.99) | 88 96 (33 32) | 84.94 (37.99) | 89 35 (31 51) | N/A<br>N/A | N/A<br>N/A | 85 97 (35 59) | 89.12 (32.58) | -0.09 |
| median [IQR] | 83.00 [65.00, 106.00] | 86.00 [66.00, 108.00] | 83.00 [64.38, 106.00] | 86.00 [67.00, 109.50] | N/A | N/A | 03.37 (33.33) | 03.11 (31.30) | 0.03 |
| Missing; n (%)<br>Lab result number-Total cholesterol (mg/dl) mean | 37,882 (81.4%) | 39,820 (77.0%) | 46,566 (98.9%) | 36,261 (98.8%) | N/A | N/A | | | |
| (only =<5000 included) v2<br>mean (sd) | 165.05 (40.75) | 166.85 (40.46) | 157.07 (50.15) | 164.40 (39.47) | N/A<br>N/A | N/A<br>N/A | 161.04 (45.72) | 165.83 (40.05) | -0.11 |
| median [IQR]<br>Missing; n (%) | | 164.00 [140.00, 191.00]<br>39,972 (77.3%) | | 164.00 [139.00, 189.00]<br>36,233 (98.7%) | N/A<br>N/A | N/A<br>N/A | | | |
| Lab result number-Triglyceride level (mg/dl) mean<br>(only =<5000 included) v2 | | | | | N/A | N/A | | | |
| mean (sd) | 132.42 (81.91)<br>114.00 (83.00, 158.00) | 121.39 (71.34)<br>106.00 [78.00, 145.00] | 143.61 (82.44)<br>129.00 [94.19, 177.00] | 139.76 (74.46)<br>124.00 [90.00, 166.00] | N/A | N/A | 138.05 (82.18) | 129.02 (72.65) | 0.12 |
| median (IQR)<br>Missing; n (%) | 114.00 [83.00, 158.00]<br>38,141 (82.0%) | 106.00 [78.00, 145.00]<br>40,060 (77.5%) | 129.00 [94.19, 177.00]<br>46,566 (98.9%) | 124.00 [90.00, 166.00]<br>36,234 (98.7%) | N/A<br>N/A | N/A<br>N/A | | | |
| Lab result number-Hemoglobin mean (only >0 included) | | | | | N/A | N/A | | | |
| mean (sd)<br>median [IQR] | 13.70 (1.63)<br>13.70 (12.70, 14.80) | 13.68 (1.63)<br>13.70 (12.70, 14.70) | 514.98 (8,374.12)<br>13.50 [12.50, 14.60] | 558.78 (9,177.87)<br>14.00 [12.90, 14.90] | N/A<br>N/A | N/A<br>N/A | 265.89 (5939.68) | 240.07 (5914.77) | 0.00 |
| Missing; n (%) Lab result number-Serum sodium mean (only > 90 | 37,380 (80.4%) | 38,689 (74.9%) | 46,538 (98.8%) | 36,147 (98.5%) | N/A | N/A | | | |
| and < 190 included) | 140.17 (2.93) | 140.38 (2.99) | 139.54 (2.89) | 139.81 (2.47) | N/A<br>N/A | N/A<br>N/A | 420.05.00.00 | 140 4442 | -0.10 |
| mean (sd)<br>median (IQR) | 140.40 [139.00, 142.00] | 141.00 [139.00, 142.00] | 140.00 [138.00, 141.00] | 140.00 [138.00, 141.00] | N/A | N/A | 139.85 (2.91) | 140.14 (2.79) | -0.10 |
| Missing; n (%) Lab result number- Albumin mean (only >0 and <=10 | 34,759 (74.7%) | 35,281 (68.3%) | 46,421 (98.6%) | 36,040 (98.2%) | N/A | N/A | | | |
| included)<br>mean (sd) | 4.14 (0.33) | 4.18 (0.33) | 3.97 (0.82) | 4.17 (0.39) | N/A<br>N/A | N/A<br>N/A | 4.05 (0.63) | 4.18 (0.36) | -0.25 |
| median [IQR] | 4.20 [3.98, 4.35] | 4.20 [4.00, 4.40] | 4.10 [3.80, 4.35] | 4.20 [4.00, 4.40] | N/A | N/A | | | |

# Table 1: Unmatched

| Missing; n (%) Lab result number-Glucose (fasting or random) mean | 36,095 (77.6%) | 37,242 (72.1%) | 46,570 (98.9%) | 36,184 (98.6%) | N/A | N/A | | | |
|---|---|---|---|---|---|---|---|---|---|
| (only 10-1000 included)<br>mean (sd)<br>median [IQR] | 110.98 (35.59)<br>101.00 [92.00, 118.00]<br>34.922 (75.1%) | 108.13 (31.46)<br>100.00 [91.67, 114.00] | 129.63 (47.03)<br>116.50 [97.50, 148.00] | 126.66 (44.91)<br>113.00 [98.00, 140.00] | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | 120.36 (41.74) | 115.83 (37.63) | 0.11 |
| Missing; n (%) Lab result number-Potassium mean (only 1-7 included) | 34,922 (/5.1%) | 35,423 (68.5%) | 46,441 (98.6%) | 36,039 (98.2%) | N/A<br>N/A | N/A<br>N/A | | | |
| mean (sd)<br>median (IQR) | 4.35 (0.43)<br>4.32 [4.10, 4.60] | 4.39 (0.42)<br>4.40 [4.10, 4.65] | 4.34 (0.42)<br>4.30 (4.10, 4.60) | 4.37 (0.42)<br>4.35 [4.10, 4.60] | N/A<br>N/A | N/A<br>N/A | 4.34 (0.43) | 4.38 (0.42) | -0.09 |
| Missing; n (%) Comorbidity Scores | 34,273 (73.7%) | 34,566 (66.9%) | 46,398 (98.5%) | 36,047 (98.2%) | N/A | N/A | | | |
| CCI (180 days)- ICD9 and ICD10 v2<br>mean (sd)<br>median (IQR) | 3.31 (1.80)<br>3.00 [2.00, 4.00] | 3.52 (1.80)<br>3.00 [2.00, 5.00] | 3.03 (1.71)<br>3.00 [2.00, 4.00] | 3.16 (1.63)<br>3.00 [2.00, 4.00] | 2.07 (1.92)<br>2.00 [0.00, 3.00] | 2.18 (2.00)<br>2.00 [1.00, 3.00] | 3.17 (1.76) | 3.37 (1.73) | -0.11 |
| Frailty Score: Qualitative Version 365 days as<br>Categories, v1 | | | | | | | | | |
| 0; n (%)<br>1 to 2; n (%) | 14,245 (30.6%)<br>16,218 (34.9%) | 28,483 (55.1%)<br>16,697 (32.3%) | 4,407 (9.4%)<br>19,921 (42.3%) | 13,475 (36.7%)<br>13,626 (37.1%) | 277,248 (100.0%)<br>0 (0.0%) | 174,898 (100.0%)<br>0 (0.0%) | 295,900 (79.8%)<br>36,139 (9.7%) | 216,856 (82.4%)<br>30,323 (11.5%) | 0.00<br>-0.01 |
| 3 or more; n (%) Frailty Score: Empirical Version 365 days as Categories, v3 | 16,055 (34.5%) | 6,504 (12.6%) | 22,768 (48.3%) | 9,613 (26.2%) | 0 (0.0%) | 0 (0.0%) | 38,823 (10.5%) | 16,117 (6.1%) | 0.02 |
| <0.12908; n (%)<br>0.12908 - 0.1631167; n (%) | 4,465 (9.6%)<br>13,374 (28.8%) | 5,291 (10.2%)<br>14,905 (28.8%) | 4,016 (8.5%)<br>12,576 (26.7%) | 3,794 (10.3%)<br>10,993 (29.9%) | 221,855 (80.0%)<br>23,931 (8.6%) | 143,801 (82.2%)<br>14,240 (8.1%) | 230,336 (62.1%)<br>49,881 (13.5%) | 152,886 (58.1%)<br>40,138 (15.2%) | 0.01<br>0.00 |
| >= 0.1631167; n (%)<br>Non-Frailty; n (%) | 28,679 (61.7%)<br>25,223 (54.2%) | 31,488 (60.9%)<br>29,309 (56.7%) | 30,504 (64.8%)<br>23,478 (49.9%) | 21,927 (59.7%)<br>18,490 (50.4%) | 31,462 (11.3%)<br>5,444 (2.0%) | 16,857 (9.6%)<br>3,205 (1.8%) | 90,645 (24.4%)<br>54,145 (14.6%) | 70,272 (26.7%)<br>51,004 (19.4%) | 0.00<br>-0.01 |
| Frailty Score (mean): Qualitative Version 365 days, v1mean (sd) | 2.12 (2.29) | 0.97 (1.59) | 2.84 (2.14) | 1.65 (1.91) | 51 (0.0%) | 23 (0.0%) | 2.48 (2.22) | 1.25 (1.73) | 0.62 |
| median [IQR]<br>Frailty Score (mean): Empirical Version 365 days, v2 | 2.00 [0.00, 3.00] | 0.00 [0.00, 1.00] | 2.00 [1.00, 4.00] | 1.00 [0.00, 3.00] | | 0 (0.0%) | | | |
| mean (sd)median [IQR] Healthcare Utilization | 0.19 (0.06)<br>0.18 [0.15, 0.21] | 0.19 (0.06)<br>0.17 [0.15, 0.21] | 0.18 (0.06)<br>0.17 [0.15, 0.21] | 0.18 (0.05)<br>0.17 [0.14, 0.20] | 12.09 [7.08, 19.38]<br>#REF! | 10.59 [5.75, 17.41]<br>#REF! | 0.18 (0.06) | 0.19 (0.06) | -0.17 |
| Any hospitalization; n (%) Any hospitalization within prior 30 days; n (%) | 8,809 (18.9%)<br>5,463 (11.7%) | 15,564 (30.1%)<br>9,233 (17.9%) | 11,202 (23.8%)<br>6,631 (14.1%) | 12,977 (35.3%)<br>8,475 (23.1%) | 63,143 (22.8%)<br>36,930 (13.3%) | 60,091 (34.4%)<br>35,816 (20.5%) | 83,154 (22.4%)<br>49,024 (13.2%) | 88,632 (33.7%)<br>53,524 (20.3%) | -0.02<br>-0.02 |
| Any hospitalization during prior 31-180 days; n (%)<br>Endocrinologist Visit; n (%) | 3,995 (8.6%)<br>1,287 (2.8%) | 7,277 (14.1%)<br>1,529 (3.0%) | 5,230 (11.1%)<br>1,484 (3.2%) | 5,135 (14.0%)<br>1,290 (3.5%) | 31,440 (11.3%)<br>10,807 (3.9%) | 29,065 (16.6%)<br>7,100 (4.1%) | 40,665 (11.0%)<br>13,578 (3.7%) | 41,477 (15.8%)<br>9,919 (3.8%) | -0.01<br>0.00 |
| Endocrinologist Visit (30 days prior); n (%) Endocrinologist Visit (31 to 180 days prior); n (%) Internal medicine/family medicine visits; n (%) | 378 (0.8%)<br>1,086 (2.3%)<br>40,302 (86.6%) | 487 (0.9%)<br>1,231 (2.4%)<br>45,027 (87.1%) | 470 (1.0%)<br>1,269 (2.7%)<br>37,673 (80.0%) | 414 (1.1%)<br>1,066 (2.9%)<br>30,010 (81.7%) | 116,999 (42.2%)<br>163,170 (58.9%)<br>228,150 (82.3%) | 106,990 (61.2%)<br>107,358 (61.4%)<br>148,191 (84.7%) | 117,847 (31.8%)<br>165,525 (44.6%)<br>306,125 (82.5%) | 107,891 (41.0%)<br>109,655 (41.6%)<br>223,228 (84.8%) | -0.02<br>0.00<br>0.00 |
| Internal medicine/family medicine visits (30 days<br>prior) v2; n (%) | 25,980 (55.8%) | 27,969 (54.1%) | 22,962 (48.8%) | 18,628 (50.7%) | ** | 140,151 (04.770) | #VALUE! | #VALUE! | #VALUE! |
| Internal medicine/family medicine visits (31 to 180 days prior) v2; n (%) | 37,369 (80.3%) | 40,783 (78.9%) | 34,952 (74.2%) | 26,875 (73.2%) | 0 | 0 | #VALUE! | #VALUE! | #VALUE! |
| Cardiologist visit; n (%) Number of Cardiologist visits (30 days prior); n (%) Number of Cardiologist visits (31 to 180 days prior); | 31,404 (67.5%)<br>18,721 (40.2%) | 43,792 (84.7%)<br>32,136 (62.2%) | 25,898 (55.0%)<br>14,126 (30.0%) | 25,364 (69.1%)<br>19,025 (51.8%) | 199,955 (72.1%)<br>138,538 (50.0%) | 148,611 (85.0%)<br>89,178 (51.0%) | 257,257 (69.4%)<br>171,385 (46.2%) | 217,767 (82.7%)<br>140,339 (53.3%) | -0.02<br>-0.01 |
| n (%)<br>Electrocardiogram v2; n (%) | 25,239 (54.3%)<br>25,997 (55.9%) | 31,683 (61.3%)<br>41,720 (80.7%) | 21,920 (46.5%)<br>26,827 (57.0%) | 18,451 (50.3%)<br>29,235 (79.6%) | 208,192 (75.1%)<br>168,037 (60.6%) | 132,225 (75.6%)<br>145,748 (83.3%) | 255,351 (68.9%)<br>220,861 (59.6%) | 182,359 (69.3%)<br>216,703 (82.3%) | 0.00<br>-0.03 |
| Use of glucose test strips; n (%)<br>Dialysis; n (%) | 423 (0.9%) | 515 (1.0%) | 405 (0.9%)<br>0 (0.0%) | 324 (0.9%)<br>0 (0.0%) | 2,878 (1.0%)<br>#REF! | 1,883 (1.1%)<br>#REF! | 3,706 (1.0%)<br>#VALUE! | 2,722 (1.0%)<br>#VALUE! | 0.00<br>#VALUE! |
| Naive new user v8 Copy; n (%)<br>N antidiabetic drugs at index date v3 Copy<br>mean (sd) | 37,301 (80.2%)<br>0.23 (0.58) | 43,095 (83.4%)<br>0.20 (0.56) | 37,454 (79.5%)<br>0.26 (0.64) | 30,197 (82.2%)<br>0.23 (0.61) | 53,264 (19.2%) | 28,431 (16.3%)<br>0.20 (0.55) | 128,019 (34.5%)<br>0.24 (0.60) | 101,723 (38.6%)<br>0.20 (0.56) | -0.01<br>0.07 |
| median [IQR]<br>number of different/distinct medication | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | | |
| prescriptionsmean (sd)median (IQR) | 8.79 (4.31)<br>8.00 [6.00, 11.00] | 9.43 (4.56)<br>9.00 [6.00, 12.00] | 9.29 (4.50)<br>9.00 [6.00, 12.00] | 9.54 (4.63)<br>9.00 (6.00, 12.00) | 9.19 (4.28)<br>9.00 [6.00, 12.00] | 9.79 (4.53)<br>9.00 [7.00, 12.00] | 9.15 (4.31) | 9.68 (4.55) | -0.12 |
| Number of Hospitalizationsmean (sd) | 0.23 (0.52) | 0.35 (0.60) | 0.27 (0.53) | 0.39 (0.57) | 0.29 (0.61) | 0.43 (0.69) | 0.28 (0.59) | 0.41 (0.66) | -0.21 |
| median (IQR)<br>Number of hospital days | 0.00 (0.00, 0.00) | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | | | |
| mean (sd)median [IQR] Number of Emergency Department (ED) visits v3 | 1.26 (4.08)<br>0.00 [0.00, 0.00] | 1.73 (4.09)<br>0.00 [0.00, 2.00] | 1.58 (4.59)<br>0.00 [0.00, 0.00] | 1.73 (3.80)<br>0.00 (0.00, 3.00) | 1.72 (5.06)<br>0.00 [0.00, 0.00] | 2.25 (5.28)<br>0.00 (0.00, 3.00) | 1.64 (4.89) | 2.08 (4.88) | -0.09 |
| mean (sd)<br>median (IQR) | 0.59 (1.33)<br>0.00 (0.00, 1.00) | 0.88 (1.63)<br>0.00 [0.00, 1.00] | 0.44 (1.86)<br>0.00 [0.00, 0.00] | 0.81 (2.41)<br>0.00 [0.00, 0.00] | 0.76 (1.63)<br>0.00 [0.00, 1.00] | 1.02 (1.82)<br>0.00 [0.00, 2.00] | 0.70 (1.63) | 0.96 (1.88) | -0.15 |
| Number of Office visits<br>mean (sd) | 5.81 (4.53) | 5.95 (4.05) | 6.57 (5.23) | 6.08 (4.28) | 14.12 (13.27) | 14.14 (12.71) | 12.12 (11.73) | 11.41 (10.63) | 0.06 |
| median [IQR] Number of Endocrinologist visitsmean (sd) | 5.00 (3.00, 8.00) | 5.00 [3.00, 8.00] | 5.00 (3.00, 9.00)<br>0.12 (1.03) | 5.00 (3.00, 8.00)<br>0.12 (1.01) | 11.00 [5.00, 19.00]<br>0.17 (1.42) | 11.00 (6.00, 18.00)<br>0.17 (1.44) | 0.15 (1.32) | 0.15 (1.30) | 0.00 |
| median [IQR]<br>Number of internal medicine/family medicine visits | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | | |
| mean (sd)<br>median (IQR) | 10.66 (13.33)<br>7.00 [2.00, 15.00] | 9.59 (12.68)<br>6.00 [2.00, 12.00] | 8.16 (11.92)<br>4.00 [1.00, 11.00] | 7.22 (10.73)<br>4.00 [1.00, 9.00] | 8.63 (10.80)<br>5.00 [1.00, 12.00] | 8.05 (9.86)<br>5.00 (2.00, 11.00) | 8.82 (11.29) | 8.24 (10.59) | 0.05 |
| Number of Cardiologist visitsmean (sd)median [IQR] | 4.51 (6.33)<br>2.00 (0.00, 6.00) | 6.12 (6.43)<br>4.00 (2.00, 9.00) | 3.39 (5.69)<br>1.00 (0.00, 4.00) | 4.21 (5.48)<br>2.00 (0.00, 6.00) | 5.31 (7.47)<br>3.00 (0.00, 7.00) | 6.15 (6.94)<br>4.00 (2.00, 8.00) | 4.97 (7.13) | 5.87 (6.66) | -0.13 |
| Number electrocardiograms received v2<br>mean (sd) | 1.52 (2.38) | 2.68 (2.89) | 1.35 (1.98) | 2.31 (2.43) | 1.59 (2.19) | 2.66 (2.59) | 1.55 (2.19) | 2.62 (2.63) | -0.44 |
| median [IQR] Number of HbA1c tests orderedmean (sd) | 1.00 (0.00, 2.00)<br>0.38 (0.69) | 2.00 [1.00, 4.00]<br>0.39 (0.67) | 1.00 (0.00, 2.00)<br>0.20 (0.53) | 2.00 [1.00, 3.00]<br>0.23 (0.55) | 1.00 [0.00, 2.00]<br>0.38 (0.70) | 2.00 [1.00, 4.00]<br>0.37 (0.68) | 0.36 (0.68) | 0.35 (0.66) | 0.01 |
| median [IQR] Number of glucose tests ordered | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | () | , | |
| mean (sd)<br>median [IQR] | 0.14 (1.31)<br>0.00 [0.00, 0.00] | 0.17 (1.72)<br>0.00 [0.00, 0.00] | 0.12 (0.69)<br>0.00 [0.00, 0.00] | 0.13 (0.75)<br>0.00 [0.00, 0.00] | 0.12 (0.56)<br>0.00 [0.00, 0.00] | 0.12 (0.57)<br>0.00 [0.00, 0.00] | 0.12 (0.71) | 0.13 (0.94) | -0.01 |
| Number of lipid tests orderedmean (sd)median [IQR] | 0.59 (0.81)<br>0.00 (0.00, 1.00) | 0.64 (0.79)<br>0.00 [0.00, 1.00] | 0.31 (0.79)<br>0.00 (0.00, 0.00) | 0.42 (0.91)<br>0.00 [0.00, 1.00] | 0.61 (0.74)<br>0.00 [0.00, 1.00] | 0.66 (0.75)<br>1.00 (0.00, 1.00) | 0.57 (0.76) | 0.62 (0.78) | -0.06 |
| Number of creatinine tests ordered<br>mean (sd) | 0.08 (0.39) | 0.08 (0.36) | 0.07 (0.42) | 0.06 (0.34) | 0.10 (0.43) | 0.10 (0.40) | 0.09 (0.42) | 0.09 (0.38) | 0.00 |
| median [IQR] Number of BUN tests orderedmean (sd) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.05 (0.33) | 0.05 (0.29) | 0.00 |
| median [IQR] Number of tests for microalbuminuria | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | , | 0.03 (0.13) | |
| mean (sd)median (IQR) Total N distinct ICD9/ICD10 diagnoses at the 3rd | 0.19 (0.63)<br>0.00 (0.00, 0.00) | 0.18 (0.60)<br>0.00 [0.00, 0.00] | 0.09 (0.44)<br>0.00 [0.00, 0.00] | 0.10 (0.43)<br>0.00 (0.00, 0.00) | 0.11 (0.40)<br>0.00 [0.00, 0.00] | 0.10 (0.40)<br>0.00 (0.00, 0.00) | 0.12 (0.44) | 0.12 (0.45) | 0.00 |
| digit level Copymean (sd) | 6.46 (8.68) | 11.88 (10.69) | 3.40 (6.52) | 7.07 (8.23) | 6.76 (9.67) | 11.41 (11.56) | 6.30 (9.21) | 10.90 (10.98) | -0.45 |
| median [IQR] For PS | 4.00 [0.00, 10.00] | 10.00 [4.00, 17.00] | 0.00 [0.00, 4.00] | 5.00 (0.00, 11.00) | 3.00 [0.00, 10.00] | 9.00 [1.00, 17.00] | | , , | |
| Hemorrhagic stroke+Other cerebrovascular<br>disease+Cerebrovascular procedure (for PS); n (%) | 1,191 (2.6%) | 1,971 (3.8%) | 1,132 (2.4%) | 1,054 (2.9%) | 267 (0.1%) | 225 (0.1%) | 2,590 (0.7%) | 3,250 (1.2%) | -0.01 |
| Occurrence of creatinine tests ordered (for PS); n (%) Occurrence of BUN tests ordered (for PS); n (%) | 2,569 (5.5%)<br>1,488 (3.2%) | 3,140 (6.1%)<br>1,620 (3.1%) | 2,388 (5.1%)<br>1,449 (3.1%) | 1,798 (4.9%)<br>1,013 (2.8%) | 12,740 (4.6%)<br>0 (0.0%) | 8,116 (4.6%)<br>0 (0.0%) | 17,697 (4.8%)<br>2,937 (0.8%) | 13,054 (5.0%)<br>2,633 (1.0%) | 0.00<br>0.00 |
| Occurrence of chronic renal insufficiency w/o CKD<br>(for PS) v2; n (%)<br>Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%) | 0 (0.0%)<br>2,864 (1.0%) | 0 (0.0%)<br>648 (0.4%) | #VALUE!<br>2,864 (0.8%) | 000 (0.0%)<br>648 (0.2%) | #VALUE!<br>0.01 |
| Chronic kidney disease Stage 3-6 (for PS); n (%) Bladder stones+Kidney stones (for PS); n (%) | 0 (0.0%)<br>653 (1.4%) | 0 (0.0%)<br>948 (1.8%) | 0 (0.0%)<br>778 (1.7%) | 0 (0.0%)<br>734 (2.0%) | 14 (0.0%) | 0 | #VALUE! | #VALUE! | #VALUE! |
| Diabetes with peripheral circulatory<br>disorders+Gangrene+Osteomyelitis(for PS) v3 with | | | | | | | | | |
| ICD10 Copy; n (%)<br>Age decile (for PS) v3<br>Age decile 1 | 1,344 (2.9%)<br>202 (0.4%) | 1,332 (2.6%)<br>393 (0.8%) | 1,122 (2.4%)<br>250 (0.5%) | 592 (1.6%)<br>474 (1.3%) | 14,208 (5.1%)<br>7,714 (2.8%) | 7,605 (4.3%)<br>5,832 (3.3%) | 16,674 (4.5%)<br>8,166 (2.2%) | 9,529 (3.6%)<br>6,699 (2.5%) | 0.00 |
| Age decile 2<br>Age decile 3 | 301 (0.6%)<br>813 (1.7%) | 542 (1.0%)<br>1,242 (2.4%) | 485 (1.0%)<br>550 (1.2%) | 883 (2.4%)<br>880 (2.4%) | 17,543 (6.3%)<br>19,750 (7.1%) | 13,018 (7.4%)<br>13,440 (7.7%) | 18,329 (4.9%)<br>21,113 (5.7%) | 14,443 (5.5%)<br>15,562 (5.9%) | 0.00<br>0.00 |
| Age decile 4<br>Age decile 5 | 863 (1.9%)<br>1,827 (3.9%) | 1,362 (2.6%)<br>2,518 (4.9%) | 916 (1.9%)<br>1,559 (3.3%) | 1,461 (4.0%)<br>2,262 (6.2%) | 21,587 (7.8%)<br>25,288 (9.1%) | 14,984 (8.6%)<br>17,244 (9.9%) | 23,366 (6.3%) 28,674 (7.7%) | 17,807 (6.8%)<br>22,024 (8.4%) | 0.00<br>0.00 |
| Age decile 6<br>Age decile 7<br>Age decile 8 | 2,950 (6.3%)<br>3,901 (8.4%)<br>6,512 (14.0%) | 3,782 (7.3%)<br>4,928 (9.5%)<br>7,553 (14.6%) | 1,531 (3.3%)<br>2,859 (6.1%)<br>3,394 (7.2%) | 2,003 (5.5%)<br>3,929 (10.7%)<br>3,911 (10.7%) | 37,490 (13.5%)<br>46,637 (16.8%)<br>73,124 (26.4%) | 23,478 (13.4%)<br>27,456 (15.7%)<br>41,582 (23.8%) | 41,971 (11.3%)<br>53,397 (14.4%)<br>83,030 (22.4%) | 29,263 (11.1%)<br>36,313 (13.8%)<br>53,046 (20.1%) | 0.00<br>0.00<br>0.00 |
| Age decile 9<br>Age decile 10 | 9,581 (20.6%)<br>19,568 (42.1%) | 10,918 (21.1%)<br>18,446 (35.7%) | 7,111 (15.1%)<br>28,441 (60.4%) | 5,307 (14.5%)<br>15,604 (42.5%) | 0 (0.0%)<br>2,335 (0.8%) | 0 (0.0%)<br>1,031 (0.6%) | 16,692 (4.5%)<br>50,344 (13.6%) | 16,225 (6.2%)<br>35,081 (13.3%) | -0.01<br>0.00 |
| Alcohol abuse or dependence+Drug abuse or<br>dependence (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 86,677 (31.3%) | 67,711 (38.7%) | 86,677 (23.4%) | 67,711 (25.7%) | 0.00 |
| Diabetes with other ophthalmic<br>manifestations+Retinal detachment, vitreous<br>hemorrhage, vitrectomy+Retinal laser coagulation | | | | | | | | | |
| therapy (for PS); n (%) Other atherosclerosis+Cardiac conduction disorders+Other CVD (for PS) v2 Copy; n (%) | 151 (0.3%)<br>17,838 (38.3%) | 183 (0.4%)<br>24,593 (47.6%) | 485 (1.0%)<br>17,553 (37.3%) | 200 (0.5%) | 22,946 (8.3%)<br>39,765 (14.3%) | 18,676 (10.7%)<br>20,259 (11.6%) | 23,582 (6.4%)<br>75.156 (20.3%) | 19,059 (7.2%)<br>60,976 (23.2%) | 0.00 |
| Previous cardiac procedure (CABG or PTCA or Stent) +<br>History of CABG or PTCA (for PS) v3; n (%) | 17,838 (38.3%)<br>3,573 (7.7%) | 24,593 (47.6%)<br>5,383 (10.4%) | 17,553 (37.3%)<br>2,289 (4.9%) | 1,844 (5.0%) | 39,765 (14.3%)<br>7,438 (2.7%) | 20,259 (11.6%)<br>5,427 (3.1%) | 13,300 (3.6%) | 12,654 (4.8%) | -0.01 |
| Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland (for PS); n (%) | 9,026 (19.4%) | 11,941 (23.1%) | 7,281 (15.5%) | 6,829 (18.6%) | 700 (0.3%) | 377 (0.2%) | 17,007 (4.6%) | 19,147 (7.3%) | -0.01<br>0.00 |
| Delirium + Psychosis (for PS); n (%)<br>Any use of Meglitinides (for PS); n (%)<br>Any use of AGIs (for PS); n (%) | 1,077 (2.3%)<br>67 (0.1%)<br>27 (0.1%) | 1,426 (2.8%)<br>58 (0.1%)<br>25 (0.0%) | 1,097 (2.3%)<br>187 (0.4%)<br>37 (0.1%) | 716 (2.0%)<br>84 (0.2%)<br>26 (0.1%) | 189 (0.1%)<br>59,061 (21.3%)<br>732 (0.3%) | 96 (0.1%)<br>37,917 (21.7%)<br>454 (0.3%) | 2,363 (0.6%)<br>59,315 (16.0%)<br>796 (0.2%) | 2,238 (0.8%)<br>38,059 (14.5%)<br>505 (0.2%) | 0.00<br>0.00<br>0.00 |
| CKD stage 3-6 + dialysis (for PS); n (%) | ** | ** | 0 (0.0%) | 0 (0.0%) | 32,383 (11.7%) | 21,697 (12.4%) | #VALUE! | #VALUE! | #VALUE! |

# Table 1: Matched

| Variable Number of patients Agemean (sd) | | | | PS-matched | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Age | Optun<br>Reference - Warfarin | Apixaban (any dose) | Truve<br>Reference - Warfarin | en<br>Apixaban (any dose) | Medio<br>Reference - Warfarin | are<br>Apixaban (any dose) | Exposure - DPP4i | POOLED<br>Exposure - DPP4i | St. Diff. |
| | 15273 | 15273 | 14849 | 14849 | 80137 | 80137 | 110,259 | 110,259 | |
| median [IQR] | 74.79 (8.86)<br>76.00 [70.00, 82.00] | 74.64 (9.26)<br>76.00 (69.00, 82.00) | 72.66 (11.86)<br>74.00 [63.00, 82.00] | 72.78 (11.72)<br>74.00 [64.00, 82.00] | 77.10 (8.28)<br>77.00 [71.00, 83.00] | 77.01 (8.32)<br>77.00 [71.00, 83.00] | 76.18 (8.92) | 76.11 (8.98) | 0.01 |
| Age categories without zero category | | | | | | | | | |
| 18 - 54; n (%)<br>55 - 64; n (%) | 412 (2.7%)<br>1,359 (8.9%) | 489 (3.2%)<br>1,466 (9.6%) | 1,005 (6.8%)<br>3,129 (21.1%) | 900 (6.1%)<br>3,175 (21.4%) | 736 (0.9%)<br>2,397 (3.0%) | 812 (1.0%)<br>2,427 (3.0%) | 2,153 (2.0%)<br>6,885 (6.2%) | 2,201 (2.0%)<br>7,068 (6.4%) | 0.00 |
| 65 - 74; n (%)<br>>=75; n (%) | 4,944 (32.4%)<br>8,558 (56.0%) | 4,931 (32.3%)<br>8,387 (54.9%) | 3,428 (23.1%)<br>7,287 (49.1%) | 3,533 (23.8%)<br>7,241 (48.8%) | 27,342 (34.1%)<br>49,662 (62.0%) | 27,427 (34.2%)<br>49,471 (61.7%) | 35,714 (32.4%)<br>65,507 (59.4%) | 35,891 (32.6%)<br>65,099 (59.0%) | 0.00 |
| Gender without zero category- United<br>Males; n (%) | 7,950 (52.1%) | 7,963 (52.1%) | 8,187 (55.1%) | 8,226 (55.4%) | 36,474 (45.5%) | 36,464 (45.5%) | 52,611 (47.7%) | 52,653 (47.8%) | 0.00 |
| Females; n (%) Race without zero category | 7,323 (47.9%) | 7,310 (47.9%) | 6,662 (44.9%) | 6,623 (44.6%) | 43,663 (54.5%) | 43,673 (54.5%) | 57,648 (52.3%) | 57,606 (52.2%) | 0.00 |
| White; n (%) | N/A | N/A | N/A | N/A | 74,275 (92.7%) | 74,299 (92.7%) | 74,275 (92.7%) | 74,299 (92.7%) | #REF! |
| Black; n (%)<br>Asian; n (%) | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | 2,826 (3.5%)<br>788 (1.0%) | 2,833 (3.5%)<br>762 (1.0%) | 2,826 (3.5%)<br>788 (1.0%) | 2,833 (3.5%)<br>762 (1.0%) | 0.00 |
| Hispanic; n (%)<br>North American Native; n (%) | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | N/A<br>N/A | 723 (0.9%)<br>253 (0.3%) | 776 (1.0%)<br>238 (0.3%) | 723 (0.9%)<br>253 (0.3%) | 776 (1.0%)<br>238 (0.3%) | 0.00 |
| Other/Unknown; n (%) Region without zero category-United v3 (lumping | N/A | N/A | N/A | N/A | 1,272 (1.6%) | 1,229 (1.5%) | 1,272 (1.6%) | 1,229 (1.5%) | 0.00 |
| missing&other category with West) | | | | | | _ | | | |
| Northeast; n (%)<br>South; n (%) | 2,074 (13.6%)<br>5,550 (36.3%) | 2,058 (13.5%)<br>5,501 (36.0%) | 3,638 (24.5%)<br>4,451 (30.0%) | 3,629 (24.4%)<br>4,448 (30.0%) | 15,635 (19.5%)<br>30,844 (38.5%) | 15,661 (19.5%)<br>30,914 (38.6%) | 21,347 (19.4%)<br>40,845 (37.0%) | 21,348 (19.4%)<br>40,863 (37.1%) | 0.00 |
| Midwest; n (%)<br>West; n (%) | 3,239 (21.2%)<br>4,410 (28.9%) | 3,229 (21.1%)<br>4,485 (29.4%) | 4,806 (32.4%)<br>1,883 (12.7%) | 4,766 (32.1%)<br>1,933 (13.0%) | 19,892 (24.8%)<br>13,766 (17.2%) | 20,032 (25.0%)<br>13,530 (16.9%) | 27,937 (25.3%)<br>20,059 (18.2%) | 28,027 (25.4%)<br>19,948 (18.1%) | 0.00 |
| Unknown+missing; n (%)<br>Calendar Time by day (March 29, 2013 to CED) | N/A | N/A | 71 (0.5%) | 73 (0.5%) | N/A | N/A | 71 (0.5%) | 73 (0.5%) | 0.00 |
| mean (sd) | 1,346.50 (640.11) | 1,295.54 (647.77) | 850.64 (519.69) | 831.37 (525.46) | 365.00 (0.00) | 365.00 (0.00) | 566.36 (305.17) | 556.71 (308.71) | 0.03 |
| median [IQR] | 376.00 [837.00, 1,868.50] 30 | 8.00 [758.00, 1,820.00] 7 | 84.00 [436.00, 1,218.00] 7 | 53.00 [410.00, 1,197.00] | 365.00 [365.00, 365.00] | 365.00 [365.00, 365.00] | | | |
| CV Covariates<br>Ischemic heart disease; n (%) | 5,440 (35.6%) | 5,555 (36.4%) | 5,202 (35.0%) | 5,293 (35.6%) | 27,989 (34.9%) | 28,209 (35.2%) | 38,631 (35.0%) | 39,057 (35.4%) | 0.00 |
| Acute MI; n (%)<br>ACS/unstable angina; n (%) | 525 (3.4%)<br>486 (3.2%) | 542 (3.5%)<br>497 (3.3%) | 510 (3.4%)<br>490 (3.3%) | 494 (3.3%)<br>475 (3.2%) | 2,314 (2.9%)<br>2,388 (3.0%) | 2,362 (2.9%)<br>2,389 (3.0%) | 3,349 (3.0%)<br>3,364 (3.1%) | 3,398 (3.1%)<br>3,361 (3.0%) | 0.00 |
| Old MI; n (%) | 875 (5.7%) | 830 (5.4%) | 522 (3.5%) | 532 (3.6%) | 4,574 (5.7%) | 4,707 (5.9%) | 5,971 (5.4%)<br>4,749 (4.3%) | 6,069 (5.5%)<br>4,783 (4.3%) | 0.00 |
| Stable angina; n (%)<br>Coronary atherosclerosis and other forms of chronic | 863 (5.7%) | 855 (5.6%) | 624 (4.2%) | 593 (4.0%) | 3,262 (4.1%) | 3,335 (4.2%) | | | |
| ischemic heart disease; n (%)<br>Other atherosclerosis with ICD10 v2 Copy; n (%) | 4,999 (32.7%)<br>201 (1.3%) | 4,972 (32.6%)<br>164 (1.1%) | 4,830 (32.5%)<br>198 (1.3%) | 4,809 (32.4%)<br>197 (1.3%) | 25,708 (32.1%)<br>984 (1.2%) | 25,961 (32.4%)<br>977 (1.2%) | 35,537 (32.2%)<br>1,383 (1.3%) | 35,742 (32.4%)<br>1,338 (1.2%) | 0.00 |
| Previous cardiac procedure (CABG or PTCA or Stent) v4; n (%) | 280 (1.8%) | 137 (0.9%) | 316 (2.1%) | 171 (1.2%) | 1,502 (1.9%) | 818 (1.0%) | 2,098 (1.9%) | 1,126 (1.0%) | 0.01 |
| History of CABG or PTCA; n (%)<br>Any stroke: n (%) | 1,401 (9.2%)<br>1,429 (9.4%) | 1,435 (9.4%) | 718 (4.8%)<br>1.356 (9.1%) | 802 (5.4%)<br>1,370 (9.2%) | 8,095 (10.1%)<br>7,131 (8.9%) | 8,580 (10.7%)<br>7,238 (9.0%) | 10,214 (9.3%)<br>9,916 (9.0%) | 10,817 (9.8%) | 0.00 |
| Ischemic stroke (w and w/o mention of cerebral | | | ,, | 1,365 (9.2%) | 7,131 (8.9%) | | 9,860 (8.9%) | 9,983 (9.1%) | 0.00 |
| infarction); n (%)<br>Hemorrhagic stroke; n (%) | 1,416 (9.3%)<br>21 (0.1%) | 1,418 (9.3%) | 1,352 (9.1%)<br>11 (0.1%) | 13 (0.1%) | 59 (0.1%) | 7,200 (9.0%)<br>62 (0.1%) | 091 (0.1%) | #VALUE! | #VALUE! |
| TIA; n (%)<br>Other cerebrovascular disease; n (%) | 561 (3.7%)<br>471 (3.1%) | 562 (3.7%)<br>470 (3.1%) | 514 (3.5%)<br>409 (2.8%) | 510 (3.4%)<br>409 (2.8%) | 2,620 (3.3%)<br>2,303 (2.9%) | 2,699 (3.4%)<br>2,287 (2.9%) | 3,695 (3.4%)<br>3,183 (2.9%) | 3,771 (3.4%)<br>3,166 (2.9%) | 0.00<br>0.00 |
| Late effects of cerebrovascular disease; n (%)<br>Cerebrovascular procedure; n (%) | 433 (2.8%)<br>14 (0.1%) | 425 (2.8%)<br>17 (0.1%) | 321 (2.2%)<br>13 (0.1%) | 335 (2.3%)<br>16 (0.1%) | 2,165 (2.7%)<br>103 (0.1%) | 2,209 (2.8%)<br>99 (0.1%) | 2,919 (2.6%)<br>130 (0.1%) | 2,969 (2.7%)<br>132 (0.1%) | 0.00 |
| Heart failure (CHF); n (%) Peripheral Vascular Disease (PVD) or PVD Surgery v2; | 4,026 (26.4%) | 4,076 (26.7%) | 3,528 (23.8%) | 3,512 (23.7%) | 18,310 (22.8%) | 18,437 (23.0%) | 25,864 (23.5%) | 26,025 (23.6%) | 0.00 |
| n (%) | 1,343 (8.8%) | 1,384 (9.1%) | 1,142 (7.7%) | 1,102 (7.4%) | 6,437 (8.0%) | 6,466 (8.1%) | 8,922 (8.1%) | 8,952 (8.1%) | 0.00 |
| Atrial fibrillation; n (%)<br>Other cardiac dysrhythmia; n (%) | 14,720 (96.4%)<br>11,951 (78.2%) | 14,720 (96.4%)<br>11,531 (75.5%) | 14,428 (97.2%)<br>8,702 (58.6%) | 14,375 (96.8%)<br>8,479 (57.1%) | 74,269 (92.7%)<br>49,385 (61.6%) | 74,268 (92.7%)<br>48,611 (60.7%) | 103,417 (93.8%)<br>70,038 (63.5%) | 103,363 (93.7%)<br>68,621 (62.2%) | 0.00<br>0.00 |
| Cardiac conduction disorders; n (%)<br>Other CVD; n (%) | 1,633 (10.7%)<br>5,937 (38.9%) | 1,697 (11.1%)<br>5,926 (38.8%) | 1,347 (9.1%)<br>5,813 (39.1%) | 1,372 (9.2%)<br>5,710 (38.5%) | 7,098 (8.9%)<br>25,840 (32.2%) | 7,032 (8.8%)<br>25,851 (32.3%) | 10,078 (9.1%)<br>37,590 (34.1%) | 10,101 (9.2%)<br>37,487 (34.0%) | 0.00 |
| Diabetes-related complications | 179 (1.2%) | 165 (1.1%) | | 134 (0.9%) | 686 (0.9%) | | 990 (0.9%) | | 0.00 |
| Diabetic retinopathy; n (%) Diabetes with other ophthalmic manifestations; n | | | 125 (0.8%) | | | 724 (0.9%) | | 1,023 (0.9%) | |
| (%) Retinal detachment, vitreous hemorrhage, | 29 (0.2%) | 25 (0.2%) | 92 (0.6%) | 93 (0.6%) | 420 (0.5%) | 437 (0.5%) | 541 (0.5%) | 555 (0.5%) | 0.00 |
| vitrectomy; n (%)<br>Retinal laser coagulation therapy; n (%) | 15 (0.1%) | 14 (0.1%)<br>12 (0.1%) | 16 (0.1%)<br>13 (0.1%) | 15 (0.1%)<br>12 (0.1%) | 58 (0.1%)<br>85 (0.1%) | 66 (0.1%)<br>90 (0.1%) | 089 (0.1%)<br>#VALUE! | 095 (0.1%)<br>114 (0.1%) | 0.00<br>#VALUE! |
| Occurrence of Diabetic Neuropathy v2 Copy; n (%)<br>Occurrence of diabetic nephropathy V3 with ICD10 | 763 (5.0%) | 784 (5.1%) | 557 (3.8%) | 568 (3.8%) | 2,858 (3.6%) | 2,971 (3.7%) | 4,178 (3.8%) | 4,323 (3.9%) | 0.00 |
| Copy; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Hypoglycemia v2; n (%)<br>Hyperglycemia; n (%) | 76 (0.5%)<br>862 (5.6%) | 80 (0.5%)<br>903 (5.9%) | 128 (0.9%)<br>505 (3.4%) | 103 (0.7%)<br>496 (3.3%) | 1,106 (1.4%)<br>5,184 (6.5%) | 1,103 (1.4%)<br>4,951 (6.2%) | 1,310 (1.2%)<br>6,551 (5.9%) | 1,286 (1.2%)<br>6,350 (5.8%) | 0.00<br>0.00 |
| Disorders of fluid electrolyte and acid-base balance; r<br>(%) | 1,693 (11.1%) | 1,852 (12.1%) | 1,339 (9.0%) | 1,402 (9.4%) | 6,132 (7.7%) | 5,838 (7.3%) | 9,164 (8.3%) | 9,092 (8.2%) | 0.00 |
| Diabetic ketoacidosis; n (%)<br>Hyperosmolar hyperglycemic nonketotic syndrome | | 13 (0.1%) | 14 (0.1%) | 11 (0.1%) | 69 (0.1%) | 80 (0.1%) | #VALUE! | 104 (0.1%) | #VALUE! |
| (HONK); n (%) Diabetes with peripheral circulatory disorders with | 18 (0.1%) | 15 (0.1%) | 16 (0.1%) | ** | 71 (0.1%) | 74 (0.1%) | 105 (0.1%) | #VALUE! | #VALUE! |
| ICD-10 v2 Copy; n (%) | 344 (2.3%) | 356 (2.3%) | 230 (1.5%) | 217 (1.5%) | 1,779 (2.2%) | 1,746 (2.2%) | 2,353 (2.1%) | 2,319 (2.1%) | 0.00 |
| Diabetic Foot; n (%)<br>Gangrene v2; n (%) | 322 (2.1%)<br>17 (0.1%) | 320 (2.1%)<br>19 (0.1%) | 339 (2.3%)<br>24 (0.2%) | 301 (2.0%)<br>25 (0.2%) | 2,082 (2.6%)<br>115 (0.1%) | 2,062 (2.6%)<br>130 (0.2%) | 2,743 (2.5%)<br>156 (0.1%) | 2,683 (2.4%)<br>174 (0.2%) | 0.00<br>0.00 |
| Lower extremity amputation; n (%)<br>Osteomyelitis; n (%) | 66 (0.4%)<br>57 (0.4%) | 49 (0.3%)<br>67 (0.4%) | 30 (0.2%)<br>58 (0.4%) | 36 (0.2%)<br>56 (0.4%) | 274 (0.3%)<br>312 (0.4%) | 275 (0.3%)<br>343 (0.4%) | 370 (0.3%)<br>427 (0.4%) | 360 (0.3%)<br>466 (0.4%) | 0.00 |
| Skin infections v2; n (%)<br>Erectile dysfunction; n (%) | 888 (5.8%)<br>278 (1.8%) | 885 (5.8%)<br>299 (2.0%) | 892 (6.0%)<br>271 (1.8%) | 905 (6.1%)<br>274 (1.8%) | 4,624 (5.8%)<br>632 (0.8%) | 4,625 (5.8%)<br>626 (0.8%) | 6,404 (5.8%)<br>1.181 (1.1%) | 6,415 (5.8%)<br>1.199 (1.1%) | 0.00 |
| Diabetes with unspecified complication; n (%) | 238 (1.6%) | 233 (1.5%) | 182 (1.2%) | 153 (1.0%) | 767 (1.0%) | 712 (0.9%) | 1,187 (1.1%) | 1,098 (1.0%) | 0.00 |
| Diabetes mellitus without mention of complications n (%) | 3,809 (24.9%) | 3,816 (25.0%) | 3,576 (24.1%) | 3,582 (24.1%) | 20,010 (25.0%) | 20,230 (25.2%) | 27,395 (24.8%) | 27,628 (25.1%) | 0.00 |
| Hypertension: 1 inpatient or 2 outpatient claims<br>within 365 days; n (%) | 13,001 (85.1%) | 12,934 (84.7%) | 11,752 (79.1%) | 11,730 (79.0%) | 71,410 (89.1%) | 71,353 (89.0%) | 96,163 (87.2%) | 96,017 (87.1%) | 0.00 |
| Hyperlipidemia v2; n (%)<br>Edema; n (%) | 8,962 (58.7%)<br>1,847 (12.1%) | 9,005 (59.0%)<br>1,843 (12.1%) | 7,798 (52.5%)<br>1,485 (10.0%) | 7,774 (52.4%)<br>1,453 (9.8%) | 41,925 (52.3%)<br>7,070 (8.8%) | 42,279 (52.8%)<br>7,141 (8.9%) | 58,685 (53.2%)<br>10,402 (9.4%) | 59,058 (53.6%)<br>10,437 (9.5%) | 0.00 |
| Renal Dysfunction (non-diabetic) v2; n (%) Occurrence of acute renal disease v2; n (%) | 15 (0.1%)<br>12 (0.1%) | ** | .,, | 12 (0.1%)<br>11 (0.1%) | 55 (0.1%)<br>46 (0.1%) | 49 (0.1%)<br>42 (0.1%) | #VALUE! | #VALUE! | #VALUE! |
| Occurrence of chronic renal insufficiency; n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| Chronic kidney disease v2; n (%)<br>CKD Stage 3-4; n (%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 000 (0.0%)<br>000 (0.0%) | 000 (0.0%)<br>000 (0.0%) | #DIV/0! |
| Occurrence of hypertensive nephropathy; n (%) Occurrence of miscellaneous renal insufficiency v2; n | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/0! |
| (%) Glaucoma or cataracts v2; n (%) | 2.873 (18.8%) | 3.064 (20.1%) | 0 (0.0%)<br>3.051 (20.5%) | 2.941 (19.8%) | 6 (0.0%)<br>16.717 (20.9%) | 6 (0.0%)<br>16.763 (20.9%) | #VALUE!<br>22.641 (20.5%) | #VALUE!<br>22,768 (20.6%) | #VALUE!<br>0.00 |
| Cellulitis or abscess of toe; n (%) | 264 (1.7%) | 293 (1.9%) | 198 (1.3%) | 195 (1.3%) | 1,108 (1.4%) | 1,212 (1.5%) | 1,570 (1.4%) | 1,700 (1.5%) | 0.00 |
| Foot ulcer; n (%)<br>Bladder stones; n (%) | 322 (2.1%)<br>18 (0.1%) | 323 (2.1%)<br>27 (0.2%) | 345 (2.3%)<br>19 (0.1%) | 304 (2.0%)<br>32 (0.2%) | 1,810 (2.3%)<br>79 (0.1%) | 1,795 (2.2%)<br>105 (0.1%) | 2,477 (2.2%)<br>116 (0.1%) | 2,422 (2.2%)<br>164 (0.1%) | 0.00<br>0.00 |
| Kidney stones; n (%)<br>Urinary tract infections (UTIs); n (%) | 222 (1.5%)<br>1,543 (10.1%) | 225 (1.5%)<br>1,671 (10.9%) | 253 (1.7%)<br>1,230 (8.3%) | 275 (1.9%)<br>1,255 (8.5%) | 1,205 (1.5%)<br>10,192 (12.7%) | 1,230 (1.5%)<br>10,461 (13.1%) | 1,680 (1.5%)<br>12,965 (11.8%) | 1,730 (1.6%)<br>13,387 (12.1%) | 0.00 |
| Dipstick urinalysis; n (%) Non-dipstick urinalysis: n (%) | 4,469 (29.3%)<br>1,692 (11.1%) | 4,791 (31.4%)<br>1,664 (10.9%) | 3,305 (22.3%)<br>852 (5.7%) | 3,551 (23.9%)<br>837 (5.6%) | 28,148 (35.1%)<br>8.405 (10.5%) | 29,526 (36.8%)<br>8,371 (10.4%) | 35,922 (32.6%)<br>10,949 (9.9%) | 37,868 (34.3%)<br>10,872 (9.9%) | 0.00 |
| Urine function test; n (%) | 469 (3.1%) | 469 (3.1%) | 599 (4.0%) | 563 (3.8%) | 3,241 (4.0%) | 3,261 (4.1%) | 4,309 (3.9%) | 4,293 (3.9%) | 0.00 |
| Cytology; n (%)<br>Cystoscopy; n (%) | 263 (1.7%)<br>280 (1.8%) | 296 (1.9%)<br>283 (1.9%) | 379 (2.6%)<br>351 (2.4%) | 334 (2.2%)<br>358 (2.4%) | 1,845 (2.3%)<br>1,868 (2.3%) | 1,923 (2.4%)<br>1,863 (2.3%) | 2,487 (2.3%)<br>2,499 (2.3%) | 2,553 (2.3%)<br>2,504 (2.3%) | 0.00<br>0.00 |
| Other Covariates<br>Liver disease; n (%) | 510 (3.3%) | 533 (3.5%) | 472 (3.2%) | 438 (2.9%) | 2,239 (2.8%) | 2,253 (2.8%) | 3,221 (2.9%) | 3,224 (2.9%) | 0.00 |
| Osteoarthritis; n (%) Other arthritis, arthropathies and musculoskeletal | 3,454 (22.6%) | 3,462 (22.7%) | 2,918 (19.7%) | 2,847 (19.2%) | 18,155 (22.7%) | 18,116 (22.6%) | 24,527 (22.2%) | 24,425 (22.2%) | 0.00 |
| pain; n (%) | 6,231 (40.8%) | 6,235 (40.8%) | 5,911 (39.8%) | 5,814 (39.2%) | 30,674 (38.3%) | 30,992 (38.7%) | 42,816 (38.8%) | 43,041 (39.0%) | 0.00 |
| Dorsopathies; n (%)<br>Fractures; n (%) | 3,580 (23.4%)<br>750 (4.9%) | 3,578 (23.4%)<br>760 (5.0%) | 3,184 (21.4%)<br>694 (4.7%) | 3,218 (21.7%)<br>680 (4.6%) | 17,414 (21.7%)<br>4,114 (5.1%) | 17,640 (22.0%)<br>4,059 (5.1%) | 24,178 (21.9%)<br>5,558 (5.0%) | 24,436 (22.2%)<br>5,499 (5.0%) | 0.00<br>0.00 |
| Falls v2; n (%)<br>Osteoporosis; n (%) | 962 (6.3%)<br>1,246 (8.2%) | 954 (6.2%)<br>1,242 (8.1%) | 483 (3.3%)<br>814 (5.5%) | 445 (3.0%)<br>803 (5.4%) | 1,949 (2.4%)<br>7,381 (9.2%) | 1,935 (2.4%)<br>7,387 (9.2%) | 3,394 (3.1%)<br>9,441 (8.6%) | 3,334 (3.0%)<br>9,432 (8.6%) | 0.00 |
| Hyperthyroidism; n (%)<br>Hypothyroidism v2; n (%) | 188 (1.2%)<br>2.823 (18.5%) | 198 (1.3%)<br>2.797 (18.3%) | 141 (0.9%)<br>2.132 (14.4%) | 176 (1.2%)<br>2.237 (15.1%) | 940 (1.2%) | 987 (1.2%) | 1,269 (1.2%)<br>14,267 (12.9%) | 1,361 (1.2%) | 0.00 |
| | 575 (3.8%) | 584 (3.8%) | 537 (3.6%) | 555 (3.7%) | 2,752 (3.4%) | 2,713 (3.4%) | 3,864 (3.5%) | 3,852 (3.5%) | 0.00 |
| Other disorders of thyroid gland V2; n (%) | 1,401 (9.2%)<br>1,672 (10.9%) | 1,452 (9.5%)<br>1,675 (11.0%) | 1,075 (7.2%)<br>1,148 (7.7%) | 1,049 (7.1%)<br>1,100 (7.4%) | 7,087 (8.8%)<br>7,191 (9.0%) | 7,141 (8.9%)<br>7,353 (9.2%) | 9,563 (8.7%)<br>10,011 (9.1%) | 9,642 (8.7%)<br>10,128 (9.2%) | 0.00<br>0.00 |
| Depression; n (%)<br>Anxiety; n (%) | 1,106 (7.2%)<br>1,054 (6.9%) | 1,225 (8.0%)<br>1,079 (7.1%) | 1,780 (12.0%)<br>796 (5.4%) | 1,831 (12.3%)<br>795 (5.4%) | 5,633 (7.0%)<br>5,565 (6.9%) | 5,896 (7.4%)<br>5,591 (7.0%) | 8,519 (7.7%)<br>7,415 (6.7%) | 8,952 (8.1%)<br>7,465 (6.8%) | 0.00 |
| Depression; n (%) | | | 261 (1.8%) | 257 (1.7%)<br>142 (1.0%) | 1,714 (2.1%)<br>1,251 (1.6%) | 1,661 (2.1%)<br>1,230 (1.5%) | 2,280 (2.1%)<br>1,575 (1.4%) | 2,206 (2.0%)<br>1,550 (1.4%) | 0.00 |
| Depression; n (%) Anxiety; n (%) Steep_Disorder; n (%) Dementia; n (%) Delirium; n (%) | 305 (2.0%) | 288 (1.9%)<br>178 (1.2%) | 149 /1 09/1 | | | | | | 0.00 |
| Depression; n (%) Anxiety, n (%) Sitep_ Disorder; n (%) Dementia; n (%) Delirium; n (%) Psychosis; n (%) Obesity, n (%) | 305 (2.0%)<br>176 (1.2%)<br>2,673 (17.5%) | 178 (1.2%)<br>2,688 (17.6%) | 148 (1.0%)<br>1,997 (13.4%) | 2,032 (13.7%) | 10,755 (13.4%) | 11,087 (13.8%) | 15,425 (14.0%) | 15,807 (14.3%) | 0.00 |
| Depression: n (%) Analety: n (%) Sleep, Disorder: n (%) Dementia; n (%) Deminum: n (%) Psychosis; n (%) Overweight: n (%) Overweight: n (%) | 305 (2.0%)<br>176 (1.2%)<br>2,673 (17.5%)<br>826 (5.4%)<br>2,920 (19.1%) | 178 (1.2%)<br>2,688 (17.6%)<br>831 (5.4%)<br>2,909 (19.0%) | 1,997 (13.4%)<br>389 (2.6%)<br>1,271 (8.6%) | 2,032 (13.7%)<br>382 (2.6%)<br>1,276 (8.6%) | 2,929 (3.7%)<br>18,325 (22.9%) | 2,932 (3.7%)<br>18,345 (22.9%) | 15,425 (14.0%)<br>4,144 (3.8%)<br>22,516 (20.4%) | 15,807 (14.3%)<br>4,145 (3.8%)<br>22,530 (20.4%) | 0.00 |
| Depression, n (%) Anniety, n (%) Sleep, Disorder, n (%) Delirium, n (%) Delirium, n (%) Deliry, n (%) Obesity, n (%) Obesity, n (%) Obesity, n (%) Smoking, n (%) Smoking, n (%) | 305 (2.0%)<br>176 (1.2%)<br>2,673 (17.5%)<br>826 (5.4%) | 178 (1.2%)<br>2,688 (17.6%)<br>831 (5.4%) | 1,997 (13.4%)<br>389 (2.6%) | 2,032 (13.7%)<br>382 (2.6%) | 2,929 (3.7%) | 2,932 (3.7%) | 15,425 (14.0%)<br>4,144 (3.8%) | 15,807 (14.3%)<br>4,145 (3.8%) | 0.00 |
| Depression, n (%) Anniety, n (%) Sleep, Disorder, n (%) Delirium, n (%) Delirium, n (%) Delirium, n (%) Desity, n (%) Obesity, n (%) Obesity, n (%) Obesity, n (%) Obesity, n (%) Obesity, n (%) Desity, n (%) Drug abuse of dependence; n (%) COP(9 n (%)) | 305 (2.0%)<br>176 (1.2%)<br>2,673 (17.5%)<br>826 (5.4%)<br>2,920 (19.1%)<br>0 (0.0%)<br>0 (0.0%)<br>2,611 (17.1%) | 178 (1.2%) 2,688 (17.6%) 831 (5.4%) 2,909 (19.0%) 0 (0.0%) 0 (0.0%) 2,687 (17.6%) | 1,997 (13.4%)<br>389 (2.6%)<br>1,271 (8.6%)<br>0 (0.0%)<br>0 (0.0%)<br>1,976 (13.3%) | 2,032 (13.7%)<br>382 (2.6%)<br>1,276 (8.6%)<br>0 (0.0%)<br>0 (0.0%)<br>1,974 (13.3%) | 2,929 (3.7%)<br>18,325 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,587 (15.7%) | 2,932 (3.7%)<br>18,345 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,821 (16.0%) | 15,425 (14.0%)<br>4,144 (3.8%)<br>22,516 (20.4%)<br>000 (0.0%)<br>000 (0.0%)<br>17,174 (15.6%) | 15,807 (14.3%)<br>4,145 (3.8%)<br>22,530 (20.4%)<br>000 (0.0%)<br>000 (0.0%)<br>17,482 (15.9%) | 0.00<br>0.00<br>#DIV/0!<br>#DIV/0!<br>0.00 |
| Depression, n (%) Anniety, n (%) Sleep, Disorder, n (%) Delirium, n (%) Delirium, n (%) Delirium, n (%) Desity, n (%) Obesity, n (%) | 305 (2.0%)<br>176 (1.2%)<br>2,673 (17.5%)<br>826 (5.4%)<br>2,920 (19.1%)<br>0 (0.0%)<br>0 (0.0%)<br>2,611 (17.1%)<br>1,068 (7.0%)<br>2,016 (13.2%) | 178 (1.2%) 2,688 (17.6%) 831 (5.4%) 2,909 (19.0%) 0 (0.0%) 0 (0.0%) 2,687 (17.6%) 1,079 (7.1%) 2,030 (13.3%) | 1,997 (13.4%)<br>389 (2.6%)<br>1,271 (8.6%)<br>0 (0.0%)<br>0 (0.0%)<br>1,976 (13.3%)<br>907 (6.1%)<br>2,129 (14.3%) | 2,032 (13.7%)<br>382 (2.6%)<br>1,276 (8.6%)<br>0 (0.0%)<br>0 (0.0%)<br>1,974 (13.3%)<br>907 (6.1%)<br>2,124 (14.3%) | 2,929 (3.7%)<br>18,325 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,587 (15.7%)<br>5,437 (6.8%)<br>7,215 (9.0%) | 2,932 (3.7%)<br>18,345 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,821 (16.0%)<br>5,528 (6.9%)<br>7,401 (9.2%) | 15,425 (14.0%)<br>4,144 (3.8%)<br>22,516 (20.4%)<br>000 (0.0%)<br>000 (0.0%)<br>17,174 (15.6%)<br>7,412 (6.7%)<br>11,360 (10.3%) | 15,807 (14.3%) 4,145 (3.8%) 22,530 (20.4%) 000 (0.0%) 000 (0.0%) 17,482 (15.9%) 7,514 (6.8%) 11,555 (10.5%) | 0.00<br>0.00<br>#DIV/0!<br>#DIV/0!<br>0.00<br>0.00 |
| Depression, n (%) Anxiety, n (%) Sleep_Disorder, n (%) Sleep_Disorder, n (%) Delirium, n (%) Delirium, n (%) Psychosis, n (%) Obesity, n (%) Obesity, n (%) Smoking, n (%) Alcohol abuse or dependence, n (%) Drug abuse or dependence, n (%) COPD; n (%) | 305 (2.0%)<br>176 (1.2%)<br>2,673 (17.5%)<br>826 (5.4%)<br>2,920 (19.1%)<br>0 (0.0%)<br>0 (0.0%)<br>2,611 (17.1%)<br>1,068 (7.0%) | 178 (1.2%) 2,688 (17.6%) 831 (5.4%) 2,909 (19.0%) 0 (0.0%) 0 (0.0%) 2,687 (17.6%) 1,079 (7.1%) | 1,997 (13.4%)<br>389 (2.6%)<br>1,271 (8.6%)<br>0 (0.0%)<br>0 (0.0%)<br>1,976 (13.3%)<br>907 (6.1%) | 2,032 (13.7%)<br>382 (2.6%)<br>1,276 (8.6%)<br>0 (0.0%)<br>0,00%)<br>1,974 (13.3%)<br>907 (6.1%) | 2,929 (3.7%)<br>18,325 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,587 (15.7%)<br>5,437 (6.8%) | 2,932 (3.7%)<br>18,345 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,821 (16.0%)<br>5,528 (6.9%) | 15,425 (14.0%)<br>4,144 (3.8%)<br>22,516 (20.4%)<br>000 (0.0%)<br>000 (0.0%)<br>17,174 (15.6%)<br>7,412 (6.7%) | 15,807 (14.3%)<br>4,145 (3.8%)<br>22,530 (20.4%)<br>000 (0.0%)<br>000 (0.0%)<br>17,482 (15.9%)<br>7,514 (6.8%) | 0.00<br>0.00<br>#DIV/0!<br>#DIV/0!<br>0.00<br>0.00<br>0.00 |
| Depression, n (%) Anxiety, n (%) Sleep, Disorder, n (%) Sleep, Disorder, n (%) Delirium, n (%) Delirium, n (%) Psychosis, n (%) Obesity, n (%) Obesity, n (%) Smoking, n (%) Smoking, n (%) Obesity, n (%) Imaging, n (%) Imaging, n (%) Imaging, n (%) | 305 (2.0%)<br>176 (1.2%)<br>2,673 (17.5%)<br>826 (5.4%)<br>2,920 (19.1%)<br>0 (0.0%)<br>0 (0.0%)<br>2,611 (17.1%)<br>1,068 (7.0%)<br>2,016 (13.2%)<br>1,033 (6.8%)<br>41 (0.3%) | 178 (1.2%) 2,688 (17.6%) 831 (5.4%) 2,909 (19.0%) 0 (0.0%) 0 (0.0%) 2,687 (17.6%) 1,079 (7.1%) 2,030 (13.3%) 1,038 (6.8%) | 1,997 (13.4%)<br>389 (2.6%)<br>1,271 (8.6%)<br>0 (0.0%)<br>0 (0.0%)<br>1,976 (13.3%)<br>907 (6.1%)<br>2,129 (14.3%)<br>966 (6.5%) | 2,032 (13.7%) 382 (2.6%) 1,276 (8.6%) 0 (0.0%) 0 (0.0%) 1,974 (13.3%) 907 (6.1%) 2,124 (14.3%) 941 (6.3%) 15 (0.1%) | 2,929 (3.7%)<br>18,325 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,587 (15.7%)<br>5,437 (6.8%)<br>7,215 (9.0%)<br>5,444 (6.8%)<br>262 (0.3%) | 2,932 (3.7%)<br>18,345 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,821 (16.0%)<br>5,528 (6.9%)<br>7,401 (9.2%)<br>5,446 (6.8%)<br>231 (0.3%) | 15,425 (14.0%)<br>4,144 (3.8%)<br>22,516 (20.4%)<br>000 (0.0%)<br>000 (0.0%)<br>17,174 (15.6%)<br>7,412 (6.7%)<br>11,360 (10.3%)<br>7,443 (6.8%) | 15,807 (14.3%) 4,145 (3.8%) 22,530 (20.4%) 000 (0.0%) 000 (0.0%) 17,482 (15.9%) 7,514 (6.8%) 11,555 (10.5%) 7,425 (6.7%) | 0.00<br>0.00<br>mDIV/0!<br>0.00<br>0.00<br>0.00<br>0.00 |
| Depression, n (%) Anxiety, n (%) Sleep, Disorder, n (%) Sleep, Disorder, n (%) Delirium, n (%) Delirium, n (%) Delirium, n (%) Psychods, n (%) Obesity, n (%) Imaging, n (%) Disbetes Medications DM Medications—Adis; n (%) MMedications—(%) MMedications—(%) MMedications—(%) | 305 (2.0%) 176 (1.2%) 2,673 (17.5%) 826 (5.4%) 2,920 (19.1%) 0,0.0%) 2,611 (17.1%) 1,068 (7.0%) 2,016 (13.2%) 1,038 (8.7%) 4,10,37% 1,031 (8.5%) 1,10,3 (8.5%) 1,10,3 (8.5%) 1,10,3 (8.5%) | 178 (1.2%) 2,688 (17.6%) 831 (5.4%) 2,909 (19.0%) 0 (0.0%) 0 (0.0%) 2,687 (17.6%) 1,079 (7.1%) 2,030 (13.3%) 1,038 (6.3%) 38 (0.2%) | 1,997 (13.4%) 389 (2.6%) 1,271 (8.6%) 0 (0.0%) 0 (0.0%) 1,976 (13.3%) 907 (6.1%) 924 (13.3%) 966 (6.5%) 35 (0.2%) | 2,032 (13.7%)<br>382 (2.6%)<br>1,276 (8.6%)<br>0 (0.0%)<br>0 (0.0%)<br>1,974 (13.3%)<br>907 (6.14.3%)<br>941 (6.3%)<br>15 (0.1%)<br>18 (0.1%) | 2,929 (3.7%)<br>18,325 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,587 (15.7%)<br>5,437 (6.8%)<br>7,215 (9.0%)<br>5,444 (6.8%)<br>262 (0.3%)<br>47 (0.1%)<br>617 (0.8%) | 2,932 (3.7%) 18,345 (22.9%) 0 (0.0%) 0 (0.0%) 12,821 (16.0%) 5,528 (6.9%) 7,401 (9.2%) 5,446 (6.8%) 231 (0.3%) 51 (0.1%) 740 (0.9%) | 15,425 (14.0 %) 4,144 (3.8 %) 22,516 (20.4 %) 000 (0.0 %) 000 (0.0 %) 17,174 (15.6 %) 7,412 (6.7 %) 11,360 (10.3 %) 7,443 (6.8 %) 338 (0.3 %) #WALUEI 879 (0.8 %) | 15,807 (14.3%) 4,145 (3.8%) 22,530 (20.4%) 000 (0.0%) 000 (0.0%) 7,514 (6.8%) 7,514 (6.8%) 11,555 (10.5%) 7,245 (6.7%) 284 (0.3%) | 0.00<br>0.00<br>#DIV/0!<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.00 |
| Depression, n (%) Anxiety, n (%) Sleep, Disorder, n (%) Sleep, Disorder, n (%) Delirium, n (%) Delirium, n (%) Delirium, n (%) Psykhods; n (%) Obesity, n (%) Obesity, n (%) Obesity, n (%) Smoking, n (%) Actorial abuse are dependence, n (%) COPO; n (%) Organize or dependence, n (%) COPO; n (%) Obstructive depayance, n (%) Destructive | 305 (2.0%) 176 (1.2%) 2,672 (1.7.5%) 826 (5.4%) 2,920 (19.1%) 0 (0.0%) 0 (0.0%) 1,068 (7.0%) 2,016 (13.2%) 1,038 (8.7%) 41 (0.3%) 12 (0.1%) 18 (0.5%) 88 (0.6%) 535 (5.5%) | 178 (1.2%) 2,688 (17.6%) 831 (5.4%) 2,999 (19.0%) 0 (0.0%) 0 (0.0%) 1,079 (7.1%) 1,079 (7.1%) 1,038 (6.5%) 38 (0.2%) | 1,997 (13.4%) 389 (2.6%) 1,271 (8.6%) 0 (0.0%) 0 (0.0%) 1,976 (13.3%) 907 (6.1%) 2,129 (14.3%) 966 (6.5%) 35 (0.2%) ** 145 (1.0%) 142 (1.0%) 550 (4.4%) | 2,032 (13.7%)<br>322 (2.6%)<br>1,276 (8.6%)<br>0 (0.0%)<br>0 (0.0%)<br>1,974 (13.3%)<br>907 (6.1%)<br>2,124 (14.3%)<br>941 (6.3%)<br>15 (0.1%)<br>18 (0.1%)<br>177 (1.2%)<br>164 (1.1%) | 2,929 (3.7%)<br>18,325 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,887 (15.7%)<br>5,437 (6.8%)<br>7,215 (9.0%)<br>5,444 (6.8%)<br>262 (0.3%)<br>47 (0.1%)<br>617 (0.8%)<br>410 (0.5%)<br>2,877 (3.6%) | 2,932 (3.7%)<br>18,345 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>12,821 (16.0%)<br>5,528 (6.9%)<br>5,446 (6.8%)<br>231 (0.3%)<br>540 (0.9%)<br>386 (0.5%)<br>386 (0.5%) | 15,425 (14.0 %) 4,144 (3.8%) 22,516 (20.4%) 000 (0.0%) 000 (0.0%) 17,174 (15.6%) 7,412 (6.7%) 11,360 (10.3%) 38 (0.3%) #VALUE! 879 (0.8%) #VALUE! 4,062 (3.7%) | 15,807 (14.3%) 4,145 (3.8%) 22,530 (20.4%) 000 (0.0%) 000 (0.0%) 17,482 (15.5%) 7,514 (6.8%) 11,555 (10.5%) 7,425 (6.7%) 284 (0.3%) WALUEL 1,083 (1.0%) #VALUEL 3,478 (3.2%) | 0.00 0.00 #DIV/0! #DIV/0! 0.00 0.00 0.00 0.00 #VALUE! 0.00 #VALUE! |
| Depression; n (S) Anxiety; n (S) Sieep_Bisorder; n (S) Sieep_Bisorder; n (S) Delinium; n (S) Psycholog; n (S) Delinium; n (S) Psycholog; n (S) Delinium; n (S) Psycholog; n (S) Delinium; n (S) Psycholog; n (S) Alcohol abuse or dependence; n (S) Alcohol abuse or dependence; n (S) Drug abuse or dependence; n (S) COPD; n (S) Alcohol abuse or dependence; n (S) COPD; n (S) Districtive dependence; n (S) Dobtructive dependence; n (S) Dobtructive dependence; n (S) Dobtructive dependence; n (S) Districtive dependence; n | 305 (2.0%) 176 (1.2%) 2,673 (17.5%) 826 (5.4%) 2,920 (19.1%) 0 (0.0%) 0 (0.0%) 2,511 (17.1%) 1,068 (7.0%) 410 (3.3) 410 (3.3) 12 (0.1%) 117 (0.5%) 88 (0.6%) | 178 (1.2%) 2,688 (17.6%) 831 (5.4%) 2,909 (19.0%) 0 (0.0%) 0 (0.0%) 2,687 (17.6%) 1,079 (7.1%) 2,030 (13.3%) 1,038 (6.5%) 38 (0.2%) | 1,997 (13.4%) 389 (2.6%) 1,271 (8.6%) 0 (0.0%) 0 (0.0%) 1,976 (13.3%) 907 (6.1%) 2,129 (14.3%) 35 (0.2%) 145 (1.0%) | 2,032 (13.7%) 382 (2.6%) 1,276 (8.6%) 0 (0.0%) 0 (0.0%) 1,974 (13.3%) 907 (6.1%) 2,124 (14.3%) 15 (0.1%) 18 (0.1%) 177 (1.2%) 164 (1.1%) | 2,929 (3.7%)<br>18,325 (2.2%)<br>0 (0.0%)<br>0 (0.0%)<br>12,587 (15.7%)<br>5,437 (6.8%)<br>7,215 (9.0%)<br>5,444 (6.8%)<br>262 (0.3%)<br>47 (0.1%)<br>617 (0.8%)<br>410 (0.5%) | 2,932 (3.7%)<br>18,345 (22.9%)<br>0 (0.0%)<br>0 (0.0%)<br>1,2821 (16.0%)<br>5,528 (6.9%)<br>7,401 (9.2%)<br>5,446 (6.8%)<br>231 (0.3%)<br>51 (0.1%)<br>740 (0.9%)<br>386 (0.5%) | 15,425 (14.0%) 4,144 (1.8%) 22,516 (20.4%) 000 (0.0%) 000 (0.0%) 17,174 (15.6%) 11,360 (10.3%) 7,412 (6.7%) 338 (0.3%) #VALUEI 879 (0.8%) #VALUEI | 15,807 (14.3%) 4,145 (3.8%) 22,530 (20.4%) 000 (0.0%) 000 (0.0%) 17,482 (15.9%) 7,514 (6.8%) 11,555 (10.5%) 7,425 (6.7%) 284 (0.3%) #VALUEI 1,083 (1.0%) #VALUEI | 0.00<br>0.00<br>#DIV/0!<br>#DIV/0!<br>0.00<br>0.00<br>0.00<br>0.00<br>#VALUE!<br>0.00 |

# Table 1: Matched

| Linagliptin; n (%) Saxagliptin; n (%) Sitagliptin; n (%) | 32 (0.2%)<br>41 (0.3%)<br>149 (1.0%) | 23 (0.2%)<br>37 (0.2%)<br>158 (1.0%) | 45 (0.3%)<br>49 (0.3%)<br>296 (2.0%) | 51 (0.3%)<br>40 (0.3%)<br>241 (1.6%) | 0.00 (0.00, 0.00)<br>0<br>0.09 (0.42) | 0.00 [0.00, 0.00]<br>0<br>0.09 (0.42) | #VALUE!<br>#VALUE!<br>#VALUE! | #VALUE!<br>#VALUE!<br>399 (0.4%) | #VALUE!<br>#VALUE!<br>#VALUE! |
|---|---|---|---|---|---|---|---|---|---|
| Concomitant initiation or current use of 2nd<br>Generation SUs; n (%) | 801 (5.2%) | 721 (4.7%) | 768 (5.2%) | 753 (5.1%) | 529 (0.7%) | 381 (0.5%) | 2,098 (1.9%) | 1,855 (1.7%) | 0.00 |
| Concomitant initiation or current use of AGIs; n (%)<br>Concomitant initiation or current use of Glitazones;<br>n (%) | 89 (0.6%) | 132 (0.9%) | 115 (0.8%) | 14 (0.1%)<br>140 (0.9%) | 0 (0.0%)<br>43 (0.1%) | 48 (0.1%) | #VALUE!<br>247 (0.2%) | #VALUE!<br>320 (0.3%) | #VALUE! |
| Concomitant initiation or current use of GLP-1 RA; n<br>(%) | 58 (0.4%) | 70 (0.5%) | 101 (0.7%) | 122 (0.8%) | 27 (0.0%) | 17 (0.0%) | 186 (0.2%) | 209 (0.2%) | 0.00 |
| Concomitant initiation or current use of Insulin; n (%) | 370 (2.4%) | 402 (2.6%) | 485 (3.3%) | 483 (3.3%) | 0 | 0 | #VALUE! | #VALUE! | #VALUE! |
| Concomitant initiation or current use of<br>Meglitinides; n (%)<br>Concomitant initiation or current use of Metformin: | 15 (0.1%) | 15 (0.1%) | 39 (0.3%) | 30 (0.2%) | 19 (0.0%) | 16 (0.0%) | 073 (0.1%) | 061 (0.1%) | 0.00 |
| n (%) Past use of 2nd Generation SUs Copy; n (%) | 1,747 (11.4%)<br>167 (1.1%) | 1,811 (11.9%)<br>183 (1.2%) | 1,584 (10.7%)<br>160 (1.1%) | 1,650 (11.1%)<br>165 (1.1%) | 1,019 (1.3%) | 824 (1.0%)<br>12 (0.0%) | 4,350 (3.9%)<br>#VALUE! | 4,285 (3.9%)<br>360 (0.3%) | 0.00<br>#VALUE! |
| Past use of AGIs Copy; n (%) Past use of Glitazones Copy; n (%) | 28 (0.2%) | 34 (0.2%) | 30 (0.2%) | **<br>37 (0.2%) | 0 (0.0%) | 0 (0.0%) | #VALUE! | #VALUE! | #VALUE! |
| Past use of GLP-1 RA Copy; n (%)<br>Past use of Insulin Copy; n (%) | 31 (0.2%)<br>165 (1.1%) | 31 (0.2%)<br>172 (1.1%) | 43 (0.3%)<br>165 (1.1%) | 42 (0.3%)<br>174 (1.2%) | | : | #VALUE! | #VALUE! | #VALUE! |
| Past use of Meglitinides Copy; n (%) Past use of metformin (final) Copy; n (%) | 5 (0.0%)<br>390 (2.6%) | 5 (0.0%)<br>386 (2.5%) | 12 (0.1%)<br>382 (2.6%) | 13 (0.1%)<br>405 (2.7%) | | :- | #VALUE! | #VALUE! | #VALUE! |
| Other Medications Use of ACE inhibitors; n (%) | 5,108 (33.4%) | 5,185 (33.9%) | 4,931 (33.2%) | 4,911 (33.1%) | 26,746 (33.4%)<br>18.865 (23.5%) | 26,769 (33.4%) | 36,785 (33.4%) | 36,865 (33.4%) | 0.00 |
| Use of ARBs; n (%) Use of Loop Diuretics - United; n (%) | 3,359 (22.0%)<br>4,236 (27.7%)<br>910 (6.0%) | 3,277 (21.5%)<br>4,204 (27.5%) | 3,611 (24.3%)<br>4,099 (27.6%)<br>979 (6.6%) | 3,632 (24.5%)<br>3,973 (26.8%)<br>1,026 (6.9%) | 18,865 (23.5%)<br>23,856 (29.8%)<br>4,712 (5.9%) | 18,827 (23.5%)<br>23,618 (29.5%) | 25,835 (23.4%)<br>32,191 (29.2%)<br>6,601 (6.0%) | 25,736 (23.3%)<br>31,795 (28.8%)<br>6,974 (6.3%) | 0.00<br>0.00<br>0.00 |
| Use of other diuretics- United; n (%) Use of nitrates-United; n (%) Use of other hypertension drugs; n (%) | 1,096 (7.2%)<br>987 (6.5%) | 954 (6.2%)<br>1,033 (6.8%)<br>1,075 (7.0%) | 1,163 (7.8%)<br>944 (6.4%) | 1,026 (6.9%)<br>1,081 (7.3%)<br>1,009 (6.8%) | 7,226 (9.0%)<br>5,421 (6.8%) | 4,994 (6.2%)<br>6,925 (8.6%)<br>5,927 (7.4%) | 9,485 (8.6%)<br>7,352 (6.7%) | 9,039 (8.2%)<br>8,011 (7.3%) | 0.00 |
| Use of digoxin- United; n (%) Use of Anti-arrhythmics; n (%) | 1,982 (13.0%)<br>2,830 (18.5%) | 1,340 (8.8%)<br>2,881 (18.9%) | 2,364 (15.9%)<br>3,408 (23.0%) | 1,677 (11.3%)<br>3,334 (22.5%) | 11,421 (14.3%)<br>16,013 (20.0%) | 8,950 (11.2%)<br>16,120 (20.1%) | 15,767 (14.3%)<br>22,251 (20.2%) | 11,967 (10.9%)<br>22,335 (20.3%) | 0.01 |
| Use of COPD/asthma meds- United; n (%) Use of statins; n (%) | 2,680 (17.5%)<br>8,379 (54.9%) | 2,826 (18.5%)<br>8,384 (54.9%) | 2,867 (19.3%)<br>8,068 (54.3%) | 2,911 (19.6%)<br>8,126 (54.7%) | 16,242 (20.3%)<br>44,642 (55.7%) | 16,177 (20.2%)<br>44,673 (55.7%) | 21,789 (19.8%)<br>61,089 (55.4%) | 21,914 (19.9%)<br>61,183 (55.5%) | 0.00<br>0.00 |
| Use of other lipid-lowering drugs; n (%) Use of antiplatelet agents; n (%) | 807 (5.3%)<br>1,518 (9.9%) | 809 (5.3%)<br>1,535 (10.1%) | 1,122 (7.6%)<br>1,870 (12.6%) | 1,135 (7.6%)<br>1,810 (12.2%) | 4,999 (6.2%)<br>9,611 (12.0%) | 5,066 (6.3%)<br>9,781 (12.2%) | 6,928 (6.3%)<br>12,999 (11.8%) | 7,010 (6.4%)<br>13,126 (11.9%) | 0.00<br>0.00 |
| Use of oral anticoagulants (Dabigatran, Rivaroxaban,<br>Apixaban, Warfarin); n (%)<br>Use of heparin and other low-molecular weight | 15,273 (100.0%) | 15,273 (100.0%) | 14,849 (100.0%) | 14,849 (100.0%) | 80,137 (100.0%) | 80,137 (100.0%) | 110,259 (100.0%) | 110,259 (100.0%) | 0.00 |
| heparins; n (%) Use of NSAIDs; n (%) | 201 (1.3%)<br>1,595 (10.4%) | 246 (1.6%)<br>1.554 (10.2%) | 1.662 (11.2%) | 1.661 (11.2%) | 838 (1.0%)<br>9,357 (11.7%) | 1,007 (1.3%)<br>9,421 (11.8%) | #VALUE!<br>12.614 (11.4%) | #VALUE!<br>12.636 (11.5%) | #VALUE!<br>0.00 |
| Use of oral corticosteroids; n (%) Use of bisphosphonate (United); n (%) | 3,107 (20.3%)<br>525 (3.4%) | 3,092 (20.2%)<br>526 (3.4%) | 2,955 (19.9%)<br>365 (2.5%) | 2,974 (20.0%)<br>355 (2.4%) | 17,909 (22.3%)<br>2,725 (3.4%) | 17,955 (22.4%)<br>2,741 (3.4%) | 23,971 (21.7%)<br>3,615 (3.3%) | 24,021 (21.8%) | 0.00 |
| Use of opioids- United; n (%) Use of antidepressants; n (%) | 3,699 (24.2%)<br>3.362 (22.0%) | 3,758 (24.6%)<br>3,379 (22.1%) | 3,918 (26.4%)<br>3.016 (20.3%) | 3,910 (26.3%)<br>3,005 (20.2%) | 21,952 (27.4%)<br>19,019 (23.7%) | 22,299 (27.8%)<br>19,236 (24.0%) | 29,569 (26.8%)<br>25,397 (23.0%) | 29,967 (27.2%)<br>25,620 (23.2%) | 0.00 |
| Use of antipsychotics; n (%) Use of antipsychotics; n (%) | 280 (1.8%)<br>1,932 (12.6%) | 283 (1.9%)<br>1,991 (13.0%) | 244 (1.6%)<br>1,587 (10.7%) | 243 (1.6%)<br>1.608 (10.8%) | 1,983 (2.5%)<br>10,833 (13.5%) | 2,058 (2.6%) | 2,507 (2.3%)<br>14,352 (13.0%) | 2,584 (2.3%)<br>14,589 (13.2%) | 0.00 |
| Use of lithium- United; n (%) Use of Benzos- United; n (%) | 12 (0.1%)<br>1,886 (12.3%) | 13 (0.1%)<br>1,904 (12.5%) | 16 (0.1%)<br>2,009 (13.5%) | 11 (0.1%)<br>1,965 (13.2%) | 59 (0.1%)<br>12,174 (15.2%) | 86 (0.1%)<br>12,263 (15.3%) | 087 (0.1%)<br>16,069 (14.6%) | 110 (0.1%)<br>16,132 (14.6%) | 0.00<br>0.00 |
| Use of anxiolytics/hypnotics-United; n (%) Use of dementia meds-United; n (%) | 699 (4.6%)<br>533 (3.5%) | 770 (5.0%)<br>499 (3.3%) | 952 (6.4%)<br>491 (3.3%) | 962 (6.5%)<br>495 (3.3%) | 5,173 (6.5%)<br>3,443 (4.3%) | 5,258 (6.6%)<br>3,510 (4.4%) | 6,824 (6.2%)<br>4,467 (4.1%) | 6,990 (6.3%)<br>4,504 (4.1%) | 0.00<br>0.00 |
| Use of antiparkinsonian meds- United; n (%)<br>Any use of pramlintide; n (%) | 444 (2.9%)<br>0 (0.0%) | 450 (2.9%)<br>0 (0.0%) | 401 (2.7%) | 389 (2.6%) | 2,817 (3.5%) | 2,844 (3.5%) | 3,662 (3.3%)<br>#VALUE! | 3,683 (3.3%)<br>#VALUE! | 0.00<br>#VALUE! |
| Any use of 1st generation sulfonylureas; n (%)<br>Entresto (sacubitril/valsartan); n (%) | 0 (0.0%)<br>65 (0.4%) | 0 (0.0%)<br>74 (0.5%) | **<br>35 (0.2%) | 20 (0.1%) | 99 (0.1%) | 114 (0.1%) | #VALUE!<br>199 (0.2%) | #VALUE!<br>208 (0.2%) | 0.00<br>0.00 |
| Initiation as monotherapy v4 Copy; n (%) Dual therapy with metformin v4 (latest based on | 0 (0.0%) | 2 (0.0%) | | | ** | ** | #VALUE! | #VALUE! | #VALUE! |
| Aetion's suggestion)- not adding to PS; n (%)<br>Labs | | ** | 13 (0.1%) | 13 (0.1%) | 194 (0.2%) | 203 (0.3%) | #VALUE!<br>30,122 | #VALUE!<br>30,122 | #VALUE! |
| Lab values- HbA1c (%) v3; n (%)<br>Lab values- HbA1c (%) (within 3 months) v3; n (%) | 2,202 (14.4%)<br>1,417 (9.3%) | 2,238 (14.7%)<br>1,436 (9.4%) | 173 (1.2%)<br>111 (0.7%) | 142 (1.0%)<br>97 (0.7%) | N/A<br>N/A | N/A<br>N/A | 2,375 (7.9%)<br>1,528 (5.1%) | 2,380 (7.9%)<br>1,533 (5.1%) | 0.00<br>0.00 |
| Lab values- HbA1c (%) (within 6 months) v3; n (%)<br>Lab values- BNP; n (%) | 2,202 (14.4%)<br>266 (1.7%) | 2,238 (14.7%)<br>324 (2.1%) | 173 (1.2%)<br>37 (0.2%) | 142 (1.0%)<br>22 (0.1%) | N/A<br>N/A | N/A<br>N/A | 2,375 (7.9%)<br>303 (1.0%) | 2,380 (7.9%)<br>346 (1.1%) | 0.00 |
| Lab values- BNP (within 3 months); n (%)<br>Lab values- BNP (within 6 months); n (%)<br>Lab values- BUN (mg/dl); n (%) | 177 (1.2%)<br>266 (1.7%)<br>4,345 (28.4%) | 226 (1.5%)<br>324 (2.1%)<br>4,694 (30.7%) | 27 (0.2%)<br>37 (0.2%)<br>258 (1.7%) | 19 (0.1%)<br>22 (0.1%)<br>231 (1.6%) | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | 204 (0.7%)<br>303 (1.0%)<br>4,603 (15.3%) | 245 (0.8%)<br>346 (1.1%)<br>4,925 (16.4%) | 0.00<br>0.00<br>0.00 |
| Lab values- BUN (mg/dl) (within 3 months); n (%) Lab values- BUN (mg/dl) (within 6 months); n (%) | 2,953 (19.3%)<br>4,345 (28.4%) | 3,245 (21.2%)<br>4,694 (30.7%) | 181 (1.2%)<br>258 (1.7%) | 155 (1.0%)<br>231 (1.6%) | N/A<br>N/A | N/A<br>N/A | 3,134 (10.4%)<br>4,603 (15.3%) | 3,400 (11.3%)<br>4,925 (16.4%) | 0.00 |
| Lab values- Creatinine (mg/dl) v2; n (%) Lab values- Creatinine (mg/dl) (within 3 months) v2; | 4,447 (29.1%) | 4,846 (31.7%) | 273 (1.8%) | 237 (1.6%) | N/A | N/A | 4,720 (15.7%) | 5,083 (16.9%) | 0.00 |
| n (%) Lab values- Creatinine (mg/dl) (within 6 months) v2; | 3,016 (19.7%) | 3,373 (22.1%) | 191 (1.3%) | 157 (1.1%) | N/A | N/A | 3,207 (10.6%) | 3,530 (11.7%) | 0.00 |
| n (%)<br>Lab values- HDL level (mg/dl); n (%) | 4,447 (29.1%)<br>2,935 (19.2%) | 4,846 (31.7%)<br>3,065 (20.1%) | 273 (1.8%)<br>175 (1.2%) | 237 (1.6%)<br>140 (0.9%) | N/A<br>N/A | N/A<br>N/A | 4,720 (15.7%)<br>3,110 (10.3%) | 5,083 (16.9%)<br>3,205 (10.6%) | 0.00 |
| Lab values-HDL level (mg/dl) (within 3 months); n (%) | 1,764 (11.5%) | 1,845 (12.1%) | 99 (0.7%) | 81 (0.5%) | N/A | N/A | 1,863 (6.2%) | 1,926 (6.4%) | 0.00 |
| Lab values-HDL level (mg/dl) (within 6 months); n (%)<br>Lab values-LDL level (mg/dl) v2; n (%) | 2,935 (19.2%)<br>3,142 (20.6%) | 3,065 (20.1%)<br>3,273 (21.4%) | 175 (1.2%)<br>192 (1.3%) | 140 (0.9%)<br>139 (0.9%) | N/A<br>N/A | N/A<br>N/A | 3,110 (10.3%)<br>3,334 (11.1%) | 3,205 (10.6%)<br>3,412 (11.3%) | 0.00 |
| Lab values-LDL level (mg/dl) (within 3 months) v2; n<br>(%) | 1,887 (12.4%) | 1,978 (13.0%) | 192 (1.3%) | 82 (0.6%) | N/A<br>N/A | N/A<br>N/A | 2,001 (6.6%) | 2,060 (6.8%) | 0.00 |
| Lab values- LDL level (mg/dl) (within 6 months) v2; n<br>(%) | 3,142 (20.6%) | 3,273 (21.4%) | 192 (1.3%) | 139 (0.9%) | N/A | N/A | 3,334 (11.1%) | 3,412 (11.3%) | 0.00 |
| Lab values- NT-proBNP; n (%)<br>Lab values- NT-proBNP (within 3 months); n (%) | 42 (0.3%)<br>34 (0.2%) | 61 (0.4%)<br>44 (0.3%) | :: | : | N/A<br>N/A | N/A<br>N/A | #VALUE!<br>#VALUE! | #VALUE! | 1 |
| Lab values- NT-proBNP (within 6 months); n (%)<br>Lab values- Total cholesterol (mg/dl) v2; n (%) | 42 (0.3%)<br>3,012 (19.7%) | 61 (0.4%)<br>3,125 (20.5%) | 174 (1.2%) | 137 (0.9%) | N/A<br>N/A | N/A<br>N/A | #VALUE!<br>3,186 (10.6%) | #VALUE!<br>3,262 (10.8%) | - 0.00 |
| Lab values-Total cholesterol (mg/dl) (within 3 months) v2; n (%) | 1,805 (11.8%) | 1,886 (12.3%) | 97 (0.7%) | 79 (0.5%) | N/A | N/A | 1,902 (6.3%) | 1,965 (6.5%) | 0.00 |
| Lab values- Total cholesterol (mg/dl) (within 6 months) v2; n (%) | 3,012 (19.7%)<br>2,951 (19.3%) | 3,125 (20.5%) | 174 (1.2%) | 137 (0.9%)<br>139 (0.9%) | N/A | N/A | 3,186 (10.6%) | 3,262 (10.8%) | 0.00 |
| Lab values-Triglyceride level (mg/dl); n (%) Lab values-Triglyceride level (mg/dl) (within 3 months); n (%) | 2,951 (19.3%)<br>1,771 (11.6%) | 3,091 (20.2%)<br>1,870 (12.2%) | 171 (1.2%)<br>98 (0.7%) | 80 (0.5%) | N/A<br>N/A | N/A<br>N/A | 3,122 (10.4%)<br>1,869 (6.2%) | 3,230 (10.7%)<br>1,950 (6.5%) | 0.00 |
| Lab values-Triglyceride level (mg/dl) (within 6<br>months); n (%) | 2,951 (19.3%) | 3,091 (20.2%) | 171 (1.2%) | 139 (0.9%) | N/A | N/A | 3.122 (10.4%) | 3,230 (10.7%) | 0.00 |
| Lab result number-HbA1c (%) mean (only 2 to 20 included) v4 | | | | | N/A | N/A | 30,122 | 30,122 | |
| mean (sd)<br>median [IQR] | 6.40 (1.12)<br>6.10 (5.75, 6.80) | 6.39 (1.20)<br>6.10 [5.70, 6.80] | 6.82 (1.24)<br>6.40 (5.93, 7.38) | 6.91 (1.52)<br>6.50 (6.00, 7.40) | N/A<br>N/A | N/A<br>N/A | 6.61 (1.18) | 6.65 (1.37) | -0.03 |
| Missing; n (%)<br>Lab result number-BNP mean v2 | 13,085 (85.7%) | 13,041 (85.4%) | 14,685 (98.9%) | 14,710 (99.1%) | N/A<br>N/A | N/A<br>N/A | 27,770 (92.2%) | 27,751 (92.1%) | #DIV/0! |
| mean (sd)<br>median [IQR] | | 327.40 (485.45)<br>199.30 [101.17, 400.30] | | 716.39 (1,080.94)<br>312.25 [137.62, 545.00] | N/A<br>N/A | N/A<br>N/A | 411.62 (538.40) | 519.16 (833.97) | -0.15 |
| Missing; n (%)<br>Lab result number-BUN (mg/dl) mean v2 | 15,007 (98.3%) | 14,949 (97.9%) | 14,812 (99.8%) | 14,827 (99.9%) | N/A<br>N/A | N/A<br>N/A | | | |
| mean (sd)<br>median (IQR) | 18.06 (6.33)<br>17.00 [14.00, 21.00] | 18.01 (6.20)<br>17.00 [14.00, 21.00] | 869.98 (13,695.52)<br>17.00 [14.00, 20.00]<br>14,591 (98.3%) | 18.61 (6.49)<br>18.00 [15.00, 21.00] | N/A<br>N/A | N/A<br>N/A | 438.02 (9615.95) | 18.31 (6.34) | 0.06 |
| Missing; n (%) Lab result number-Creatinine (mg/dl) mean (only 0.1 to 15 included) v3 | 10,928 (71.6%) | 10,579 (69.3%) | 14,591 (98.3%) | 14,618 (98.4%) | N/A<br>N/A | N/A<br>N/A | | | |
| mean (sd)<br>median (IQR) | 0.97 (0.25)<br>0.94 [0.80, 1.10] | 0.97 (0.23)<br>0.94 [0.81, 1.09] | 0.97 (0.24)<br>0.94 [0.80, 1.08] | 1.00 (0.25)<br>0.98 [0.85, 1.13] | N/A<br>N/A | N/A<br>N/A | 0.97 (0.25) | 0.98 (0.24) | -0.04 |
| Missing; n (%) Lab result number- HDL level (mg/dl) mean (only | 10,873 (71.2%) | 10,470 (68.6%) | 14,582 (98.2%) | 14,615 (98.4%) | N/A | N/A | | | |
| =<5000 included) v2<br>mean (sd) | 51.89 (16.24) | 52.65 (17.24) | 45.20 (16.08) | 45.00 (13.88) | N/A<br>N/A | N/A<br>N/A | 48.59 (16.16) | 48.88 (15.67) | -0.02 |
| median (IQR)<br>Missing; n (%) | 49.50 [41.00, 60.25]<br>12,338 (80.8%) | 50.00 [41.00, 62.00]<br>12,208 (79.9%) | 43.25 [35.88, 52.00]<br>14,675 (98.8%) | 44.00 [35.12, 52.75]<br>14,709 (99.1%) | N/A<br>N/A | N/A<br>N/A | | | |
| Lab result number-LDL level (mg/dl) mean (only<br>=<\$000 included) v2 | | | | | N/A | N/A | | | |
| mean (sd)<br>median (IQR) | 90.04 (33.51)<br>87.00 (67.00, 111.00) | 87.75 (33.30)<br>84.00 [65.00, 106.50] | 88.64 (36.83)<br>85.00 [64.00, 109.25] | 88.11 (32.58)<br>87.10 [64.75, 111.25] | N/A<br>N/A | N/A<br>N/A | 89.35 (35.19) | 87.93 (32.95) | 0.04 |
| Missing; n (%) Lab result number-Total cholesterol (mg/dl) mean | 12,217 (80.0%) | 12,075 (79.1%) | 14,680 (98.9%) | 14,719 (99.1%) | N/A<br>N/A | N/A<br>N/A | | | |
| (only=<5000 included) v2<br>mean (sd)<br>median [IQR] | 168.20 (41.65) | 165.29 (40.13)<br>162.00 [138.00, 190.00] | 160.92 (47.56) | 160.86 (41.76)<br>164.00 [132.50, 187.00] | N/A<br>N/A<br>N/A | N/A<br>N/A<br>N/A | 164.61 (44.66) | 163.11 (40.94) | 0.04 |
| Missing; n (%) Lab result number-Triglyceride level (mg/dl) mean | 12,266 (80.3%) | 12,150 (79.6%) | 14,676 (98.8%) | 14,712 (99.1%) | N/A | N/A | | | |
| (only =<5000 included) v2<br>mean (sd) | 128.76 (82.61) | 122.22 (73.94) | 137.46 (73.77) | 140.81 (71.38) | N/A<br>N/A | N/A<br>N/A | 133.05 (78.38) | 131.38 (72.69) | 0.02 |
| median (IQR)<br>Missing; n (%) | 112.00 [82.00, 153.50]<br>12,322 (80.7%) | | 125.50 [94.00, 164.00]<br>14,679 (98.9%) | 130.00 [96.50, 167.00]<br>14,710 (99.1%) | N/A<br>N/A | N/A<br>N/A | | | |
| Lab result number-Hemoglobin mean (only >0 included) | | | | | N/A | N/A | | | |
| mean (sd)<br>median [IQR] | 13.62 (1.68)<br>13.60 (12.60, 14.70) | 13.67 (1.62)<br>13.70 [12.65, 14.70] | 699.98 (9,732.82)<br>13.55 [12.53, 14.72] | 13.69 (1.84)<br>13.70 [12.87, 14.76] | N/A<br>N/A | N/A<br>N/A | 351.97 (6833.64) | 13.68 (1.73) | 0.07 |
| Missing; n (%) Lab result number-Serum sodium mean (only > 90 | 11,942 (78.2%) | 11,699 (76.6%) | 14,648 (98.6%) | 14,667 (98.8%) | N/A | N/A | | | |
| and < 190 included)mean (sd) | 140.28 (2.98) | 140.22 (3.00) | 139.19 (2.88) | 139.82 (2.30) | N/A<br>N/A | N/A<br>N/A | 139.74 (2.93) | 140.02 (2.68) | -0.10 |
| median [IQR]Missing; n (%) Lab result number-Albumin mean (only >0 and <=10 | 11,075 (72.5%) | 140.50 [139.00, 142.00]<br>10,754 (70.4%) | 14,595 (98.3%) | 14,639 (98.6%) | N/A<br>N/A | N/A<br>N/A | | | |
| included)mean (sd) | 4.15 (0.34) | 4.17 (0.34) | 3.98 (0.77) | 4.13 (0.47) | N/A<br>N/A | N/A<br>N/A | 4.07 (0.59) | 4.15 (0.41) | -0.16 |
| median [IQR] | 4.20 [4.00, 4.40] | 4.20 [4.00, 4.40] | 4.10 [3.80, 4.40] | 4.20 [3.90, 4.40] | N/A | N/A | | | |

# Table 1: Matched

| Missing; n (%)<br>Lab result number-Glucose (fasting or random) mean | 11,535 (75.5%) | 11,360 (74.4%) | 14,655 (98.7%) | 14,686 (98.9%) | N/A | N/A | | | |
|---|---|---|---|---|---|---|---|---|---|
| (only 10-1000 included)<br>mean (sd) | 110.11 (33.77) | 110.43 (36.05) | 128.77 (45.98) | 131.44 (51.52) | N/A<br>N/A | N/A<br>N/A | 119.31 (40.26) | 120.79 (44.36) | -0.03 |
| median (IQR)Missing; n (%) | 101.00 [92.00, 117.00]<br>11,123 (72.8%) | 101.00 [92.00, 116.00]<br>10,823 (70.9%) | 115.00 [97.00, 144.75]<br>14,600 (98.3%) | 116.25 [97.83, 143.31]<br>14,639 (98.6%) | N/A<br>N/A | N/A<br>N/A | | | |
| Lab result number-Potassium mean (only 1-7<br>included) | | | | | N/A | N/A | | | |
| mean (sd)<br>median [IQR] | 4.36 (0.44)<br>4.35 [4.10, 4.60] | 4.39 (0.43)<br>4.40 [4.10, 4.65] | 4.32 (0.41)<br>4.30 [4.10, 4.57] | 4.37 (0.40)<br>4.40 [4.10, 4.60] | N/A<br>N/A | N/A<br>N/A | 4.34 (0.43) | 4.38 (0.42) | -0.09 |
| Missing; n (%) Comorbidity Scores | 10,855 (71.1%) | 10,470 (68.6%) | 14,599 (98.3%) | 14,632 (98.5%) | N/A | N/A | | | |
| CCI (180 days)- ICD9 and ICD10 v2<br>mean (sd) | 3.50 (1.86) | 3.50 (1.84) | 3.22 (1.73) | 3.20 (1.71) | 2.20 (2.00) | 2.22 (2.02) | 3.36 (1.80) | 3.35 (1.78) | 0.01 |
| median [IQR]<br>Frailty Score: Qualitative Version 365 days as | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | 3.00 [2.00, 4.00] | 3.00 [2.00, 4.00] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | | | |
| Categories, v1<br>0; n (%) | 6,480 (42.4%) | 5,808 (38.0%) | 2,847 (19.2%) | 2,765 (18.6%) | 80,137 (100.0%) | 80,137 (100.0%) | 89,464 (81.1%) | 88,710 (80.5%) | 0.00 |
| 1 to 2; n (%)<br>3 or more; n (%) | 4,987 (32.7%)<br>3,806 (24.9%) | 5,444 (35.6%)<br>4,021 (26.3%) | 5,982 (40.3%)<br>6,020 (40.5%) | 6,121 (41.2%)<br>5,963 (40.2%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 10,969 (9.9%)<br>9,826 (8.9%) | 11,565 (10.5%)<br>9,984 (9.1%) | 0.00<br>0.00 |
| Frailty Score: Empirical Version 365 days as<br>Categories, v3 | 1 344 (8 8%) | | | | | 63 584 (79 3%) | | | |
| <0.12908; n (%)<br>0.12908 - 0.1631167; n (%) | 4,185 (27.4%) | 1,533 (10.0%)<br>4,252 (27.8%)<br>9,488 (62.1%) | 1,237 (8.3%)<br>4,009 (27.0%) | 1,288 (8.7%)<br>4,061 (27.3%) | 63,958 (79.8%)<br>7,169 (8.9%) | 7,168 (8.9%) | 66,539 (60.3%)<br>15,363 (13.9%) | 66,405 (60.2%)<br>15,481 (14.0%)<br>28.373 (25.7%) | 0.00 |
| >= 0.1631167; n (%)<br>Non-Frailty; n (%) | 9,744 (63.8%)<br>8,075 (52.9%) | 9,488 (62.1%)<br>8,222 (53.8%) | 9,603 (64.7%)<br>7,317 (49.3%) | 9,500 (64.0%)<br>7,321 (49.3%) | 9,010 (11.2%)<br>1,831 (2.3%) | 9,385 (11.7%)<br>1,475 (1.8%) | 28,357 (25.7%)<br>17,223 (15.6%) | 28,373 (25.7%)<br>17,018 (15.4%) | 0.00<br>0.00 |
| Frailty Score (mean): Qualitative Version 365 days, v1mean (sd) | 1.62 (2.14) | 1.69 (2.07) | 2.40 (2.09) | 2.39 (2.08) | 0.09 (0.06) | 0.09 (0.06) | 2.00 (2.12) | 2.04 (2.07) | -0.02 |
| median (IQR) Frailty Score (mean): Empirical Version 365 days, v2 | 1.00 [0.00, 2.00] | 1.00 [0.00, 3.00] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0.07 [0.05, 0.12] | 0.07 [0.04, 0.12] | 2.00 (2.12) | 2.04 (2.07) | -0.02 |
| mean (sd)median (IQR) | 0.19 (0.06)<br>0.18 [0.15, 0.22] | 0.19 (0.06)<br>0.18 [0.15, 0.22] | 0.18 (0.05)<br>0.17 (0.15, 0.21) | 0.18 (0.05)<br>0.17 [0.15, 0.21] | 13.79 (10.60)<br>11.48 [6.52, 18.58] | 13.94 (11.23)<br>11.41 [6.23, 18.92] | 0.19 (0.06) | 0.19 (0.06) | 0.00 |
| Healthcare Utilization Any hospitalization; n (%) | 4.088 (26.8%) | 4.353 (28.5%) | 4.929 (33.2%) | 4.940 (33.3%) | 27.061 (33.8%) | 27.502 (34.3%) | 36.078 (32.7%) | 36.795 (33.4%) | 0.00 |
| Any hospitalization within prior 30 days; n (%)<br>Any hospitalization during prior 31-180 days; n (%) | 2,665 (17.4%)<br>1,771 (11.6%) | 2,680 (17.5%)<br>1,906 (12.5%) | 3,263 (22.0%)<br>1,940 (13.1%) | 3,266 (22.0%)<br>1,967 (13.2%) | 17,754 (22.2%)<br>11,741 (14.7%) | 17,978 (22.4%) | 23,682 (21.5%)<br>15,452 (14.0%) | 23,924 (21.7%)<br>15,663 (14.2%) | 0.00 |
| Endocrinologist Visit; n (%) Endocrinologist Visit (30 days prior); n (%) | 423 (2.8%)<br>121 (0.8%) | 422 (2.8%)<br>130 (0.9%) | 485 (3.3%)<br>169 (1.1%) | 480 (3.2%)<br>151 (1.0%) | 3,229 (4.0%)<br>956 (1.2%) | 3,111 (3.9%)<br>926 (1.2%) | 4,137 (3.8%)<br>1,246 (1.1%) | 4,013 (3.6%)<br>1,207 (1.1%) | 0.00 |
| Endocrinologist Visit (31 to 180 days prior); n (%)<br>Internal medicine/family medicine visits; n (%) | 357 (2.3%)<br>13,081 (85.6%) | 341 (2.2%)<br>13,272 (86.9%) | 394 (2.7%)<br>12,120 (81.6%) | 399 (2.7%)<br>11.913 (80.2%) | 2,719 (3.4%)<br>66,414 (82.9%) | 2,622 (3.3%)<br>67,563 (84.3%) | 3,470 (3.1%)<br>91,615 (83.1%) | 3,362 (3.0%)<br>92,748 (84.1%) | 0.00<br>0.00 |
| Internal medicine/family medicine visits (30 days<br>prior) v2; n (%) | 8,371 (54.8%) | 8,426 (55.2%) | 7,582 (51.1%) | 7,465 (50.3%) | 42,114 (52.6%) | 41,751 (52.1%) | 58,067 (52.7%) | 57,642 (52.3%) | 0.00 |
| Internal medicine/family medicine visits (31 to 180 days prior) v2; n (%) | 11,810 (77.3%) | 11,921 (78.1%) | 11,016 (74.2%) | 10,766 (72.5%) | 58,410 (72.9%) | 59,572 (74.3%) | 81,236 (73.7%) | 82,259 (74.6%) | 0.00 |
| Cardiologist visit; n (%)<br>Number of Cardiologist visits (30 days prior); n (%) | 11,538 (75.5%)<br>8,214 (53.8%) | 12,069 (79.0%)<br>8,242 (54.0%) | 9,253 (62.3%)<br>6,208 (41.8%) | 9,102 (61.3%)<br>6,079 (40.9%) | 63,920 (79.8%)<br>46,109 (57.5%) | 66,537 (83.0%)<br>46,119 (57.6%) | 84,711 (76.8%)<br>60,531 (54.9%) | 87,708 (79.5%)<br>60,440 (54.8%) | 0.00<br>0.00 |
| Number of Cardiologist visits (31 to 180 days prior);<br>n (%) | 8,453 (55.3%) | 8,712 (57.0%) | 7,212 (48.6%) | 6,953 (46.8%) | 46,069 (57.5%) | 47,552 (59.3%) | 61,734 (56.0%) | 63,217 (57.3%) | 0.00 |
| Electrocardiogram v2; n (%)<br>Use of glucose test strips; n (%) | 10,536 (69.0%)<br>138 (0.9%) | 11,542 (75.6%)<br>157 (1.0%) | 10,205 (68.7%)<br>114 (0.8%) | 11,063 (74.5%)<br>133 (0.9%) | 60,573 (75.6%)<br>907 (1.1%) | 64,303 (80.2%)<br>988 (1.2%) | 81,314 (73.7%)<br>1,159 (1.1%) | 86,908 (78.8%)<br>1,278 (1.2%) | -0.01<br>0.00 |
| Dialysis; n (%)<br>Naive new user v8 Copy; n (%) | 1 (0.0%)<br>12,399 (81.2%) | 0 (0.0%)<br>12,421 (81.3%) | 0 (0.0%)<br>12,023 (81.0%) | 0 (0.0%)<br>11,989 (80.7%) | 14,760 (18.4%) | 14,638 (18.3%) | #VALUE!<br>39,182 (35.5%) | #VALUE!<br>39,048 (35.4%) | #VALUE!<br>0.00 |
| N antidiabetic drugs at index date v3 Copy<br>mean (sd) | 0.22 (0.56) | 0.22 (0.58) | 0.24 (0.62) | 0.24 (0.63) | 0.23 (0.58) | 0.22 (0.57) | 0.23 (0.58) | 0.22 (0.58) | 0.02 |
| median [IQR]<br>number of different/distinct medication<br>prescriptions | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | | |
| mean (sd) | 9.21 (4.49)<br>9.00 [6.00, 12.00] | 9.27 (4.57)<br>9.00 (6.00, 12.00) | 9.70 (4.58)<br>9.00 (6.00, 12.00) | 9.69 (4.72)<br>9.00 (6.00, 12.00) | 9.75 (4.49)<br>9.00 [7.00, 12.00] | 9.84 (4.55)<br>9.00 [7.00, 12.00] | 9.67 (4.50) | 9.74 (4.58) | -0.02 |
| Number of Hospitalizations<br>mean (sd) | 0.33(0.61) | 0.33 (0.57) | 0.38 (0.59) | 0.38 (0.58) | 0.43 (0.70) | 0.43 (0.70) | 0.41 (0.67) | 0.41 (0.67) | 0.00 |
| median [IQR]<br>Number of hospital days | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | | | |
| mean (sd)<br>median [IQR] | 1.71 (4.11)<br>0.00 (0.00, 2.00) | 1.72 (4.67)<br>0.00 [0.00, 2.00] | 1.94 (3.92)<br>0.00 (0.00, 3.00) | 1.92 (4.82)<br>0.00 [0.00, 3.00] | 2.42 (5.05)<br>0.00 (0.00, 3.00) | 2.41 (6.24)<br>0.00 [0.00, 3.00] | 2.26 (4.79) | 2.25 (5.87) | 0.00 |
| Number of Emergency Department (ED) visits v3<br>mean (sd) | 0.75 (1.46) | 0.76 (1.44) | 0.67 (2.44) | 0.69 (2.09) | 0.96 (1.92) | 1.00 (1.88) | 0.89 (1.94) | 0.93 (1.86) | -0.02 |
| median (IQR) Number of Office visits | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 2.00] | 0.00 [0.00, 2.00] | | | 0.00 |
| mean (sd)median [IQR] Number of Endocrinologist visits | 5.55 (4.15)<br>5.00 [3.00, 8.00] | 5.59 (3.91)<br>5.00 (3.00, 7.00) | 6.05 (4.59)<br>5.00 [3.00, 8.00] | 5.98 (4.28)<br>5.00 [3.00, 8.00] | 13.20 (12.77)<br>10.00 [5.00, 17.00] | 13.26 (11.74)<br>10.00 [6.00, 17.00] | 11.18 (11.12) | 11.22 (10.24) | 0.00 |
| mean (sd)median [IQR] | 0.09 (0.86)<br>0.00 (0.00, 0.00) | 0.09 (0.88)<br>0.00 (0.00, 0.00) | 0.12 (1.05)<br>0.00 (0.00, 0.00) | 0.10 (0.95)<br>0.00 [0.00, 0.00] | 0.16 (1.33)<br>0.00 [0.00, 0.00] | 0.16 (1.33)<br>0.00 [0.00, 0.00] | 0.14 (1.24) | 0.14 (1.23) | 0.00 |
| Number of internal medicine/family medicine visitsmean (sd) | 9.28 (12.23) | 9.34 (12.11) | 7.57 (11.66) | 7.44 (11.28) | 7.89 (9.77) | 7.90 (9.87) | 8.04 (10.41) | 8.04 (10.40) | 0.00 |
| median (IQR) Number of Cardiologist visits | 6.00 [2.00, 12.00] | 6.00 [2.00, 12.00] | 4.00 [1.00, 9.00] | 4.00 [1.00, 9.00] | 5.00 [1.00, 11.00] | 5.00 [2.00, 11.00] | | , | |
| mean (sd)<br>median (IQR) | 5.17 (6.51)<br>3.00 [1.00, 7.00] | 5.26 (5.88)<br>4.00 [1.00, 8.00] | 3.57 (5.21)<br>2.00 (0.00, 5.00) | 3.55 (5.23)<br>2.00 [0.00, 5.00] | 5.65 (7.11)<br>3.00 [1.00, 8.00] | 5.72 (6.54)<br>4.00 [1.00, 8.00] | 5.30 (6.80) | 5.36 (6.29) | -0.01 |
| Number electrocardiograms received v2<br>mean (sd) | 2.16 (2.89) | 2.23 (2.51) | 1.90 (2.42) | 1.89 (2.05) | 2.32 (2.61) | 2.36 (2.40) | 2.24 (2.63) | 2.28 (2.37) | -0.02 |
| median [IQR]<br>Number of HbA1c tests ordered | 1.00 [0.00, 3.00] | 2.00 [1.00, 3.00] | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | | | |
| mean (sd)median [IQR] | 0.36 (0.67)<br>0.00 (0.00, 1.00) | 0.37 (0.66)<br>0.00 (0.00, 1.00) | 0.19 (0.50)<br>0.00 (0.00, 0.00) | 0.19 (0.50)<br>0.00 [0.00, 0.00] | 0.38 (0.68)<br>0.00 [0.00, 1.00] | 0.38 (0.68)<br>0.00 [0.00, 1.00] | 0.35 (0.66) | 0.35 (0.66) | 0.00 |
| Number of glucose tests orderedmean (sd)median (IOR) | 0.15 (2.00) | 0.18 (2.20) | 0.10 (0.49) | 0.13 (0.68) | 0.12 (0.53) | 0.14 (0.66) | 0.12 (0.89) | 0.14 (1.02) | -0.02 |
| median [IQR] Number of lipid tests orderedmean (sd) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 (0.00, 0.00) | 0.57 (0.76) | 0.58 (0.74) | -0.01 |
| median [IQR] Number of creatinine tests ordered | 0.00 (0.00, 1.00) | 0.00 [0.00, 1.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.57 (0.76) | 0.38 (0.74) | -0.01 |
| mean (sd) | 0.07 (0.36)<br>0.00 (0.00, 0.00) | 0.07 (0.37) | 0.06 (0.34) | 0.06 (0.33) | 0.10 (0.42)<br>0.00 [0.00, 0.00] | 0.10 (0.40)<br>0.00 (0.00, 0.00) | 0.09 (0.40) | 0.09 (0.39) | 0.00 |
| Number of BUN tests ordered<br>mean (sd) | 0.04(0.26) | 0.04 (0.27) | 0.04 (0.25) | 0.04 (0.27) | 0.06 (0.32) | 0.06 (0.30) | 0.05 (0.30) | 0.05 (0.29) | 0.00 |
| median [IQR]<br>Number of tests for microalbuminuria | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 (0.00, 0.00) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | | | |
| mean (sd)median [IQR] | 0.18 (0.62)<br>0.00 (0.00, 0.00) | 0.17 (0.59)<br>0.00 (0.00, 0.00) | 0.08 (0.40)<br>0.00 (0.00, 0.00) | 0.08 (0.40)<br>0.00 [0.00, 0.00] | 0.11 (0.40)<br>0.00 [0.00, 0.00] | 0.11 (0.40)<br>0.00 [0.00, 0.00] | 0.12 (0.44) | 0.11 (0.43) | 0.02 |
| Total N distinct ICD9/ICD10 diagnoses at the 3rd<br>digit level Copy | | | | | | | | | |
| mean (sd)<br>median (IQR) | 9.31 (10.15)<br>7.00 (0.00, 14.00) | 9.08 (10.16)<br>6.00 [0.00, 14.00] | 5.28 (7.97)<br>2.00 (0.00, 7.00) | 5.18 (7.95)<br>1.00 [0.00, 7.00] | 9.65 (11.24)<br>6.00 (0.00, 15.00) | 9.65 (11.37)<br>6.00 (0.00, 15.00) | 9.01 (10.71) | 8.97 (10.81) | 0.00 |
| For PS<br>Hemorrhagic stroke+Other cerebrovascular<br>disease+Cerebrovascular procedure (for PS); n (%) | 400 /2 20/1 | 400 (2.29/) | 421 (2.99/) | 435 (3.08) | 2 424 (2 09) | 3 410 /3 09/1 | 2 242 (2 0%) | 2 224 (2 09/) | 0.00 |
| Occurrence of creatinine tests ordered (for PS); n (%) | 498 (3.3%)<br>843 (5.5%) | 488 (3.2%)<br>852 (5.6%) | 421 (2.8%)<br>705 (4.7%) | 426 (2.9%)<br>700 (4.7%) | 2,424 (3.0%)<br>6,314 (7.9%) | 2,410 (3.0%)<br>6,358 (7.9%) | 3,343 (3.0%)<br>7,862 (7.1%) | 3,324 (3.0%)<br>7,910 (7.2%) | 0.00 |
| Occurrence of BUN tests ordered (for PS); n (%) Occurrence of chronic renal insufficiency w/o CKD | 448 (2.9%) | 467 (3.1%) | 406 (2.7%) | 414 (2.8%) | 3,672 (4.6%) | 3,754 (4.7%) | 4,526 (4.1%) | 4,635 (4.2%) | 0.00 |
| (for PS) v2; n (%)<br>Chronic kidney disease Stage 1-2 (for PS); n (%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%)<br>#VALUE! | 000 (0.0%)<br>#VALUE! | #DIV/0!<br>#VALUE! |
| Chronic kidney disease Stage 3-6 (for PS); n (%)<br>Bladder stones+Kidney stones (for PS); n (%) | 0 (0.0%)<br>234 (1.5%) | 0 (0.0%)<br>240 (1.6%) | 0 (0.0%)<br>263 (1.8%) | 0 (0.0%)<br>293 (2.0%) | 0 (0.0%)<br>1,254 (1.6%) | 0 (0.0%)<br>1,293 (1.6%) | 000 (0.0%)<br>1,751 (1.6%) | 000 (0.0%)<br>1,826 (1.7%) | #DIV/0!<br>0.00 |
| Diabetes with peripheral circulatory<br>disorders+Gangrene+Osteomyelitis(for PS) v3 with | | | | | | | | | |
| ICD10 Copy; n (%)<br>Age decile (for PS) v3 | 400 (2.6%) | 420 (2.7%) | 295 (2.0%) | 281 (1.9%) | 2,113 (2.6%) | 2,100 (2.6%) | 2,808 (2.5%) | 2,801 (2.5%) | 0.00 |
| Age decile 1<br>Age decile 2 | 84 (0.5%)<br>125 (0.8%) | 109 (0.7%)<br>125 (0.8%) | 138 (0.9%)<br>228 (1.5%) | 104 (0.7%)<br>201 (1.4%) | 4,207 (5.2%)<br>4,785 (6.0%) | 4,193 (5.2%)<br>4,825 (6.0%) | 4,429 (4.0%)<br>5,138 (4.7%) | 4,406 (4.0%)<br>5,151 (4.7%) | 0.00 |
| Age decile 3<br>Age decile 4 | 285 (1.9%)<br>290 (1.9%) | 344 (2.3%)<br>336 (2.2%) | 229 (1.5%)<br>410 (2.8%) | 231 (1.6%)<br>364 (2.5%) | 2,686 (3.4%)<br>5,791 (7.2%) | 2,680 (3.3%)<br>5,956 (7.4%) | 3,200 (2.9%)<br>6,491 (5.9%) | 3,255 (3.0%)<br>6,656 (6.0%) | 0.00<br>0.00 |
| Age decile 5<br>Age decile 6 | 615 (4.0%)<br>1,006 (6.6%) | 661 (4.3%)<br>1,023 (6.7%) | 626 (4.2%)<br>596 (4.0%) | 626 (4.2%)<br>538 (3.6%) | 6,235 (7.8%)<br>6,771 (8.4%) | 6,207 (7.7%)<br>6,805 (8.5%) | 7,476 (6.8%)<br>8,373 (7.6%) | 7,494 (6.8%)<br>8,366 (7.6%) | 0.00 |
| Age decile 7<br>Age decile 8 | 1,391 (9.1%)<br>2,357 (15.4%) | 1,463 (9.6%)<br>2,204 (14.4%) | 1,072 (7.2%)<br>1,109 (7.5%) | 1,099 (7.4%)<br>1,214 (8.2%) | 7,738 (9.7%)<br>10,840 (13.5%) | 7,940 (9.9%)<br>10,712 (13.4%) | 10,201 (9.3%)<br>14,306 (13.0%) | 10,502 (9.5%)<br>14,130 (12.8%) | 0.00 |
| Age decide 9Age decide 10 | 3,302 (21.6%)<br>5,818 (38.1%) | 3,097 (20.3%)<br>5,911 (38.7%) | 2,371 (16.0%)<br>8,070 (54.3%) | 2,419 (16.3%)<br>8,053 (54.2%) | 12,490 (15.6%)<br>18,594 (23.2%) | 12,405 (15.5%)<br>18,414 (23.0%) | 18,163 (16.5%)<br>32,482 (29.5%) | 17,921 (16.3%)<br>32,378 (29.4%) | 0.00<br>0.00 |
| Alcohol abuse or dependence+Drug abuse or<br>dependence (for PS); n (%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | 000 (0.0%) | 000 (0.0%) | #DIV/01 |
| Diabetes with other ophthalmic<br>manifestations+Retinal detachment, vitreous<br>hemorrhage, vitrectomy+Retinal laser coagulation | | | | | | | | | |
| therapy (for PS); n (%) Other atherosclerosis+Cardiac conduction | 51 (0.3%) | 51 (0.3%) | 117 (0.8%) | 116 (0.8%) | 555 (0.7%) | 579 (0.7%) | 723 (0.7%) | 746 (0.7%) | 0.00 |
| disorders+Other CVD (for PS) v2 Copy; n (%)<br>Previous cardiac procedure (CABG or PTCA or Stent) + | 6,723 (44.0%) | 6,783 (44.4%) | 6,490 (43.7%) | 6,462 (43.5%) | 29,955 (37.4%) | 29,898 (37.3%) | 43,168 (39.2%) | 43,143 (39.1%) | 0.00 |
| History of CABG or PTCA (for PS) v3; n (%)<br>Hyperthyroidism + Hypothyroidism + Other disorders | 1,500 (9.8%) | 1,484 (9.7%) | 877 (5.9%) | 876 (5.9%) | 8,694 (10.8%) | 8,876 (11.1%) | 11,071 (10.0%) | 11,236 (10.2%) | 0.00 |
| of thyroid gland (for PS); n (%) Delirium + Psychosis (for PS); n (%) | 3,257 (21.3%)<br>444 (2.9%) | 3,193 (20.9%)<br>425 (2.8%) | 2,528 (17.0%)<br>371 (2.5%) | 2,647 (17.8%)<br>371 (2.5%) | 10,893 (13.6%)<br>2,665 (3.3%) | 11,074 (13.8%)<br>2,620 (3.3%) | 16,678 (15.1%)<br>3,480 (3.2%) | 16,914 (15.3%)<br>3,416 (3.1%) | 0.00 |
| Any use of Meglitinides (for PS); n (%) Any use of AGIs (for PS); n (%) CKD stage 3.6.4 diabatic (for PS): n (%) | 20 (0.1%)<br>12 (0.1%)<br>1 (0.0%) | 20 (0.1%) | 51 (0.3%) | 43 (0.3%)<br>18 (0.1%) | 172 (0.2%)<br>47 (0.1%) | 204 (0.3%)<br>51 (0.1%) | 243 (0.2%)<br>#VALUE!<br>#VALUE! | 267 (0.2%)<br>#VALUE!<br>#VALUE! | 0.00<br>#VALUE!<br>#VALUE! |
| CKD stage 3-6 + dialysis (for PS); n (%) | 1 (0.0%) | 0 (0.0%) | 0 (0.0%) | 0 (0.0%) | | | #VALUE! | #VALUE! | #VALUE! |